Replication of Ticagrelor versus Clopidogrel in Patients with Acute Coronary Syndromes (PLATO Trial)

January 13, 2020

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Ticagrelor versus Clopidogrel in Patients with Acute Coronary Syndromes (PLATO trial)

#### 1.2 <u>Intended aim(s)</u>

Compared ticagrelor (180-mg loading dose, 90 mg twice daily thereafter) and clopidogrel (300-to-600-mg loading dose, 75 mg daily thereafter) for the prevention of cardiovascular events in 18,624 patients admitted to the hospital with an acute coronary syndrome, with or without ST-segment elevation.

#### 1.3 Primary endpoint for replication and RCT finding

a composite of death from vascular causes, myocardial infarction, or stroke

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Estimated that 1780 such events would be required to achieve 90% power to detect a relative risk reduction of 13.5% in the rate of the primary end point in the ticagrelor group as compared with the clopidogrel group, given an event rate of 11% in the clopidogrel group at 12 months.

#### 1.5 Primary trial estimate targeted for replication

HR = 0.84 (95% CI 0.77–0.92) comparing ticagrelor to clopidogrel (Wallentin et al., 2009)

### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

#### 3. Data Source(s)

United/Optum, MarketScan

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing ticagrelor 90mg twice daily to clopidogrel 75mg daily. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of ticagrelor 90mg or the comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation.

#### 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

#### 5.2.1 Eligible cohort entry dates

Market availability of ticagrelor in the U.S. started on 2011-07-20.

- For Marketscan: 2011-07-20 to 2017-12-31 (end of data availability).
- For Optum: 2011-07-20 to 2019-03-31 (end of data availability).

#### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

### 5.3 Flowchart of the study cohort assembly

| | Optum | | MarketScan | |
|---|---|---|---|---|
| | Less Excluded | Remaining | | Remaining |
| Less Excluded Patients | Patients | Patients | Less Excluded Patients | Patients |
| All patients | | 75,524,500 | | 191,990,035 |
| Met cohort entry criteria: | | | | |
| Patients with hospitalization for potential ST-segment elevation or non-ST segment | -75275676 | 248,824 | -191715444 | 274,591 |
| elevation Acute Coronary Syndrome | | | | |

| Patients with sufficient enrollment period in the claims database | -33452 | 215,372 | -67391 | 207,200 |
|---|---|---|---|---|
| Parent: Excluded based on Start of Clopidogrel 75mg OR Ticagrelor 90mg (if never began 14 days after discharge) | -136791 | 78,581 | -119212 | 87,988 |
| Parent: Excluded based on Enrollment with allowed gap- from hospital discharge to 14 days after discharge | -610 | 77,971 | -1431 | 86,557 |
| Parent: Final cohort | | 77,971 | | 86,557 |
| Patients who initiate clopidogrel 75mg or ticagrelor 90mg 14 days within discharge from the ACS hospitalization | -245 | 77,726 | -23 | 86,534 |
| Patients with sufficient enrollment period covering post 14 days hospital discharge. | 0 | 77,726 | 0 | 86,534 |
| Patients with no prior use of clopidogrel | -5415 | 72,311 | -4841 | 81,693 |
| Patients with no prior use of ticagrelor | -842 | 71,469 | -799 | 80,894 |
| Patients without qualification in >1 exposure category | -46 | 71,423 | -44 | 80,850 |
| Patients with age 18 or older | 0 | 71,423 | -1 | 80,849 |
| Patients with risk factors such as age >=60, previous MI, CABG, TIA, Carotid stenosis, cerebral revascularizations, diabetes mellitus, peripheral artery disease, chronic renal dysfunction | -16839 | 54,584 | -22689 | 58,160 |
| Patients without contraindication to clopidogrel: moderate/severe liver disease 180 days prior to drug initiation | -3508 | 51,076 | -2609 | 55,551 |
| Patients without contraindication to clopidogrel: active bleeding or bleeding history 180 days prior to drug initiation | -978 | 50,098 | -2631 | 52,920 |
| Patients without contraindication to clopidogrel: major surgery 30 days prior to drug initiation | -549 | 49,549 | -482 | 52,438 |
| Patients not on concomitant oral/IV therapy with CYP3A inhibitors 90 days prior to drug initiation | -1011 | 48,538 | -1010 | 51,428 |
| Patients who do not require dialysis 180 days prior to drug initiation | -654 | 47,884 | -457 | 50,971 |
| Patients without clinically significant thrombocytopenia 180 days prior to drug initiation | -1108 | 46,776 | -1396 | 49,575 |
| Patients without clinically significant anemia 180 days prior to drug initiation | -3559 | 43,217 | -4869 | 44,706 |
| Excluded based on Exclusion #11 - Any other condition that may put the patient at risk- 180 days prior to drug initiation Patients without conditions that put individuals at risk or influence study results such as cardiogenic shock, severe hemodynamic instability, or active cancer 180 days prior to drug initiation. | -1764 | 41,453 | -3848 | 40,858 |
| Excluded based on Exclusion #13 - Pregnancy- 180 days prior to drug initiation Patients not pregnant | -7 | 41,446 | -9 | 40,849 |

Final cohort 41,446 40,849

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of ticagrelor. Initiation will be defined as starting treatment with ticagrelor or a comparator drug with no prior use of the corresponding drug in the past 6 months (washout period).

#### Comparator agents:

- Initiators of ticagrelor 90mg will be compared to initiators of
  - o Clopidogrel 75mg

#### 6.2 Preliminary covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Primary outcome</u>: 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality
- Secondary outcomes: Individual components:
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - o Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in Marketscan
    - In Optum, all-cause inpatient mortality + all-cause mortality for Medicare Advantage patients is used

Control outcome of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

- 1. Major bleeding (we expect to see a null association; Wallentin et al., 2009)
- 2. Pneumonia (we expect to see a null association)

#### **Control outcome definition**

| Outcome | Definition | Comments |
|---|---|---|
| Control Outcomes | | |
| Major bleeding | Any inpatient diagnosis of major bleeding code list provided in <b>Appendix A</b> | Same code list used for both outcome and major bleed exclusion criteria |
| Pneumonia | Any inpatient diagnosis of pneumonia: * 481 - PNEUMOCOCCAL PNEUMONIA [STREPTOCOCCUS PNEUMONIAE PNEUMONIA] * 482 - OTHER BACTERIAL PNEUMONIA * 483 - PNEUMONIA DUE TO OTHER SPECIFIED ORGANISM * 485 - BRONCHOPNEUMONIA ORGANISM UNSPECIFIED * 486 - PNEUMONIA ORGANISM UNSPECIFIED * 487.0 - INFLUENZA WITH PNEUMONIA * 507 - PNEUMONITIS DUE TO SOLIDS AND LIQUIDS * 482.0 - PNEUMONIA DUE TO KLEBSIELLA PNEUMONIAE * 482.1 - PNEUMONIA DUE TO PSEUDOMONAS * 482.2 - PNEUMONIA DUE TO HEMOPHILUS INFLUENZAE * 482.3 - PNEUMONIA DUE TO STREPTOCOCCUS * 482.30 - PNEUMONIA DUE TO STREPTOCOCCUS GROUP A * 482.32 - PNEUMONIA DUE TO STREPTOCOCCUS GROUP A | PPV = 85% (Aronsky, et al.; 2005); Note- The corresponding ICD-10 codes will also be used |

| * 482.39 - PNEUMONIA DUE TO OTHER STREPTOCOCCUS |
|---------------------------------------------------------------------------|
| * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS |
| * 482.40 - PNEUMONIA DUE TO STAPHYLOCOCCUS UNSPECIFIED |
| * 482.41 - METHICILLIN SUSCEPTIBLE PNEUMONIA DUE TO STAPHYLOCOCCUS AUREUS |
| * 482.42 - METHICILLIN RESISTANT PNEUMONIA DUE TO STAPHYLOCOCCUS AUREUS |
| * 482.49 - OTHER STAPHYLOCOCCUS PNEUMONIA |
| * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA |
| * 482.81 - PNEUMONIA DUE TO ANAEROBES |
| * 482.82 - PNEUMONIA DUE TO ESCHERICHIA COLI [E.COLI] |
| * 482.83 - PNEUMONIA DUE TO OTHER GRAM-NEGATIVE BACTERIA |
| * 482.84 - PNEUMONIA DUE TO LEGIONNAIRES' DISEASE |
| * 482.89 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA |
| * 482.9 - BACTERIAL PNEUMONIA UNSPECIFIED |
| * 483.0 - PNEUMONIA DUE TO MYCOPLASMA PNEUMONIAE |
| * 483.1 - PNEUMONIA DUE TO CHLAMYDIA |
| * 483.8 - PNEUMONIA DUE TO OTHER SPECIFIED ORGANISM |
| * 507.0 - PNEUMONITIS DUE TO INHALATION OF FOOD OR VOMITUS |
| * 507.1 - PNEUMONITIS DUE TO INHALATION OF OILS AND ESSENCES |
| * 507.8 - PNEUMONITIS DUE TO OTHER SOLIDS AND LIQUIDS |

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of ticagrelor and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.

Effectiveness research with Real World Data to support FDA's regulatory decision making

- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (ticagrelor and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator.
- Initiation of prasugrel

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7. Initial Feasibility Analysis

#### Aetion report links:

Optum: https://bwh-dope.aetion.com/projects/details/948/results/45952/result/0 Marketscan: https://bwh-dope.aetion.com/projects/details/949/results/45949/result/0

Date conducted: December 12, 2019

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of the overall study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report links:

<u>Optum:</u> https://bwh-dope.aetion.com/projects/details/948/results/45953/result/6 <u>Marketscan:</u> https://bwh-dope.aetion.com/projects/details/949/results/45950/result/6 Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

Date conducted: December 12, 2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/16/2019 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 1/3/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 9. Balance Assessment after PS matching

### Aetion report links (Ticagrelor vs. clopidogrel):

Optum: https://bwh-dope.aetion.com/projects/details/948/results/46989/result/0 Marketscan: https://bwh-dope.aetion.com/projects/details/949/results/46990/result/0

Date conducted: 01/05/2020

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 194 (0.69%) | 108 (0.77%) | 86 (0.62%) |
| Start of an additional exposure | 3,375 (12.07%) | 254 (1.82%) | 3,121 (22.32%) |
| End of index exposure | 11,280 (40.34%) | 5,799 (41.48%) | 5,481 (39.21%) |
| Specified date reached | 5,755 (20.58%) | 3,626 (25.94%) | 2,129 (15.23%) |
| End of patient enrollment | 5,042 (18.03%) | 3,039 (21.74%) | 2,003 (14.33%) |
| Switch to Prasugrel (for censoring) + nursing home admission | 2,314 (8.28%) | 1,154 (8.25%) | 1,160 (8.30%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|------------------------------------|--------------|---------------|
| Patient Group | Optum | Marketscan |
| Overall Patient Population | 163 [58-387] | 219 [85-409] |
| Referent | 228 [81-444] | 259 [113-451] |
| Exposure | 114 [40-310] | 179 [59-381] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan |
|--------------------------------|-------|------------|
| Risk per 1,000 patients (MACE) | 75.73 | 56.46 |

### **10. Final Power Assessment**

### Date conducted:

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).

#### o Pooled

For ticagrelor 90mg vs. clopidogrel 75mg (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 13,980 | Reference | 13,980 |
| Exposed | 13,980 | Exposed | 13,980 |
| Risk per 1,000 patients | 66.10 | Risk per 1,000 patients | 66.10 |
| Desired HR from RCT | 0.865 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1848.156 | Number of events expected | 1848.156 |
| Power | 0.876441293 | Power | 0.999883191 |

#### o Optum

■ For ticagrelor 90mg vs. clopidogrel 75mg (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 6,697 | Reference | 6,697 |
| Exposed | 6,697 | Exposed | 6,697 |
| Risk per 1,000 patients | 75.73 | Risk per 1,000 patients | 75.73 |
| Desired HR from RCT | 0.865 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1014.32762 | Number of events expected | 1014.32762 |
| Power | 0.636639088 | Power | 0.986722295 |

## MarketScan

For ticagrelor 90mg vs. clopidogrel 75mg (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 7,283 | Reference | 7,283 |
| Exposed | 7,283 | Exposed | 7,283 |
| Risk per 1,000 patients | 56.46 | Risk per 1,000 patients | 56.46 |
| Desired HR from RCT | 0.865 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 822.39636 | Number of events expected | 822.39636 |
| Power | 0.54759547 | Power | 0.964227735 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/16/2019 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 01/03/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns: 1/10/20

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.

### 12. Register study protocol on clinicalTrials.gov

#### **Date conducted:**

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

#### 13.1 For primary analysis:

• In the PS-matched cohort from Section 9, calculate the HR for each outcome for ticagrelor versus clopidogrel patients using a Cox proportional hazards model.

#### 13.2 For secondary analyses:

• In both pre-matched cohorts, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for ticagrelor versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

#### 14. Requested Results

#### 14.1 Results from primary and secondary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 15. References

Aronsky, Dominik, et al. Accuracy of Administrative Data for Identifying Patients with Pneumonia. American Journal of Medical Quality. 2005: 20(6);319–28. doi:10.1177/1062860605280358.

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. **page** 177

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

Wallentin L, Becker RC, Budaj A, et al. N Engl J Med 2009; 361:1045-1057

| ш | PLATO trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| - | FEATO trial definitions | Implementation in routine care | neleielices/ rationale | Color coding |
| | Trial details- Hazard Ratio, 0.84; S | 95% confidence interval [CI], 0.77 to 0.92 ) | Please see the following Google Drive for further details or any missing information:<br>https://drive.google.com/open?id=1WD618wrywXjEaXzHTcuk-VCrchb6b.gV. | Adequate mapping in claims |
| | EXPOSURE | E vs. COMPARISON | Not all ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping: https://www.nber.ore/data/icd9-icd-10-cm-and-ocs-crosswalk-general-equivalence-mapping.html | Intermediate mapping in claims |
| | Ticagrelor (90 mg twice daily) vs Clopidogrel (75mg daily) | Exposure) Ticagrelor<br>Reference) Clopidogrel | KEY TIME POINTS: Index event: Onset of Acute coronary syndrome (ACS) which becomes the indication for study drug (ticagregor or clopidogred) initiation Index hospitalization: Hospitalization for the treatment of index event Drug Initiation dates. New prescription claim for the study drug in patients with a record of index hospitalization in the previous 2 weeks. * We assume that the patient first initiates study drug in hospital and continues to be part of the initiator group as long as a prescription is filled within 2 weeks of discharge of ACS event. | Poor mapping or cannot be measured in claims |
| | PRIM | ARY OUTCOME | | Can't be measured in claims but not<br>important for the analysis |
| | The primary efficacy end point is time to first occurrence of death from vascular causes, myocardial infarction, or stroke. | Measured 1 day after drug initiation in diagnosis position specified below and inpatient care setting: Inpatient mortality/Mi/Stroke For Mi Any diagnosis position in inpatient care setting ICD-9 Dx 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care) For stroke Primary diagnosis position in inpatient care setting ICD-9 discharge diagnosis: 430.xx Subarachnoid hemorrhage (SAH) 431.xx Intracerebral hemorrhage (ICH) 433.xx1 Occlusion and stenosis of precerebral arteries with cerebral infarction 434.xx (excluding 434.xv) Occlusion and stenosis of cerebral arteries with cerebral infarction 436.x Acute, but ill-defined cerebrovascular events Mortality- See Mortality Sheet. | For MI: →PPV 94% in Medicare claims data [Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avom J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: solitorial positive predictive value on the basis of review of hospital records. American heart journal 2004;148:99-104.] →PPV 88.4% in commercially-insured population [Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. Pharmacoepidemiology and Drug Safety 2010;19:596-603.] For stroke: PPV angling from 80% to 98% for hemorrhagic stroke PPV rangling from 80% to 98% for hemorrhagic stroke PPV rangling from 80% to 98% for hemorrhagic stroke of identifying cerebrovascular accident or transient ischemic attack using administrative data. →[Tirschwell Dt, Longstreth WT, Jr. Validating administrative data in stroke research. Stroke; a journal of cerebral circulation 2002;33:2465-70.] →[Roumie Ct, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR, Validation of ICD-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | |
| | | SION CRITERIA | | |
| $\vdash$ | 1-4 ALL FO | DUR ARE REQUIRED | | |
| 1 | Hospitalized for potential ST-segment elevation or non - ST-segment elevation ACS, with onset during the previous 24 hours, documented by cardiac ischemic symptoms due to atherosclerosis of ≥10 minutes' duration at rest | Meesured 2 weeks prior to Index hospitalization in Inpatient, primary diagnosis position Acute MI: ICD-9 Dx 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care) ICD-10: I21.0x, I21.1x, I21.2x, I21.3x, I21.4x, I22.0x, I22.0x, I22.1x, I22.2x, I22.8x, I22.9x, I25.2x Unstable angina: ICD-9: 411.x ICD-10: I24.1x, I20.0x, I25.1x, I25.7x, I24.0x, I24.8x, I24.9x | | |
| 2 | ≥18 years of age | Measured at Index hospitalization Age >=18 | | |
| 3 | Not pregnant. Urinary and/or blood pregnancy tests are to be performed in women of child-bearing potential and repeated at least every 6 months. Women of child-bearing potential must be using ≥2 forms of reliable contraception, including one barrier method. | Please see exclusion #13 | | |
| 4 | With informed consent | N/A MEET COITEDIA BA OD BB | | |
| <u>-</u> | IN ADDITION TO 1-4, MEET CRITERIA 5A OR 5B | | | |
| 5A | ≥2 of the following 3 risk factors 1. ST-segment changes on ECG indicating ischemia. | * Note) In the claims, we are unable to measure ≥2 of the 3 risk factors | | |
| I | 1. 51 segment changes on ECG indicating scrienna. ST-segment depression or transient elevation ≥ 1 mm in two or more 2 contiguous leads | N/A | | |

| 3. One of the following: (a) ≥60 y of age Measured at Index hospitalization Age >= 60 Measured at Index hospitalization in any diagnosis position and inpatient or outpatient care setting as offerhed below: M: ICD 9 Active Mi: 410.xx. Old Mi: 412.xx CABG: Inpatient CPT-4: 33510 - 33536, 33545, 33572. Or Inpatient or outpatient ICD-9 procedure: 36.1x, 36.2x (c) CAD with ≥50% stenosis in ≥2 vessels N/A Measured any time prior to index hospitalization in any diagnosis position and inpatient or outpatient care setting as defined below: (coexpton: That -inpatient diagnosis only) Isohemic stroke: ICD 9: 435.xx TA (inpatient care) (d) Previous isohemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization Measured any time prior to index hospitalization in any diagnosis position and inpatient or outpatient care setting as defined below: (coexpton: That -inpatient diagnosis only) Isohemic stroke: ICD 9: 435.xx TA (inpatient diagnosis, any position): ICD 9: 435.xx Carotid stenosis: Carotid stenosis: Carotid stenos | ort study.* BMJ 2018;360:k119 of Heart Failure Hospitalization in gliflozin Comparative Effectiveness and it: |
|---|---|
| (a) ≥60 y of age Age >= 60 | ort study." BMJ 2018;360:k119 of Heart Failure Hospitalization in gliflozin Comparative Effectiveness and it: |
| Measured any time prior to index hospitalization in any diagnosis position and inpatient or outpatient care setting as defined below: MI: ICD 9 Acute MI: 410.xx, Old MI: 412.xx CABB: Inpatient CPT-4: 33510 - 33536, 33545, 33572. Or Inpatient or outpatient ICD-9 procedure: 36.1x, 36.2x (c) CAD with ≥50% stenosis in ≥2 vessels N/A Measured any time prior to index hospitalization in any diagnosis position and inpatient or outpatient care setting as defined below: (exception: TIA - Inpatient diagnosis only) Isobernal stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization (d) Previous ischemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization ME CABB: Inpatient or outpatient ICD-9 procedure: 36.1x, 36.2x N/A N/A Measured any time prior to index hospitalization in any diagnosis position and inpatient or outpatient care setting as defined below: (exception: TIA - Inpatient diagnosis only) Isobernal stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization (d) Previous ischemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization (d) Previous ischemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization (d) Previous ischemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization (d) Previous ischemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revescularization (exception: TIA - Inpatient diagnosis, any position): (CD-9: 435.xx TIA (Inpatient diagnosis, any position): (CD-9: 435.xx Carotid stenosis: (CD-9: 435.xx) Carotid s | ort study.* BMJ 2018;360:k119 of Heart Failure Hospitalization in gliflozin Comparative Effectiveness and it: |
| defined below: MI: ICD 9 Acute MI: 410.xx, Old MI: 412.xx Patrom, Elisabetta et al. "Cardiovascular outcomes assoning fillozin antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/bmj.k119 Patromo, Elisabetta et al. "Empagliflozin and the Risk of Routine Clinical Care: A First Analysis from the Empagliflozin and the Risk of Routine Clinical Care: A First Analysis | ort study.* BMJ 2018;360:k119 of Heart Failure Hospitalization in gliflozin Comparative Effectiveness and it: |
| Measured any time prior to Index hospitalization in any diagnosis position and Inpatient or outpatient care setting as defined below: (exception: TIA - Inpatient diagnosis only) Ischemic stroke: ICD-9: 433.x, 434. x Patorno, Elisabetta et al. *Cardiovascular outcomes ass non-giffician antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/pmj.k119 revascularization Measured any time prior to Index hospitalization in any diagnosis position and Inpatient or outpatient care setting as defined below: (exception: TIA - Inpatient diagnosis only) Ischemic stroke: ICD-9: 433.x, 434. x Patorno, Elisabetta et al. *Cardiovascular outcomes ass non-giffician antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/pmj.k119 revascularization Cardiovascular outcomes ass non-giffician antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/pmj.k119 Patorno, Elisabetta et al. *Cardiovascular outcomes ass non-giffician antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/pmj.k119 revascularization Cardiovascular outcomes ass non-giffician antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/pmj.k119 Patorno, Elisabetta et al. *Cardiovascular outcomes ass non-giffician antidiabetic drugs: population based cohor http:/ | |
| defined below: (exception: TIA - Inpetient diagnosis only) Ischemic stroke: ICD-9: 433.x, 434. x Patorno, Elisabetta et al. "Cardiovascular outcomes ass non-gliflozin antidiabetic drugs: population based cohor http://dx.doi.org/10.1136/mnj.k119 TIA (Inpetient diagnosis, any position): ICD-9: 435.xx TIA (Inpetient diagnosis, any position): ICD-9: 435.xx Carotid stenoels: Carotid stenoels: Return Ca | |
| Safety (EMPRISE) Study.* Circulation. 2019 Apr 8. doi: Coerbral reveasoularization: ICD-9 procedure code Carotid endarterectomy (38.12), Angioplasty/atherectomy of precerebral vessels (00.61) Carotid artery stenting (00.63). | gliflozin Comparative Effectiveness and |
| Measured 385 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting as defined below: Diabetes type 1: (e) Diabetes mellitus Diabetes mellitus (bC) 9: 250.x0 r 250.x2 Diabetes type 2: (CD) 9: 250.x0 or 250.x2 (CD) 9: 250.x0 or 250.x2 (CD) 9: 250.x0 r 250.x2 (CD) 9: 250. | ort study." BMJ 2018;360:k119 of Heart Failure Hospitalization in gliflozin Comparative Effectiveness and |
| Measured 365 days prior drug Initiation in any diagnosis position and inpatient or outpatient care setting as defined below. (f) Peripheral artery disease (f) Peripheral vascular disease (DD-9: 440.20 - 440.24, 440.29 - 440.32, 440.3, 440.4, 443.9 Patorno, Elisabetta et al. "Cardiovascular outcomes ass non-giffloria natidiabetic drugs: population based cohor hittp://dx.doi.org/10.1136/bmj.k112 Patorno, Elisabetta et al. "Englishetta et a | ort study." BMJ 2018;360:k119 of Heart Failure Hospitalization in gliflozin Comparative Effectiveness and |
| Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting as defined below: (g) Chronic renal dysfunction (g) Chronic renal dysfunction | ort study." BMJ 2018;360:k119 |
| Chronic Iddney disease: Patorno, Elisabetta et al. "Empagliflozin and the Risk of ICD-9: Septiment of Chronic Iddney disease: Patorno, Elisabetta et al. "Empagliflozin and the Risk of ICD-9: Septiment of Chronic Iddney disease: Septiment of Chronic Iddney Chronic Id | gliflozin Comparative Effectiveness and |
| UK B Persistent ST-segment elevation ≥1 mm (not known to be preexisting or due to a coexisting disorder) in ≥2 contiguous leads or new LB8B plus primary PCI planned. | |
| EXCLUSION CRITERIA | |
| Drug related | |

| 1 | 1. Contraindication to clopidogrel or other reason that study drug should not be administered (eg, hypersensitivity, moderate or severe liver disease, active bleeding or bleeding history, major surgery within 30 days) | Moderate/severe liver disease: Measured 190 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting ICD-9 diagnosis codes: 070.xx, 570.xx 573.xx 456.0x.456.2x, 576.8x, 782.4x, 789.5x ICD-9 procedure codes: 391.x, 42.91 Active bleeding or bleeding history: Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting Codes are in the sheet "Major Bleeding" Majory surgery (except cardiac surgeries): Measured 30 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting Major surgery selected from ICD-9 procedure codes range 40.x-84.x (procedures 35.x-39.x [cardiovascular procedures] are excluded) | Patorno, Elisabetta et al. *Cardiovascular outcomes associated with canagliflozin versus other non-giffozin antidiabetic drugs: population based cohort study.* BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. *Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study.* Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA118.039177 |
|---|---|---|---|
| 2 | 2. Oral anticoagulation therapy that cannot be stopped | N/A | |
| 3 | 3. Fibrinolytic therapy planned or within the previous 24 h | N/A | |
| 4 | 4. Concomitant oral or IV therapy with strong CYP3A inhibitors (ketoconazole, traconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin/rifampicin, phenytoin, carbamazepine) | Prescription claim for following CYP3A inhibitors, CYP3A substrates, or strong CYP3A inducers Measured 90 days prior to drug initiation Ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir Cyclosporine, quinidine Rifampin, rifampicin/rifampin, phenytoin, carbamazepine | |
| | Treat | tment Related | |
| 5 | 1. Index event is an acute complication of PCI | N/A | |
| 6 | 2. PCI after index event and before first study dose | N/A | |
| | | dical Related | |
| 8 | Increased risk of bradycardiac events Dialysis required | N/A Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpetient care setting Codes are in the sheet 'Dialysis' | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagilifozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (FMDRS) Stuty." (Circulation 2019 Apr & Roi: |
| 9 | 3. Known clinically important thrombocytopenia | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting Thrombocytopenia ICD-9: 287.3x, 287.4x, 287.5x | Salety LEMPRISE 1 Study. Cilculation, 2019 Aut 6, 000. |
| 10 | 4. Known clinically important anemia | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting Anemia (unspecified anemia including anemia of chronic illness, sideroblastic anemia) ICD-9: 285.x | |
| 11 | 5. Any other condition that may put the patient at risk or influence study results in the investigators' opinion (eg, cardiogenic shock, severe hemodynamic instability, active cancer) | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpetient care setting Cardiogenic shook: ICD-9: 785.51 Severe hemodynamic instability: ICD-9: 785.59 Other shock without mention of trauma 785.59 Septic shock, 785.50 shock, unspecified Active cancer: ICD-9: History of mallignant neoplasm 140.xx.208.xx (except 173.xx, non-melanoma skin cancer) | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-<br>gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119<br>http://dx.doi.org/10.136/pmj.k119<br>Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical<br>Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study."<br>Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | | General | |
| 12 | Participant in another investigational drug or device study within 30 days | N/A | |

| 13 | 2. Pregnancy or lactation | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting |
|---|---|---|
| | | Codes are in the sheet "Pregnancy" |
| 14 | 3. Any condition that increases the risk for noncompliance or being lost to follow-up | N/A |
| 15 | 4. Involvement in the planning or conduct of the study | N/A |
| 16 | 5. Previous enrollment or randomization in this study | N/A |

| Trial ID | pNDA10 |
|---|---|
| Trial Name (with web links) | <u>PLATO</u> |
| Trial Name (with pdf links) | <u>PLATO</u> |
| <u>NCT</u> | NCT00391872 |
| Trial category | Primary indication |
| Run-in period Description | |
| Run-in period | |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | Antiplatelets |
| RCT Category | 1a- Intended S with label change |
| Brand Name | <u>Brilinta</u> |
| Generic Name | ticagrelor |
| <u>Sponsor</u> | AstraZeneca |
| <u>Year</u> | 2011 |
| Measurable endpoint | Primary composite endpoint of cardiovascular death, non-fatal MI (excluding silent MI), or non-fatal stroke |
| <u>Exposure</u> | Ticagrelor |
| <u>Comparator</u> | Clopidogrel |
| <u>Population</u> | Patients admitted to the hospital with<br>an acute coronary syndrome, with or<br>without ST-segment elevation. 89%<br>patients on Beta-blocker, 76% ACE<br>inhibitors, 89% on statins |
| Trial finding | RR = 0.84 (95% CI 0.77–0.92) |
| <u>Notes</u> | |
| No. of Patients | 18,624 |
| Non-inferiority margin | - |
| Assay Sens. Outcome | |
| Assay Sens. Endpoint (from trial) | |

| Finding for potential Assay Sens. Outcome | |
|---|---|
| from trial- | |
| <u>Power</u> | 0.90 to detect a relative risk reduction of 13.5% in the rate of the primary end point |
| Blinding | Double-blinded |
| Statistical Method | |
| Approval indication | For the reduction of thrombotic events in patients with acute coronary syndrome |

#### Mortality-Dependent on data source.

1. All-cause mortality / inpatient mortality Identified using the vital status file-

#### Medicare

Identified using the discharge status codes-

#### Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)

- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

#### 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare at a later date. We will conduct secondary analyses using CV mortality at that time.

| Major bleeding control outcome: 1 inpatient (any position) | |
|---|---|
| Major bleedin | Major bleeding exclusion criteria: 1 inpatient (any position) or 2 outpatient diagnosis (separated by 7-365 days) |
| 562.02 | (ICD9) DIVERTICULOSIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.03 | (ICD9) DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.12 | (ICD9) DIVERTICULOSIS OF COLON WITH HEMORRHAGE |
| 562.13 | (ICD9) DIVERTICULITIS OF COLON WITH HEMORRHAGE |
| 568.81 | (ICD9) HEMOPERITONEUM (NONTRAUMATIC) |
| 569.3 | (ICD9) HEMORRHAGE OF RECTUM AND ANUS |
| 569.83 | (ICD9) PERFORATION OF INTESTINE |
| 569.85 | (ICD9) ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE |
| 569.86 | (ICD9) DIEULAFOY LESION (HEMORRHAGIC) OF INTESTINE |
| 578 | (ICD9) HEMATEMESIS |
| 578.9 | (ICD9) HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED |
| 423 | (ICD9) HEMOPERICARDIUM |
| 432 | (ICD9) NONTRAUMATIC EXTRADURAL HEMORRHAGE |
| 432.1 | (ICD9) SUBDURAL HEMORRHAGE |
| 432.9 | (ICD9) UNSPECIFIED INTRACRANIAL HEMORRHAGE |
| 459 | (ICD9) HEMORRHAGE UNSPECIFIED |
| 531 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE |
| 531 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.01 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.2 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.2 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.21 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 531.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE |
| 531.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.41 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.61 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE |
| 532 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.01 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 532.2 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |

| 532.2 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
|---|---|
| 532.21 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532.4 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE |
| 532.4 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.41 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 532.6 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 532.6 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 532.61 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 533 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| 533 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 533.01 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| 533.2 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 533.2 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 533.21 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 533.4 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| 533.4 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 533.41 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| 533.6 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 533.6 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 533.61 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.01 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 534.2 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.2 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.21 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.41 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 534.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.61 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 578.1 | (ICD9) BLOOD IN STOOL |
| 719.1 | (ICD9) HEMARTHROSIS |
| 719.1 | (ICD9) HEMARTHROSIS SITE UNSPECIFIED |

| 719.11 | (ICD9) HERARTHROSIS INVOLVING SHOULDER REGION |
|---|---|
| 719.12 | (ICD9) HEMARTHORSIS INVOLVING UPPER ARM |
| 719.13 | (ICD9) HEMARTHROSIS INVOLVING FOREARM |
| 719.14 | (ICD9) HEMARTHROSIS INVOLVING HAND |
| 719.15 | (ICD9) HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH |
| 719.16 | (ICD9) HEMARTHROSIS INVOLVING LOWER LEG |
| 719.17 | (ICD9) HEMARTHROSIS INVOLVING ANKLE AND FOOT |
| 719.18 | (ICD9) HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES |
| 719.19 | (ICD9) HEMARTHROSIS INVOLVING MULTIPLE SITES |
| 430 | (ICD9) SUBARACHNOID HEMORRHAGE |
| 431 | (ICD9) INTRACEREBRAL HEMORRHAGE |
| I31.2 | (ICD10) Hemopericardium, not elsewhere classified |
| 160.00 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified carotid siphon and bifurcation |
| 160.01 | (ICD10) Nontraumatic subarachnoid hemorrhage from right carotid siphon and bifurcation |
| 160.02 | (ICD10) Nontraumatic subarachnoid hemorrhage from left carotid siphon and bifurcation |
| 160.10 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified middle cerebral artery |
| 160.11 | (ICD10) Nontraumatic subarachnoid hemorrhage from right middle cerebral artery |
| 160.12 | (ICD10) Nontraumatic subarachnoid hemorrhage from left middle cerebral artery |
| 160.2 | (ICD10) Nontraumatic subarachnoid hemorrhage from anterior communicating artery |
| 160.30 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified posterior communicating artery |
| 160.31 | (ICD10) Nontraumatic subarachnoid hemorrhage from right posterior communicating artery |
| 160.32 | (ICD10) Nontraumatic subarachnoid hemorrhage from left posterior communicating artery |
| 160.4 | (ICD10) Nontraumatic subarachnoid hemorrhage from basilar artery |
| 160.50 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified vertebral artery |
| 160.51 | (ICD10) Nontraumatic subarachnoid hemorrhage from right vertebral artery |
| 160.52 | (ICD10) Nontraumatic subarachnoid hemorrhage from left vertebral artery |
| 160.6 | (ICD10) Nontraumatic subarachnoid hemorrhage from other intracranial arteries |
| 160.7 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified intracranial artery |
| 160.8 | (ICD10) Other nontraumatic subarachnoid hemorrhage |
| 160.9 | (ICD10) Nontraumatic subarachnoid hemorrhage, unspecified |
| I61.0 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, subcortical |
| I61.1 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, cortical |
| I61.2 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, unspecified |
| I61.3 | (ICD10) Nontraumatic intracerebral hemorrhage in brain stem |
| 161.4 | (ICD10) Nontraumatic intracerebral hemorrhage in cerebellum |

| 161.5 | (ICD10) Nontraumatic intracerebral hemorrhage, intraventricular |
|---|---|
| 161.6 | (ICD10) Nontraumatic intracerebral hemorrhage, multiple localized |
| 161.8 | (ICD10) Other nontraumatic intracerebral hemorrhage |
| 161.9 | (ICD10) Nontraumatic intracerebral hemorrhage, unspecified |
| 162.00 | (ICD10) Nontraumatic subdural hemorrhage, unspecified |
| 162.01 | (ICD10) Nontraumatic acute subdural hemorrhage |
| 162.02 | (ICD10) Nontraumatic subacute subdural hemorrhage |
| 162.03 | (ICD10) Nontraumatic chronic subdural hemorrhage |
| 162.1 | (ICD10) Nontraumatic extradural hemorrhage |
| 162.9 | (ICD10) Nontraumatic intracranial hemorrhage, unspecified |
| K25.0 | (ICD10) Acute gastric ulcer with hemorrhage |
| K25.2 | (ICD10) Acute gastric ulcer with both hemorrhage and perforation |
| K25.4 | (ICD10) Chronic or unspecified gastric ulcer with hemorrhage |
| K25.6 | (ICD10) Chronic or unspecified gastric ulcer with both hemorrhage and perforation |
| K26.0 | (ICD10) Acute duodenal ulcer with hemorrhage |
| K26.2 | (ICD10) Acute duodenal ulcer with both hemorrhage and perforation |
| K26.4 | (ICD10) Chronic or unspecified duodenal ulcer with hemorrhage |
| K26.6 | (ICD10) Chronic or unspecified duodenal ulcer with both hemorrhage and perforation |
| K27.0 | (ICD10) Acute peptic ulcer, site unspecified, with hemorrhage |
| K27.2 | (ICD10) Acute peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K27.4 | (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage |
| K27.6 | (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K28.0 | (ICD10) Acute gastrojejunal ulcer with hemorrhage |
| K28.2 | (ICD10) Acute gastrojejunal ulcer with both hemorrhage and perforation |
| K28.4 | (ICD10) Chronic or unspecified gastrojejunal ulcer with hemorrhage |
| K28.6 | (ICD10) Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation |
| K55.21 | (ICD10) Angiodysplasia of colon with hemorrhage |
| K56.60 | (ICD10) Unspecified intestinal obstruction |
| K57.01 | (ICD10) Diverticulitis of small intestine with perforation and abscess with bleeding |
| K57.11 | (ICD10) Diverticulosis of small intestine without perforation or abscess with bleeding |
| K57.13 | (ICD10) Diverticulitis of small intestine without perforation or abscess with bleeding |
| K57.21 | (ICD10) Diverticulitis of large intestine with perforation and abscess with bleeding |
| K57.31 | (ICD10) Diverticulosis of large intestine without perforation or abscess with bleeding |
| K57.33 | (ICD10) Diverticulitis of large intestine without perforation or abscess with bleeding |
| K57.41 | (ICD10) Diverticulitis of both small and large intestine with perforation and abscess with bleeding |

| K57.51 | (ICD10) Diverticulosis of both small and large intestine without perforation or abscess with bleeding |
|---|---|
| K57.53 | (ICD10) Diverticulitis of both small and large intestine without perforation or abscess with bleeding |
| K57.81 | (ICD10) Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding |
| K57.91 | (ICD10) Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding |
| K57.93 | (ICD10) Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding |
| K62.5 | (ICD10) Hemorrhage of anus and rectum |
| K63.1 | (ICD10) Perforation of intestine (nontraumatic) |
| K63.81 | (ICD10) Dieulafoy lesion of intestine |
| K66.1 | (ICD10) Hemoperitoneum |
| K92.0 | (ICD10) Hematemesis |
| K92.1 | (ICD10) Melena |
| K92.2 | (ICD10) Gastrointestinal hemorrhage, unspecified |
| M25.00 | (ICD10) Hemarthrosis, unspecified joint |
| M25.011 | (ICD10) Hemarthrosis, right shoulder |
| M25.012 | (ICD10) Hemarthrosis, left shoulder |
| M25.019 | (ICD10) Hemarthrosis, unspecified shoulder |
| M25.021 | (ICD10) Hemarthrosis, right elbow |
| M25.022 | (ICD10) Hemarthrosis, left elbow |
| M25.029 | (ICD10) Hemarthrosis, unspecified elbow |
| M25.031 | (ICD10) Hemarthrosis, right wrist |
| M25.032 | (ICD10) Hemarthrosis, left wrist |
| M25.039 | (ICD10) Hemarthrosis, unspecified wrist |
| M25.041 | (ICD10) Hemarthrosis, right hand |
| M25.042 | (ICD10) Hemarthrosis, left hand |
| M25.049 | (ICD10) Hemarthrosis, unspecified hand |
| M25.051 | (ICD10) Hemarthrosis, right hip |
| M25.052 | (ICD10) Hemarthrosis, left hip |
| M25.059 | (ICD10) Hemarthrosis, unspecified hip |
| M25.061 | (ICD10) Hemarthrosis, right knee |
| M25.062 | (ICD10) Hemarthrosis, left knee |
| M25.069 | (ICD10) Hemarthrosis, unspecified knee |
| M25.071 | (ICD10) Hemarthrosis, right ankle |
| M25.072 | (ICD10) Hemarthrosis, left ankle |
| M25.073 | (ICD10) Hemarthrosis, unspecified ankle |
| M25.074 | (ICD10) Hemarthrosis, right foot |

| M25.075 | (ICD10) Hemarthrosis, left foot |
|---|---|
| M25.076 | (ICD10) Hemarthrosis, unspecified foot |
| M25.08 | (ICD10) Hemarthrosis, other specified site |
| R58 | (ICD10) Hemorrhage, not elsewhere classified |
| R04 | (ICD10) Hemorrhage from respiratory passages |
| R04.0 | (ICD10) Epistaxis |
| R04.1 | (ICD10) Hemorrhage from throat |
| R04.2 | (ICD10) Hemoptysis |
| R04.8 | (ICD10) Hemorrhage from other sites in respiratory passages |
| R04.81 | (ICD10) Acute idiopathic pulmonary hemorrhage in infants |
| R04.89 | (ICD10) Hemorrhage from other sites in respiratory passages |
| R04.9 | (ICD10) Hemorrhage from respiratory passages, unspecified |
| R31 | (ICD10) Hematuria |
| R31.0 | (ICD10) Gross hematuria |
| R31.1 | (ICD10) Benign essential microscopic hematuria |
| R31.2 | (ICD10) Other microscopic hematuria |
| R31.21 | |
| R31.29 | |
| R31.9 | (ICD10) Hematuria, unspecified |
| 784.7 | (ICD9) EPISTAXIS |
| 784.8 | (ICD9) HEMORRHAGE FROM THROAT |
| 599.7 | (ICD9) HEMATURIA |
| 599.7 | (ICD9) HEMATURIA UNSPECIFIED |
| 599.71 | (ICD9) GROSS HEMATURIA |
| 599.72 | (ICD9) MICROSCOPIC HEMATURIA |
| 786.3 | (ICD9) HEMOPTYSIS |
| 786.3 | (ICD9) HEMOPTYSIS UNSPECIFIED |
| 786.31 | (ICD9) ACUTE IDIOPATHIC PULMONARY HEMORRHAGE IN INFANTS |
| 786.39 | (ICD9) OTHER HEMOPTYSIS |
| The occurren | ce of Inpatient with the following attributes: Procedure Code (Any Position) is any of: { "44.43", "43255", "0W3P8ZZ" } |
| 44.43 | (ICD9) ENDOSCOPIC CONTROL OF GASTRIC OR DUODENAL BLEEDING |
| 43255 | (HCPCS) Esophagogastroduodenoscopy, flexible, transoral; with control of bleeding, any method / Upper gastrointestinal endoscopy |
| 43233 | including esophagus, stomach, and either the duodenum and/or jejunum as appropriate; with control of bleeding, any method |
| 0W3P8ZZ | (ICD10) Control Bleeding in Gastrointestinal Tract, Via Natural or Artificial Opening Endoscopic |

#### **Dialysis codes**

ESRD, defined as 2 codes (either inpatient or outpatient), separated by at least 30 days

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

- ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512. Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

tor the adequacy or natition, etc. m2 or 5 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

## **Pregnancy** Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION

- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS


The c-statistics for the propensity score model, pre-matching was 0.744. The post-matching c-statistic was 0.538.

The c-statistics for the propensity score model, pre-matching was 0.722. The post-matching c-statistic was 0.528.



Figure 64: Post-matching propensity score overlap



Figure 64: Post-matching propensity score overlap

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| | | | | Un | matched | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opt | um | | Tru | ven | | POOL | LED | |
| Variable | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. |
| Number of patients | 34,251 | 7,078 | | 32,565 | 8,264 | | 66,816 | 15,342 | |
| Age | | | | | | | | | |
| mean (sd) | 70.43 (10.74) | 67.99 (10.81) | 0.23 | 66.08 (12.03) | 62.10 (10.28) | 0.36 | 68.31 (11.39) | 64.82 (10.53) | 0.32 |
| median [IQR] | 71.00 [64.00, 79.00] | 69.00 [61.00, 76.00] | 0.19 | 64.00 [59.00, 74.00] | 62.00 [56.00, 67.00] | 0.18 | 67.59 (11.39) | 65.23 (10.53) | 0.22 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 2,810 (8.2%) | 821 (11.6%) | -0.11 | 4,940 (15.2%) | 1,688 (20.4%) | -0.14 | 7,750 (11.6%) | 2,509 (16.4%) | -0.14 |
| 55 - 64; n (%) | 6,438 (18.8%) | 1,599 (22.6%) | -0.09 | 12,321 (37.8%) | 4,014 (48.6%) | -0.22 | 18,759 (28.1%) | 5,613 (36.6%) | -0.18 |
| 65 - 74; n (%) | 12,095 (35.3%) | 2,625 (37.1%) | -0.04 | 7,185 (22.1%) | 1,526 (18.5%) | 0.09 | 19,280 (28.9%) | 4,151 (27.1%) | 0.04 |
| >= 75; n (%) | 12,908 (37.7%) | 2,033 (28.7%) | 0.19 | 8,119 (24.9%) | 1,036 (12.5%) | 0.32 | 21,027 (31.5%) | 3,069 (20.0%) | 0.27 |
| Gender | | , , , | | | | | . , , | , , , | |
| Males; n (%) | 21,162 (61.8%) | 4,536 (64.1%) | -0.05 | 21,484 (66.0%) | 5,919 (71.6%) | -0.12 | 42,646 (63.8%) | 10,455 (68.1%) | -0.09 |
| Females; n (%) | 13,089 (38.2%) | 2,542 (35.9%) | 0.05 | 11,081 (34.0%) | 2,345 (28.4%) | 0.12 | 24,170 (36.2%) | 4,887 (31.9%) | 0.09 |
| Region | | , , | | | , , | | , , , | , , | |
| Northeast; n (%) | 4,152 (12.1%) | 804 (11.4%) | 0.02 | 6,331 (19.4%) | 1,562 (18.9%) | 0.01 | 10,483 (15.7%) | 2,366 (15.4%) | 0.01 |
| South; n (%) | 14,216 (41.5%) | 3,335 (47.1%) | -0.11 | 9,450 (29.0%) | 2,199 (26.6%) | 0.05 | 23,666 (35.4%) | 5,534 (36.1%) | -0.01 |
| Midwest; n (%) | 8,706 (25.4%) | 1,626 (23.0%) | 0.06 | 11,688 (35.9%) | 3,597 (43.5%) | -0.16 | 20,394 (30.5%) | 5,223 (34.0%) | -0.07 |
| West; n (%) | 7,177 (21.0%) | 1,313 (18.6%) | 0.06 | 4,769 (14.6%) | 868 (10.5%) | 0.12 | 11,946 (17.9%) | 2,181 (14.2%) | 0.10 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 327 (1.0%) | 38 (0.5%) | 0.06 | 327 (0.5%) | 38 (0.2%) | 0.05 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 34,251 (100.0%) | 7,078 (100.0%) | #DIV/0! | 32,565 (100.0%) | 8,264 (100.0%) | #DIV/0! | 66,816 (100.0%) | 15,342 (100.0%) | #DIV/0! |
| Acute MI; n (%) | 31,334 (91.5%) | 6,496 (91.8%) | -0.01 | 31,063 (95.4%) | 7,831 (94.8%) | 0.03 | 62397 (93.4%) | 14327 (93.4%) | 0.00 |
| ACS/unstable angina; n (%) | 14,701 (42.9%) | 2,968 (41.9%) | 0.02 | 11,618 (35.7%) | 2,960 (35.8%) | 0.00 | 26319 (39.4%) | 5928 (38.6%) | 0.02 |
| Old MI; n (%) | 5,865 (17.1%) | 1,180 (16.7%) | 0.01 | 3,170 (9.7%) | 720 (8.7%) | 0.03 | 9035 (13.5%) | 1900 (12.4%) | 0.03 |
| Stable angina; n (%) | 8,209 (24.0%) | 1,781 (25.2%) | -0.03 | 4,741 (14.6%) | 1,380 (16.7%) | -0.06 | 12,950 (19.4%) | 3,161 (20.6%) | -0.03 |
| Coronary atherosclerosis and other forms | 32,438 (94.7%) | 6,799 (96.1%) | -0.07 | 29,092 (89.3%) | 7,630 (92.3%) | -0.10 | 61,530 (92.1%) | 14,429 (94.0%) | -0.07 |
| of chronic ischemic heart disease; n (%) | | | | | | | | | |
| Other atherosclerosis with ICD10; n (%) | 634 (1.9%) | 84 (1.2%) | 0.06 | 632 (1.9%) | 89 (1.1%) | 0.07 | 1266 (1.9%) | 173 (1.1%) | 0.07 |
| Previous cardiac procedure (CABG or PTCA | 25,241 (73.7%) | 6,564 (92.7%) | -0.53 | 24,229 (74.4%) | 7,510 (90.9%) | -0.45 | 49470 (74.0%) | 14074 (91.7%) | -0.48 |
| or Stent); n (%) | | | | | | | | | |
| History of CABG or PTCA; n (%) | 12,033 (35.1%) | 2,459 (34.7%) | 0.01 | 5,974 (18.3%) | 1,489 (18.0%) | 0.01 | 18,007 (27.0%) | 3,948 (25.7%) | 0.03 |
| Any stroke; n (%) | 4,738 (13.8%) | 622 (8.8%) | 0.16 | 3,006 (9.2%) | 433 (5.2%) | 0.16 | 7,744 (11.6%) | 1,055 (6.9%) | 0.16 |
| Ischemic stroke (w and w/o mention of | 4,698 (13.7%) | 619 (8.7%) | 0.16 | 2,999 (9.2%) | 433 (5.2%) | 0.16 | 7,697 (11.5%) | 1,052 (6.9%) | 0.16 |
| cerebral infarction); n (%) | | | | | | | | | |
| Hemorrhagic stroke; n (%) | 77 (0.2%) | 8 (0.1%) | 0.03 | 9 (0.0%) | 0 (0.0%) | #DIV/0! | 86 (0.1%) | 8 (0.1%) | 0.00 |
| TIA; n (%) | 829 (2.4%) | 128 (1.8%) | 0.04 | 595 (1.8%) | 81 (1.0%) | 0.07 | 1424 (2.1%) | 209 (1.4%) | 0.05 |
| Other cerebrovascular disease; n (%) | 1,088 (3.2%) | 153 (2.2%) | 0.06 | 565 (1.7%) | 77 (0.9%) | 0.07 | 1653 (2.5%) | 230 (1.5%) | 0.07 |
| Late effects of cerebrovascular disease; n (%) | 888 (2.6%) | 139 (2.0%) | 0.04 | 337 (1.0%) | 54 (0.7%) | 0.03 | 1225 (1.8%) | 193 (1.3%) | 0.04 |
| Cerebrovascular procedure; n (%) | 71 (0.2%) | 8 (0.1%) | 0.03 | 49 (0.2%) | 4 (0.0%) | 0.06 | 120 (0.2%) | 12 (0.1%) | 0.03 |
| Heart failure (CHF); n (%) | 10,773 (31.5%) | 1,796 (25.4%) | 0.14 | 7,073 (21.7%) | 1,226 (14.8%) | 0.18 | 17,846 (26.7%) | 3,022 (19.7%) | 0.17 |
| Peripheral Vascular Disease (PVD) or PVD | 4,708 (13.7%) | 884 (12.5%) | 0.04 | 2,400 (7.4%) | 428 (5.2%) | 0.09 | 7,108 (10.6%) | 1,312 (8.6%) | 0.07 |
| Surgery; n (%) | 1,700 (13.770) | 304 (12.370) | 0.04 | 2,500 (7.570) | 120 (3.270) | 0.03 | ,,100 (10.0/0) | 1,312 (0.070) | 0.57 |
| Atrial fibrillation; n (%) | 6,613 (19.3%) | 833 (11.8%) | 0.21 | 4,094 (12.6%) | 587 (7.1%) | 0.19 | 10,707 (16.0%) | 1,420 (9.3%) | 0.20 |
| Other cardiac dysrhythmia; n (%) | 13,828 (40.4%) | 2,626 (37.1%) | 0.07 | 9,711 (29.8%) | 2,478 (30.0%) | 0.00 | 23,539 (35.2%) | 5,104 (33.3%) | 0.04 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Cardiac conduction disorders; n (%) | 5,955 (17.4%) | 1,074 (15.2%) | 0.06 | 3,681 (11.3%) | 813 (9.8%) | 0.05 | 9636 (14.4%) | 1887 (12.3%) | 0.06 |
|---|---|---|---|---|---|---|---|---|---|
| Other CVD; n (%) | 14,535 (42.4%) | 2,682 (37.9%) | 0.09 | 9,954 (30.6%) | 2,194 (26.5%) | 0.09 | 24,489 (36.7%) | 4,876 (31.8%) | 0.10 |
| Diabetes-related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 1,230 (3.6%) | 273 (3.9%) | -0.02 | 633 (1.9%) | 154 (1.9%) | 0.00 | 1,863 (2.8%) | 0,427 (2.8%) | 0.00 |
| Diabetes with other ophthalmic | 105 (0.3%) | 36 (0.5%) | -0.03 | 422 (1.3%) | 75 (0.9%) | 0.04 | 0,527 (0.8%) | 0,111 (0.7%) | 0.01 |
| manifestations; n (%) | | | | | | | | | |
| Retinal detachment, vitreous hemorrhage, | 147 (0.4%) | 17 (0.2%) | 0.04 | 74 (0.2%) | 24 (0.3%) | -0.02 | 221 (0.3%) | 41 (0.3%) | 0.00 |
| vitrectomy; n (%) | | | | | | | | | |
| Retinal laser coagulation therapy; n (%) | 127 (0.4%) | 31 (0.4%) | 0.00 | 113 (0.3%) | 36 (0.4%) | -0.02 | 240 (0.4%) | 67 (0.4%) | 0.00 |
| Occurrence of Diabetic Neuropathy; n (%) | 3,634 (10.6%) | 902 (12.7%) | -0.07 | 1,671 (5.1%) | 430 (5.2%) | 0.00 | 5,305 (7.9%) | 1,332 (8.7%) | -0.03 |
| Occurrence of diabetic nephropathy with ICD10 ; n (%) | 3,723 (10.9%) | 859 (12.1%) | -0.04 | 1,057 (3.2%) | 259 (3.1%) | 0.01 | 4,780 (7.2%) | 1,118 (7.3%) | 0.00 |
| Hypoglycemia; n (%) | 529 (1.5%) | 40 (0.6%) | 0.09 | 598 (1.8%) | 96 (1.2%) | 0.05 | 1,127 (1.7%) | 0,136 (0.9%) | 0.07 |
| Hyperglycemia; n (%) | 2,999 (8.8%) | 639 (9.0%) | -0.01 | 1,715 (5.3%) | 497 (6.0%) | -0.03 | 4,714 (7.1%) | 1,136 (7.4%) | -0.01 |
| Disorders of fluid electrolyte and acid-base | 7,300 (21.3%) | 1,404 (19.8%) | 0.04 | 3,644 (11.2%) | 793 (9.6%) | 0.05 | 10,944 (16.4%) | 2,197 (14.3%) | 0.06 |
| balance; n (%) | | | | | | | | | |
| Diabetic ketoacidosis; n (%) | 217 (0.6%) | 40 (0.6%) | 0.00 | 189 (0.6%) | 49 (0.6%) | 0.00 | 406 (0.6%) | 89 (0.6%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK); n (%) | 154 (0.4%) | 34 (0.5%) | -0.01 | 56 (0.2%) | 13 (0.2%) | 0.00 | 210 (0.3%) | 47 (0.3%) | 0.00 |
| Diabetes with peripheral circulatory disorders with ICD-10; n (%) | 1,964 (5.7%) | 470 (6.6%) | -0.04 | 652 (2.0%) | 145 (1.8%) | 0.01 | 2,616 (3.9%) | 0,615 (4.0%) | -0.01 |
| Diabetic Foot; n (%) | 655 (1.9%) | 104 (1.5%) | 0.03 | 412 (1.3%) | 74 (0.9%) | 0.04 | 1067 (1.6%) | 178 (1.2%) | 0.03 |
| Gangrene ; n (%) | 80 (0.2%) | 9 (0.1%) | 0.03 | 38 (0.1%) | 4 (0.0%) | 0.04 | 118 (0.2%) | 13 (0.1%) | 0.03 |
| Lower extremity amputation; n (%) | 258 (0.8%) | 45 (0.6%) | 0.02 | 70 (0.2%) | 17 (0.2%) | 0.00 | 328 (0.5%) | 62 (0.4%) | 0.01 |
| Osteomyelitis; n (%) | 144 (0.4%) | 30 (0.4%) | 0.00 | 88 (0.3%) | 23 (0.3%) | 0.00 | 232 (0.3%) | 53 (0.3%) | 0.00 |
| Skin infections ; n (%) | 1,789 (5.2%) | 325 (4.6%) | 0.03 | 1,272 (3.9%) | 294 (3.6%) | 0.02 | 3,061 (4.6%) | 0,619 (4.0%) | 0.03 |
| Erectile dysfunction; n (%) | 895 (2.6%) | 230 (3.2%) | -0.04 | 634 (1.9%) | 197 (2.4%) | -0.03 | 1,529 (2.3%) | 0,427 (2.8%) | -0.03 |
| Diabetes with unspecified complication; n (%) | 1,412 (4.1%) | 409 (5.8%) | -0.08 | 758 (2.3%) | 278 (3.4%) | -0.07 | 2,170 (3.2%) | 0,687 (4.5%) | -0.07 |
| Diabetes mellitus without mention of complications; n (%) | 15,987 (46.7%) | 3,767 (53.2%) | -0.13 | 13,028 (40.0%) | 3,410 (41.3%) | -0.03 | 29,015 (43.4%) | 7,177 (46.8%) | -0.07 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 29,781 (86.9%) | 6,140 (86.7%) | 0.01 | 24,582 (75.5%) | 6,362 (77.0%) | -0.04 | 54,363 (81.4%) | 12,502 (81.5%) | 0.00 |
| Hyperlipidemia ; n (%) | 28,216 (82.4%) | 5,950 (84.1%) | -0.05 | 21,320 (65.5%) | 5,887 (71.2%) | -0.12 | 49,536 (74.1%) | 11,837 (77.2%) | -0.07 |
| Edema; n (%) | 2,760 (8.1%) | 463 (6.5%) | 0.06 | 1,232 (3.8%) | 240 (2.9%) | 0.05 | 3,992 (6.0%) | 0,703 (4.6%) | 0.06 |
| Renal Dysfunction (non-diabetic); n (%) | 10,997 (32.1%) | 2,153 (30.4%) | 0.04 | 5,565 (17.1%) | 1,067 (12.9%) | 0.12 | 16,562 (24.8%) | 3,220 (21.0%) | 0.09 |
| Occurrence of acute renal disease; n (%) | 5,186 (15.1%) | 967 (13.7%) | 0.04 | 2,495 (7.7%) | 464 (5.6%) | 0.08 | 7681 (11.5%) | 1431 (9.3%) | 0.07 |
| Occurrence of chronic renal insufficiency; n (%) | 8,114 (23.7%) | 1,581 (22.3%) | 0.03 | 3,144 (9.7%) | 565 (6.8%) | 0.11 | 11,258 (16.8%) | 2,146 (14.0%) | 0.08 |
| Chronic kidney disease ; n (%) | 7,938 (23.2%) | 1,541 (21.8%) | 0.03 | 3,053 (9.4%) | 537 (6.5%) | 0.11 | 10,991 (16.4%) | 2,078 (13.5%) | 0.08 |
| CKD Stage 3-4; n (%) | 5,647 (16.5%) | 1,103 (15.6%) | 0.02 | 1,963 (6.0%) | 358 (4.3%) | 0.08 | 7,610 (11.4%) | 1,461 (9.5%) | 0.06 |
| Occurrence of hypertensive nephropathy; n (%) | 6,374 (18.6%) | 1,237 (17.5%) | 0.03 | 2,370 (7.3%) | 390 (4.7%) | 0.11 | 8744 (13.1%) | 1627 (10.6%) | 0.08 |
| Occurrence of miscellaneous renal insufficiency; n (%) | 3,321 (9.7%) | 626 (8.8%) | 0.03 | 1,555 (4.8%) | 344 (4.2%) | 0.03 | 4,876 (7.3%) | 0,970 (6.3%) | 0.04 |
| Glaucoma or cataracts ; n (%) | 5,574 (16.3%) | 1,117 (15.8%) | 0.01 | 4,135 (12.7%) | 898 (10.9%) | 0.06 | 9,709 (14.5%) | 2,015 (13.1%) | 0.04 |
| Cellulitis or abscess of toe; n (%) | 474 (1.4%) | 87 (1.2%) | 0.02 | 184 (0.6%) | 56 (0.7%) | -0.01 | 658 (1.0%) | 143 (0.9%) | 0.01 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Foot ulcer; n (%) | 661 (1.9%) | 107 (1.5%) | 0.03 | 415 (1.3%) | 72 (0.9%) | 0.04 | 1076 (1.6%) | 179 (1.2%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Bladder stones; n (%) | 78 (0.2%) | 9 (0.1%) | 0.03 | 30 (0.1%) | 9 (0.1%) | 0.00 | 108 (0.2%) | 18 (0.1%) | 0.03 |
| Kidney stones; n (%) | 961 (2.8%) | 220 (3.1%) | -0.02 | 521 (1.6%) | 148 (1.8%) | -0.02 | 1,482 (2.2%) | 0,368 (2.4%) | -0.01 |
| Urinary tract infections (UTIs); n (%) | 3,662 (10.7%) | 627 (8.9%) | 0.06 | 1,767 (5.4%) | 308 (3.7%) | 0.08 | 5,429 (8.1%) | 0,935 (6.1%) | 0.08 |
| Dipstick urinalysis; n (%) | 9,527 (27.8%) | 1,976 (27.9%) | 0.00 | 6,727 (20.7%) | 1,658 (20.1%) | 0.01 | 16,254 (24.3%) | 3,634 (23.7%) | 0.01 |
| Non-dipstick urinalysis; n (%) | 5,596 (16.3%) | 1,400 (19.8%) | -0.09 | 3,038 (9.3%) | 864 (10.5%) | -0.04 | 8,634 (12.9%) | 2,264 (14.8%) | -0.06 |
| Urine function test; n (%) | 867 (2.5%) | 162 (2.3%) | 0.01 | 619 (1.9%) | 156 (1.9%) | 0.00 | 1,486 (2.2%) | 0,318 (2.1%) | 0.01 |
| Cytology; n (%) | 410 (1.2%) | 84 (1.2%) | 0.00 | 179 (0.5%) | 37 (0.4%) | 0.01 | 589 (0.9%) | 121 (0.8%) | 0.01 |
| Cystos; n (%) | 597 (1.7%) | 106 (1.5%) | 0.02 | 233 (0.7%) | 43 (0.5%) | 0.03 | 830 (1.2%) | 149 (1.0%) | 0.02 |
| Other Covariates | | | | | | | | | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0,000 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 7,052 (20.6%) | 1,438 (20.3%) | 0.01 | 4,240 (13.0%) | 988 (12.0%) | 0.03 | 11,292 (16.9%) | 2,426 (15.8%) | 0.03 |
| Other arthritis, arthropathies and | 13,667 (39.9%) | 2,723 (38.5%) | 0.03 | 10,227 (31.4%) | 2,471 (29.9%) | 0.03 | 23,894 (35.8%) | 5,194 (33.9%) | 0.04 |
| musculoskeletal pain; n (%) | | | | | | | | | |
| Dorsopathies; n (%) | 9,026 (26.4%) | 1,846 (26.1%) | 0.01 | 6,582 (20.2%) | 1,668 (20.2%) | 0.00 | 15,608 (23.4%) | 3,514 (22.9%) | 0.01 |
| Fractures; n (%) | 1,178 (3.4%) | 202 (2.9%) | 0.03 | 737 (2.3%) | 153 (1.9%) | 0.03 | 1,915 (2.9%) | 0,355 (2.3%) | 0.04 |
| Falls; n (%) | 1,563 (4.6%) | 267 (3.8%) | 0.04 | 370 (1.1%) | 70 (0.8%) | 0.03 | 1933 (2.9%) | 337 (2.2%) | 0.04 |
| Osteoporosis; n (%) | 2,018 (5.9%) | 328 (4.6%) | 0.06 | 1,062 (3.3%) | 164 (2.0%) | 0.08 | 3,080 (4.6%) | 0,492 (3.2%) | 0.07 |
| Hyperthyroidism; n (%) | 239 (0.7%) | 47 (0.7%) | 0.00 | 134 (0.4%) | 29 (0.4%) | 0.00 | 373 (0.6%) | 76 (0.5%) | 0.01 |
| Hypothyroidism ; n (%) | 5,722 (16.7%) | 1,155 (16.3%) | 0.01 | 3,460 (10.6%) | 809 (9.8%) | 0.03 | 9,182 (13.7%) | 1,964 (12.8%) | 0.03 |
| Other disorders of thyroid gland; n (%) | 1,009 (2.9%) | 246 (3.5%) | -0.03 | 684 (2.1%) | 176 (2.1%) | 0.00 | 1,693 (2.5%) | 0,422 (2.8%) | -0.02 |
| Depression; n (%) | 4,071 (11.9%) | 818 (11.6%) | 0.01 | 2,357 (7.2%) | 499 (6.0%) | 0.05 | 6,428 (9.6%) | 1,317 (8.6%) | 0.03 |
| Anxiety; n (%) | 4,488 (13.1%) | 986 (13.9%) | -0.02 | 2,477 (7.6%) | 682 (8.3%) | -0.03 | 6,965 (10.4%) | 1,668 (10.9%) | -0.02 |
| SleepDisorder; n (%) | 2,233 (6.5%) | 322 (4.5%) | 0.09 | 2,524 (7.8%) | 461 (5.6%) | 0.09 | 4,757 (7.1%) | 0,783 (5.1%) | 0.08 |
| Dementia; n (%) | 2,499 (7.3%) | 310 (4.4%) | 0.12 | 1,211 (3.7%) | 120 (1.5%) | 0.14 | 3710 (5.6%) | 430 (2.8%) | 0.14 |
| Delirium; n (%) | 1,054 (3.1%) | 159 (2.2%) | 0.06 | 505 (1.6%) | 73 (0.9%) | 0.06 | 1559 (2.3%) | 232 (1.5%) | 0.06 |
| Psychosis; n (%) | 499 (1.5%) | 64 (0.9%) | 0.06 | 252 (0.8%) | 37 (0.4%) | 0.05 | 751 (1.1%) | 101 (0.7%) | 0.04 |
| Obesity; n (%) | 7,787 (22.7%) | 1,982 (28.0%) | -0.12 | 5,186 (15.9%) | 1,595 (19.3%) | -0.09 | 12,973 (19.4%) | 3,577 (23.3%) | -0.10 |
| Overweight; n (%) | 1,859 (5.4%) | 522 (7.4%) | -0.08 | 666 (2.0%) | 250 (3.0%) | -0.06 | 2,525 (3.8%) | 0,772 (5.0%) | -0.06 |
| Smoking; n (%) | 14,843 (43.3%) | 3,268 (46.2%) | -0.06 | 8,437 (25.9%) | 2,368 (28.7%) | -0.06 | 23,280 (34.8%) | 5,636 (36.7%) | -0.04 |
| Alcohol abuse or dependence; n (%) | 838 (2.4%) | 166 (2.3%) | 0.01 | 556 (1.7%) | 122 (1.5%) | 0.02 | 1394 (2.1%) | 288 (1.9%) | 0.01 |
| Drug abuse or dependence; n (%) | 883 (2.6%) | 198 (2.8%) | -0.01 | 380 (1.2%) | 105 (1.3%) | -0.01 | 1263 (1.9%) | 303 (2.0%) | -0.01 |
| COPD; n (%) | 7,224 (21.1%) | 1,272 (18.0%) | 0.08 | 4,050 (12.4%) | 686 (8.3%) | 0.13 | 11,274 (16.9%) | 1,958 (12.8%) | 0.12 |
| Asthma; n (%) | 2,569 (7.5%) | 519 (7.3%) | 0.01 | 1,779 (5.5%) | 406 (4.9%) | 0.03 | 4,348 (6.5%) | 0,925 (6.0%) | 0.02 |
| Obstructive sleep apnea; n (%) | 3,355 (9.8%) | 841 (11.9%) | -0.07 | 2,502 (7.7%) | 709 (8.6%) | -0.03 | 5,857 (8.8%) | 1,550 (10.1%) | -0.04 |
| Pneumonia; n (%) | 2,786 (8.1%) | 472 (6.7%) | 0.05 | 1,673 (5.1%) | 234 (2.8%) | 0.12 | 4,459 (6.7%) | 0,706 (4.6%) | 0.09 |
| Imaging; n (%) | 835 (2.4%) | 216 (3.1%) | -0.04 | 4,135 (12.7%) | 113 (1.4%) | 0.45 | 1227 (1.8%) | 329 (2.1%) | -0.02 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 18,168 (53.0%) | 3,711 (52.4%) | 0.01 | 18,195 (55.9%) | 4,684 (56.7%) | -0.02 | 36,363 (54.4%) | 8,395 (54.7%) | -0.01 |
| Use of ARBs; n (%) | 7,250 (21.2%) | 1,772 (25.0%) | -0.09 | 6,486 (19.9%) | 1,768 (21.4%) | -0.04 | 13,736 (20.6%) | 3,540 (23.1%) | -0.06 |
| Use of Loop Diuretics - ; n (%) | 7,459 (21.8%) | 1,065 (15.0%) | 0.18 | 5,065 (15.6%) | 615 (7.4%) | 0.26 | 12,524 (18.7%) | 1,680 (11.0%) | 0.22 |
| Use of other diuretics-; n (%) | 1,797 (5.2%) | 346 (4.9%) | 0.01 | 1,516 (4.7%) | 346 (4.2%) | 0.02 | 3,313 (5.0%) | 0,692 (4.5%) | 0.02 |
| Use of nitrates-; n (%) | 15,391 (44.9%) | 3,062 (43.3%) | 0.03 | 15,249 (46.8%) | 3,618 (43.8%) | 0.06 | 30,640 (45.9%) | 6,680 (43.5%) | 0.05 |
| Use of other hypertension drugs; n (%) | 3,062 (8.9%) | 529 (7.5%) | 0.05 | 2,130 (6.5%) | 372 (4.5%) | 0.09 | 5,192 (7.8%) | 0,901 (5.9%) | 0.08 |
| Use of digoxin-; n (%) | 772 (2.3%) | 72 (1.0%) | 0.10 | 703 (2.2%) | 64 (0.8%) | 0.12 | 1475 (2.2%) | 136 (0.9%) | 0.11 |
| Use of Anti-arrhythmics; n (%) | 1,992 (5.8%) | 204 (2.9%) | 0.14 | 1,521 (4.7%) | 157 (1.9%) | 0.16 | 3513 (5.3%) | 361 (2.4%) | 0.15 |
| Use of COPD/asthma meds-; n (%) | 5,251 (15.3%) | 1,080 (15.3%) | 0.00 | 4,557 (14.0%) | 990 (12.0%) | 0.06 | 9,808 (14.7%) | 2,070 (13.5%) | 0.03 |
| Use of statins; n (%) | 30,368 (88.7%) | 6,399 (90.4%) | -0.06 | 29,034 (89.2%) | 7,587 (91.8%) | -0.09 | 59,402 (88.9%) | 13,986 (91.2%) | -0.08 |
| 1 | • ' | . , | | · · | . , | | . , | • • | |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Use of other lipid-lowering drugs; n (%) | 2,561 (7.5%) | 545 (7.7%) | -0.01 | 2,974 (9.1%) | 754 (9.1%) | 0.00 | 5,535 (8.3%) | 1,299 (8.5%) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Use of oral anticoagulants (Dabigatran, | 3,350 (9.8%) | 353 (5.0%) | 0.18 | 2,682 (8.2%) | 321 (3.9%) | 0.18 | 6,032 (9.0%) | 0,674 (4.4%) | 0.18 |
| Rivaroxaban, Apixaban, Warfarin); n (%) | | | | | | | | | |
| Use of heparin and other low-molecular | 384 (1.1%) | 41 (0.6%) | 0.05 | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 387 (0.6%) | 41 (0.3%) | 0.04 |
| weight heparins; n (%) | | | | | | | | | |
| Use of NSAIDs; n (%) | 4,499 (13.1%) | 1,078 (15.2%) | -0.06 | 4,253 (13.1%) | 1,298 (15.7%) | -0.07 | 8,752 (13.1%) | 2,376 (15.5%) | -0.07 |
| Use of oral corticosteroids; n (%) | 6,426 (18.8%) | 1,272 (18.0%) | 0.02 | 5,175 (15.9%) | 1,257 (15.2%) | 0.02 | 11,601 (17.4%) | 2,529 (16.5%) | 0.02 |
| Use of bisphosphonate (); n (%) | 783 (2.3%) | 114 (1.6%) | 0.05 | 554 (1.7%) | 67 (0.8%) | 0.08 | 1337 (2.0%) | 181 (1.2%) | 0.06 |
| Use of opioids-; n (%) | 10,025 (29.3%) | 1,741 (24.6%) | 0.11 | 8,554 (26.3%) | 1,758 (21.3%) | 0.12 | 18,579 (27.8%) | 3,499 (22.8%) | 0.12 |
| Use of antidepressants; n (%) | 6,765 (19.8%) | 1,410 (19.9%) | 0.00 | 5,528 (17.0%) | 1,302 (15.8%) | 0.03 | 12,293 (18.4%) | 2,712 (17.7%) | 0.02 |
| Use of antipsychotics; n (%) | 665 (1.9%) | 145 (2.0%) | -0.01 | 418 (1.3%) | 74 (0.9%) | 0.04 | 1,083 (1.6%) | 0,219 (1.4%) | 0.02 |
| Use of anticonvulsants; n (%) | 4,151 (12.1%) | 968 (13.7%) | -0.05 | 2,669 (8.2%) | 652 (7.9%) | 0.01 | 6,820 (10.2%) | 1,620 (10.6%) | -0.01 |
| Use of lithium- ; n (%) | 41 (0.1%) | 11 (0.2%) | -0.03 | 35 (0.1%) | 6 (0.1%) | 0.00 | 76 (0.1%) | 17 (0.1%) | 0.00 |
| Use of Benzos- ; n (%) | 3,677 (10.7%) | 793 (11.2%) | -0.02 | 3,590 (11.0%) | 852 (10.3%) | 0.02 | 7,267 (10.9%) | 1,645 (10.7%) | 0.01 |
| Use of anxiolytics/hypnotics-; n (%) | 1,644 (4.8%) | 316 (4.5%) | 0.01 | 1,835 (5.6%) | 441 (5.3%) | 0.01 | 3,479 (5.2%) | 0,757 (4.9%) | 0.01 |
| Use of dementia meds-; n (%) | 924 (2.7%) | 123 (1.7%) | 0.07 | 648 (2.0%) | 61 (0.7%) | 0.11 | 1572 (2.4%) | 184 (1.2%) | 0.09 |
| Use of antiparkinsonian meds-; n (%) | 805 (2.4%) | 159 (2.2%) | 0.01 | 576 (1.8%) | 117 (1.4%) | 0.03 | 1,381 (2.1%) | 0,276 (1.8%) | 0.02 |
| Entresto (sacubitril/valsartan); n (%) | 58 (0.2%) | 16 (0.2%) | 0.00 | 9 (0.0%) | 3 (0.0%) | #DIV/0! | 67 (0.1%) | 19 (0.1%) | 0.00 |
| Labs | | | | | | | 0 | 0 | |
| Lab values- HbA1c (%) ; n (%) | 5,587 (16.3%) | 1,481 (20.9%) | -0.12 | 570 (1.8%) | 128 (1.5%) | 0.02 | 6,157 (9.2%) | 1,609 (10.5%) | -0.04 |
| Lab values- HbA1c (%) (within 3 months); n | 3,598 (10.5%) | 955 (13.5%) | -0.09 | 395 (1.2%) | 93 (1.1%) | 0.01 | 3,993 (6.0%) | 1,048 (6.8%) | -0.03 |
| (%) | , , | , , | | , , | | | , , | . , , | |
| Lab values- HbA1c (%) (within 6 months) ; n<br>(%) | 5,587 (16.3%) | 1,481 (20.9%) | -0.12 | 570 (1.8%) | 128 (1.5%) | 0.02 | 6,157 (9.2%) | 1,609 (10.5%) | -0.04 |
| Lab values- BNP; n (%) | 376 (1.1%) | 75 (1.1%) | 0.00 | 44 (0.1%) | 2 (0.0%) | 0.04 | 420 (0.6%) | 77 (0.5%) | 0.01 |
| Lab values- BNP (within 3 months); n (%) | 290 (0.8%) | 54 (0.8%) | 0.00 | 39 (0.1%) | 1 (0.0%) | 0.04 | 329 (0.5%) | 55 (0.4%) | 0.01 |
| Lab values- BNP (within 6 months); n (%) | 376 (1.1%) | 75 (1.1%) | 0.00 | 44 (0.1%) | 2 (0.0%) | 0.04 | 420 (0.6%) | 77 (0.5%) | 0.01 |
| Lab values- BUN (mg/dl); n (%) | 8,281 (24.2%) | 2,014 (28.5%) | -0.10 | 452 (1.4%) | 141 (1.7%) | -0.02 | 8,733 (13.1%) | 2,155 (14.0%) | -0.03 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 5,410 (15.8%) | 1,335 (18.9%) | -0.08 | 310 (1.0%) | 88 (1.1%) | -0.01 | 5,720 (8.6%) | 1,423 (9.3%) | -0.02 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 8,281 (24.2%) | 2,014 (28.5%) | -0.10 | 452 (1.4%) | 141 (1.7%) | -0.02 | 8,733 (13.1%) | 2,155 (14.0%) | -0.03 |
| Lab values- Creatinine (mg/dl); n (%) | 8,490 (24.8%) | 2,074 (29.3%) | -0.10 | 475 (1.5%) | 152 (1.8%) | -0.02 | 8,965 (13.4%) | 2,226 (14.5%) | -0.03 |
| Lab values- Creatinine (mg/dl) (within 3 | 5,559 (16.2%) | 1,382 (19.5%) | -0.09 | 322 (1.0%) | 98 (1.2%) | -0.02 | 5,881 (8.8%) | 1,480 (9.6%) | -0.03 |
| months); n (%) | | | | , , | , , | | , , , | | |
| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 8,490 (24.8%) | 2,074 (29.3%) | -0.10 | 475 (1.5%) | 152 (1.8%) | -0.02 | 8,965 (13.4%) | 2,226 (14.5%) | -0.03 |
| Lab values- HDL level (mg/dl); n (%) | 6,291 (18.4%) | 1,583 (22.4%) | -0.10 | 482 (1.5%) | 121 (1.5%) | 0.00 | 6,773 (10.1%) | 1,704 (11.1%) | -0.03 |
| Lab values- HDL level (mg/dl) (within 3 | 3,750 (10.9%) | 955 (13.5%) | -0.08 | 304 (0.9%) | 71 (0.9%) | 0.00 | 4,054 (6.1%) | 1,026 (6.7%) | -0.02 |
| months); n (%) | , , | | | | | | | | |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 6,291 (18.4%) | 1,583 (22.4%) | -0.10 | 482 (1.5%) | 121 (1.5%) | 0.00 | 6,773 (10.1%) | 1,704 (11.1%) | -0.03 |
| Lab values- LDL level (mg/dl); n (%) | 6,448 (18.8%) | 1,656 (23.4%) | -0.11 | 546 (1.7%) | 129 (1.6%) | 0.01 | 6,994 (10.5%) | 1,785 (11.6%) | -0.04 |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 3,851 (11.2%) | 1,012 (14.3%) | -0.09 | 367 (1.1%) | 78 (0.9%) | 0.02 | 4,218 (6.3%) | 1,090 (7.1%) | -0.03 |
| Lab values- LDL level (mg/dl) (within 6 months) ; n (%) | 6,448 (18.8%) | 1,656 (23.4%) | -0.11 | 546 (1.7%) | 129 (1.6%) | 0.01 | 6,994 (10.5%) | 1,785 (11.6%) | -0.04 |
| Lab values- NT-proBNP; n (%) | 61 (0.2%) | 11 (0.2%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 62 (0.1%) | 12 (0.1%) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Lab values- NT-proBNP (within 3 months); n (%) | 47 (0.1%) | 7 (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 48 (0.1%) | 8 (0.1%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- NT-proBNP (within 6 months);<br>n (%) | 61 (0.2%) | 11 (0.2%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 62 (0.1%) | 12 (0.1%) | 0.00 |
| Lab values- Total cholesterol (mg/dl); n (%) | 6,353 (18.5%) | 1,612 (22.8%) | -0.11 | 471 (1.4%) | 123 (1.5%) | -0.01 | 6,824 (10.2%) | 1,735 (11.3%) | -0.04 |
| Lab values-Total cholesterol (mg/dl)<br>(within 3 months); n (%) | 3,786 (11.1%) | 970 (13.7%) | -0.08 | 298 (0.9%) | 71 (0.9%) | 0.00 | 4,084 (6.1%) | 1,041 (6.8%) | -0.03 |
| Lab values- Total cholesterol (mg/dl)<br>(within 6 months); n (%) | 6,353 (18.5%) | 1,612 (22.8%) | -0.11 | 471 (1.4%) | 123 (1.5%) | -0.01 | 6,824 (10.2%) | 1,735 (11.3%) | -0.04 |
| Lab values- Triglyceride level (mg/dl); n (%) | 6,221 (18.2%) | 1,597 (22.6%) | -0.11 | 472 (1.4%) | 119 (1.4%) | 0.00 | 6,693 (10.0%) | 1,716 (11.2%) | -0.04 |
| Lab values- Triglyceride level (mg/dl)<br>(within 3 months); n (%) | 3,695 (10.8%) | 963 (13.6%) | -0.09 | 296 (0.9%) | 70 (0.8%) | 0.01 | 3,991 (6.0%) | 1,033 (6.7%) | -0.03 |
| Lab values-Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 6,221 (18.2%) | 1,597 (22.6%) | -0.11 | 472 (1.4%) | 119 (1.4%) | 0.00 | 6,693 (10.0%) | 1,716 (11.2%) | -0.04 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 5,556 | 1,478 | | 464 | 125 | | 0 | 0 | |
| mean (sd) | 7.20 (1.75) | 7.29 (1.78) | -0.05 | 8.06 (1.91) | 7.73 (1.79) | 0.18 | 7.62 (1.83) | 7.53 (1.79) | 0.05 |
| median [IQR] | 6.70 [6.00, 7.90] | 6.80 [6.00, 8.08] | -0.06 | 7.55 [6.60, 9.20] | 7.30 [6.30, 9.00] | 0.14 | 7.11 (1.83) | 7.07 (1.79) | 0.02 |
| Missing; n (%) | 28,695 (83.8%) | 5,600 (79.1%) | 0.12 | 32,101 (98.6%) | 8,139 (98.5%) | 0.01 | 60,796 (91.0%) | 13,739 (89.6%) | 0.05 |
| Lab result number- BNP mean | 376 | 75 | | 44 | 2 | | 0 | 0 | |
| mean (sd) | 527.10 (1,591.70) | 345.44 (674.53) | 0.15 | 900.99 (2,781.11) | 334.50 (0.71) | 0.29 | 709.33 (2251.31) | 339.55 (458.16) | 0.23 |
| median [IQR] | 163.50 [67.92,<br>456.20] | 99.00 [44.50, 280.00] | 0.05 | 180.00 [51.75,<br>426.75] | 334.50 [334.00,<br>335.00] | -0.08 | 171.54 (2251.31) | 225.85 (458.16) | -0.03 |
| Missing; n (%) | 33,875 (98.9%) | 7,003 (98.9%) | 0.00 | 32,521 (99.9%) | 8,262 (100.0%) | -0.04 | 66,396 (99.4%) | 15,265 (99.5%) | -0.01 |
| Lab result number- BUN (mg/dl) mean | 8,281 | 2,014 | | 452 | 141 | | 0 | 0 | |
| mean (sd) | 19.75 (9.07) | 18.87 (7.63) | 0.10 | 571.73 (8,364.27) | 2,768.72 (19,247.11) | -0.15 | 288.78 (5839.34) | 1500.08 (14126.08) | -0.11 |
| median [IQR] | 18.00 [14.00, 23.00] | 17.00 [14.00, 22.00] | 0.12 | 17.00 [14.00, 21.46] | 17.00 [13.50, 21.00] | 0.00 | 17.51 (5839.34) | 17.00 (14126.08) | 0.00 |
| Missing; n (%) | 25,970 (75.8%) | 5,064 (71.5%) | 0.10 | 32,113 (98.6%) | 8,123 (98.3%) | 0.02 | 58,083 (86.9%) | 13,187 (86.0%) | 0.03 |
| Lab result number- Creatinine (mg/dl)<br>mean (only 0.1 to 15 included) | 8,378 | 2,055 | | 426 | 124 | | 0 | 0 | |
| ` . '. | 1.11 (0.46) | 1.08 (0.40) | 0.07 | 1.05 (0.59) | 1.00 (0.23) | 0.11 | 1.08 (0.53) | 1.04 (0.32) | 0.09 |
| mean (sd)<br>median [IQR] | 1.01 [0.85, 1.24] | 1.00 [0.84, 1.21] | 0.07 | 0.98 [0.83, 1.12] | 1.00 (0.23) | -0.04 | 1.00 (0.53) | 1.04 (0.32) | 0.09 |
| Missing; n (%) | 25,873 (75.5%) | 5,023 (71.0%) | 0.02 | 32,139 (98.7%) | 8,140 (98.5%) | 0.02 | 58,012 (86.8%) | 13,163 (85.8%) | 0.03 |
| Lab result number- HDL level (mg/dl) mean (only =<5000 included) | 6,291 | 1,583 | 0.10 | 480 | 121 | 0.02 | 0 | 0 | 0.03 |
| mean (sd) | 47.14 (15.16) | 46.42 (13.96) | 0.05 | 41.22 (13.28) | 42.43 (12.34) | -0.09 | 44.25 (14.27) | 44.27 (13.11) | 0.00 |
| median [IQR] | 45.00 [37.00, 55.00] | 44.00 [37.00, 54.00] | 0.07 | • • | 40.00 [35.00, 50.00] | 0.00 | 42.56 (14.27) | 41.85 (13.11) | 0.05 |
| Missing; n (%) | 27,960 (81.6%) | 5,495 (77.6%) | 0.10 | 32,085 (98.5%) | 8,143 (98.5%) | 0.00 | 60,045 (89.9%) | 13,638 (88.9%) | 0.03 |
| Lab result number- LDL level (mg/dl) mean (only =<5000 included) | 6,290 | 1,620 | | 465 | 114 | | 0 | 0 | |
| mean (sd) | 99.66 (43.64) | 103.21 (43.70) | -0.08 | 95.58 (49.98) | 97.40 (47.25) | -0.04 | 97.67 (46.84) | 100.08 (45.65) | -0.05 |
| median [IQR] | 97.00 [72.00, 126.00] | 100.00 [75.00,<br>130.00] | -0.07 | 92.00 [66.00,<br>125.75] | 104.00 [61.75,<br>130.38] | -0.25 | 94.56 (46.84) | 102.15 (45.65) | -0.16 |
| Missing; n (%) | 27,961 (81.6%) | 5,458 (77.1%) | 0.11 | 32,100 (98.6%) | 8,150 (98.6%) | 0.00 | 60,061 (89.9%) | 13,608 (88.7%) | 0.04 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included) | 6,335 | 1,608 | | 469 | 122 | | 0 | 0 | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 183.83 (52.62) | 187.10 (48.78) | -0.06 | 181.89 (60.15) | 191.08 (49.85) | -0.17 | 182.88 (56.42) | 189.24 (49.36) | -0.12 |
| median [IQR] | 178.00 [150.00, | 182.00 [154.00, | -0.08 | 178.00 [145.25, | 190.00 (45.05) | -0.22 | 178.00 (56.42) | 186.31 (49.36) | -0.16 |
| median [regit] | 211.00] | 216.00] | 0.00 | 215.50] | 223.50] | 0.22 | 170.00 (50.42) | 100.51 (45.50) | 0.10 |
| Missing; n (%) | 27,916 (81.5%) | 5,470 (77.3%) | 0.10 | 32,096 (98.6%) | 8,142 (98.5%) | 0.01 | 60,012 (89.8%) | 13,612 (88.7%) | 0.04 |
| Lab result number- Triglyceride level | 6.217 | 1,597 | 0.10 | 470 | 118 | 0.01 | 00,012 (03.070) | 0 | 0.04 |
| (mg/dl) mean (only =<5000 included) | 0,217 | 1,557 | | 470 | 110 | | O | v | |
| mean (sd) | 167.43 (139.68) | 173.67 (120.45) | -0.05 | 192.52 (165.88) | 209.43 (138.42) | -0.11 | 179.66 (153.01) | 192.93 (130.44) | -0.09 |
| median [IQR] | 136.00 [97.00, | 144.50 [105.00, | -0.07 | 157.33 [109.00, | 167.00 [131.75, | -0.06 | 146.40 (153.01) | 156.62 (130.44) | -0.07 |
| median [regit] | 195.50] | 206.00] | 0.07 | 214.50] | 247.75] | 0.00 | 140.40 (155.01) | 130.02 (130.44) | 0.07 |
| Missing; n (%) | 28,034 (81.8%) | 5,481 (77.4%) | 0.11 | 32,095 (98.6%) | 8,146 (98.6%) | 0.00 | 60,129 (90.0%) | 13,627 (88.8%) | 0.04 |
| Lab result number- Hemoglobin mean | 6,311 | 1,527 | 0.11 | 322 | 91 | 0.00 | 0 | 0 | 0.04 |
| (only >0 included) | 0,311 | 1,327 | | 322 | 31 | | O . | Ü | |
| mean (sd) | 13.63 (1.82) | 13.86 (1.78) | -0.13 | 13.56 (2.07) | 111,610.08 | -0.15 | 13.60 (1.95) | 60125.39 | -0.11 |
| () | , | ( | | , , | (1,048,228.73) | | ( , | (769329.27) | |
| median [IQR] | 13.70 [12.40, 14.90] | 14.00 [12.67, 15.10] | -0.17 | 13.70 [12.50, 15.00] | 14.30 [13.00, 15.00] | 0.00 | 13.70 (1.95) | 14.16 (769329.27) | 0.00 |
| | . , . | . , . | | . , . | . , . | | , , | , | |
| Missing; n (%) | 27,940 (81.6%) | 5,551 (78.4%) | 0.08 | 32,243 (99.0%) | 8,173 (98.9%) | 0.01 | 60,183 (90.1%) | 13,724 (89.5%) | 0.02 |
| Lab result number- Serum sodium mean | 8,155 | 2,011 | | 425 | 137 | | 0 | 0 | |
| (only > 90 and < 190 included) | | | | | | | | | |
| mean (sd) | 139.83 (2.95) | 140.07 (2.79) | -0.08 | 138.91 (2.74) | 139.30 (2.58) | -0.15 | 139.38 (2.85) | 139.66 (2.68) | -0.10 |
| median [IQR] | 140.00 [138.00, | 140.00 [138.50, | 0.00 | 139.00 [137.00, | 139.50 [137.75, | -0.19 | 139.51 (2.85) | 139.73 (2.68) | -0.08 |
| | 142.00] | 142.00] | | 141.00] | 141.00] | | | | |
| Missing; n (%) | 26,096 (76.2%) | 5,067 (71.6%) | 0.10 | 32,140 (98.7%) | 8,127 (98.3%) | 0.03 | 58,236 (87.2%) | 13,194 (86.0%) | 0.04 |
| Lab result number- Albumin mean (only >0 | 7,380 | 1,825 | | 361 | 118 | | 0 | 0 | |
| and <=10 included) | | | | | | | | | |
| mean (sd) | 4.16 (0.35) | 4.21 (0.34) | -0.14 | 4.04 (0.65) | 4.01 (0.48) | 0.05 | 4.10 (0.52) | 4.10 (0.42) | 0.00 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.10 [4.00, 4.40] | 4.00 [4.00, 4.30] | 0.18 | 4.15 (0.52) | 4.09 (0.42) | 0.13 |
| Missing; n (%) | 26,871 (78.5%) | 5,253 (74.2%) | 0.10 | 32,204 (98.9%) | 8,146 (98.6%) | 0.03 | 59,075 (88.4%) | 13,399 (87.3%) | 0.03 |
| Lab result number- Glucose (fasting or | 8,076 | 2,007 | | 418 | 139 | | 0 | 0 | |
| random) mean (only 10-1000 included) | | | | | | | | | |
| mean (sd) | 131.19 (59.23) | 135.47 (61.82) | -0.07 | 166.36 (68.04) | 156.18 (62.58) | 0.16 | 148.33 (63.68) | 146.63 (62.23) | 0.03 |
| median [IQR] | 110.50 [95.00, | 114.00 [97.00, | -0.06 | 148.17 [117.50, | 142.00 [111.00, | 0.09 | 128.86 (63.68) | 129.08 (62.23) | 0.00 |
| | 146.38] | 152.50] | | 193.17] | 188.00] | | | | |
| Missing; n (%) | 26,175 (76.4%) | 5,071 (71.6%) | 0.11 | 32,147 (98.7%) | 8,125 (98.3%) | 0.03 | 58,322 (87.3%) | 13,196 (86.0%) | 0.04 |
| Lab result number-Potassium mean (only | 8,373 | 2,050 | | 437 | 133 | | 0 | 0 | |
| 1-7 included) | | | | | | | | | |
| mean (sd) | 4.42 (0.45) | 4.46 (0.44) | -0.09 | 4.32 (0.48) | 4.16 (0.44) | 0.35 | 4.37 (0.46) | 4.30 (0.44) | 0.16 |
| median [IQR] | 4.40 [4.10, 4.70] | 4.44 [4.20, 4.70] | -0.09 | 4.30 [4.00, 4.60] | 4.10 [4.00, 4.40] | 0.43 | 4.35 (0.46) | 4.26 (0.44) | 0.20 |
| Missing; n (%) | 25,878 (75.6%) | 5,028 (71.0%) | 0.10 | 32,128 (98.7%) | 8,131 (98.4%) | 0.03 | 58,006 (86.8%) | 13,159 (85.8%) | 0.03 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 4.00 (2.59) | 3.69 (2.41) | 0.12 | 2.50 (1.89) | 2.21 (1.61) | 0.17 | 3.27 (2.28) | 2.89 (2.02) | 0.18 |
| median [IQR] | 4.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 0.40 | 2.00 [1.00, 4.00] | 2.00 [1.00, 3.00] | 0.00 | 3.03 (2.28) | 2.46 (2.02) | 0.26 |
| Frailty Score (mean): Empirical Version 365 | | | | | | | | | |
| days, | | | | | | | | | |
| mean (sd) | 0.20 (0.06) | 0.20 (0.05) | 0.00 | 0.18 (0.05) | 0.18 (0.04) | 0.00 | 0.19 (0.06) | 0.19 (0.04) | 0.00 |
| • | - | | | | | | | | |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| median [IQR]<br>Healthcare Utilization | 0.19 [0.17, 0.23] | 0.19 [0.16, 0.22] | 0.00 | 0.18 [0.15, 0.20] | 0.17 [0.15, 0.19] | 0.22 | 0.19 (0.06) | 0.18 (0.04) | 0.20 |
|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization; n (%) | 34,191 (99.8%) | 7,071 (99.9%) | -0.03 | 32,565 (100.0%) | 8,264 (100.0%) | #DIV/0! | 66,756 (99.9%) | 15,335 (100.0%) | -0.04 |
| Any hospitalization during prior 31-180 | 2,482 (7.2%) | 418 (5.9%) | 0.05 | 1,256 (3.9%) | 199 (2.4%) | 0.09 | 3,738 (5.6%) | 0,617 (4.0%) | 0.07 |
| days; n (%) | 2,402 (7.270) | 410 (3.370) | 0.03 | 1,230 (3.370) | 133 (2.470) | 0.03 | 3,738 (3.0%) | 0,017 (4.070) | 0.07 |
| Endocrinologist Visit; n (%) | 2,043 (6.0%) | 497 (7.0%) | -0.04 | 1,587 (4.9%) | 464 (5.6%) | -0.03 | 3,630 (5.4%) | 0,961 (6.3%) | -0.04 |
| Endocrinologist Visit (30 days prior); n (%) | 1,167 (3.4%) | 255 (3.6%) | -0.01 | 910 (2.8%) | 244 (3.0%) | -0.01 | 2,077 (3.1%) | 0,499 (3.3%) | -0.01 |
| | 1)107 (51.70) | 255 (5.675) | 0.01 | 310 (21070) | 2 (5.5%) | 0.02 | 2,077 (0.170) | 0) 133 (3.375) | 0.01 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 1,161 (3.4%) | 321 (4.5%) | -0.06 | 877 (2.7%) | 286 (3.5%) | -0.05 | 2,038 (3.1%) | 0,607 (4.0%) | -0.05 |
| Internal medicine/family medicine visits; n (%) | 29,770 (86.9%) | 6,033 (85.2%) | 0.05 | 23,203 (71.3%) | 5,917 (71.6%) | -0.01 | 52,973 (79.3%) | 11,950 (77.9%) | 0.03 |
| Internal medicine/family medicine visits (30 days prior); n (%) | 25,267 (73.8%) | 5,047 (71.3%) | 0.06 | 15,093 (46.3%) | 3,669 (44.4%) | 0.04 | 40,360 (60.4%) | 8,716 (56.8%) | 0.07 |
| Internal medicine/family medicine visits (31 to 180 days prior); n (%) | 22,710 (66.3%) | 4,564 (64.5%) | 0.04 | 18,942 (58.2%) | 4,760 (57.6%) | 0.01 | 41,652 (62.3%) | 9,324 (60.8%) | 0.03 |
| Cardiologist visit; n (%) | 31,825 (92.9%) | 6,595 (93.2%) | -0.01 | 12,667 (38.9%) | 3,160 (38.2%) | 0.01 | 44,492 (66.6%) | 9,755 (63.6%) | 0.06 |
| Number of Cardiologist visits (30 days prior); n (%) | 31,454 (91.8%) | 6,555 (92.6%) | -0.03 | 10,251 (31.5%) | 2,599 (31.4%) | 0.00 | 41,705 (62.4%) | 9,154 (59.7%) | 0.06 |
| Number of Cardiologist visits (31 to 180 | 8,575 (25.0%) | 1,530 (21.6%) | 0.08 | 4,839 (14.9%) | 1,058 (12.8%) | 0.06 | 13,414 (20.1%) | 2,588 (16.9%) | 0.08 |
| days prior); n (%) | | | | | | | | | |
| Electrocardiogram ; n (%) | 32,129 (93.8%) | 6,630 (93.7%) | 0.00 | 19,485 (59.8%) | 4,518 (54.7%) | 0.10 | 51,614 (77.2%) | 11,148 (72.7%) | 0.10 |
| Use of glucose test strips; n (%) | 610 (1.8%) | 134 (1.9%) | -0.01 | 427 (1.3%) | 124 (1.5%) | -0.02 | 1,037 (1.6%) | 0,258 (1.7%) | -0.01 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 10.48 (5.03) | 10.47 (5.09) | 0.00 | 9.73 (4.54) | 9.33 (4.39) | 0.09 | 10.11 (4.80) | 9.86 (4.73) | 0.05 |
| median [IQR] | 10.00 [7.00, 13.00] | 10.00 [7.00, 13.00] | 0.00 | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 9.51 (4.80) | 9.46 (4.73) | 0.01 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 1.17 (0.48) | 1.13 (0.44) | 0.09 | 1.10 (0.35) | 1.06 (0.26) | 0.13 | 1.14 (0.42) | 1.09 (0.35) | 0.13 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.42) | 1.00 (0.35) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 5.07 (4.30) | 4.37 (3.53) | 0.18 | 4.34 (3.10) | 3.58 (2.06) | 0.29 | 4.71 (3.76) | 3.94 (2.83) | 0.23 |
| median [IQR] | 4.00 [3.00, 6.00] | 3.00 [3.00, 5.00] | 0.25 | 3.00 [3.00, 5.00] | 3.00 [3.00, 4.00] | 0.00 | 3.51 (3.76) | 3.00 (2.83) | 0.15 |
| Number of Emergency Department (ED) | | | | | | | | | |
| visits | | | | | | | | | |
| mean (sd) | 1.26 (1.65) | 1.17 (1.73) | 0.05 | 3.03 (5.26) | 3.33 (5.85) | -0.05 | 2.12 (3.86) | 2.33 (4.45) | -0.05 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 0.00 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.00 | 1.49 (3.86) | 1.54 (4.45) | -0.01 |
| Number of Office visits | | 0.00 (0.70) | | 0.00 (0.50) | 0.05 (0.00) | | 0 = 4 (0 = 5) | 0.40.40.45 | |
| mean (sd) | 4.08 (3.94) | 3.98 (3.73) | 0.03 | 3.39 (3.56) | 3.06 (3.22) | 0.10 | 3.74 (3.76) | 3.48 (3.46) | 0.07 |
| median [IQR] | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 0.00 | 2.00 [1.00, 5.00] | 2.00 [1.00, 4.00] | 0.00 | 2.51 (3.76) | 2.46 (3.46) | 0.01 |
| Number of Endocrinologist visits | 0.05 (4.50) | 0.00(4.00) | | 0.04 (4.00) | 0.04 (4.54) | | 0.75 (4.50) | 0.57 (4.50) | |
| mean (sd) | 0.26 (1.62) | 0.30 (1.89) | -0.02 | 0.21 (1.33) | 0.24 (1.51) | -0.02 | 0.75 (1.50) | 0.67 (1.62) | 0.05 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.51 (1.50) | 0.46 (1.62) | 0.03 |
| Number of internal medicine/family | | | | | | | | | |
| medicine visits | 40.20/44.40\ | 0.76 (42.22) | 0.05 | E 04 /2 06\ | 4 5 4 /7 34 ) | 0.00 | 7.76 (44.56) | C OF /40 46\ | 0.07 |
| mean (sd) | 10.38 (14.10) | 9.76 (13.28) | 0.05 | 5.01 (8.06) | 4.54 (7.21) | 0.06 | 7.76 (11.56) | 6.95 (10.46) | 0.07 |
| median [IQR] | 6.00 [2.00, 13.00] | 6.00 [2.00, 12.00] | 0.00 | 3.00 [0.00, 6.00] | 2.00 [0.00, 6.00] | 0.13 | 4.54 (11.56) | 3.85 (10.46) | 0.06 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Number of Cardiologist visits | | | | | | | | | I |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 9.25 (6.90) | 9.65 (6.77) | -0.06 | 1.38 (2.87) | 1.29 (2.61) | 0.03 | 5.41 (5.33) | 5.15 (4.98) | 0.05 |
| median [IQR] | 8.00 [5.00, 12.00] | 9.00 [6.00, 12.00] | -0.15 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 4.10 (5.33) | 4.15 (4.98) | -0.01 |
| Number electrocardiograms received | | | | | | | | | |
| mean (sd) | 3.66 (3.02) | 3.56 (2.99) | 0.03 | 1.26 (1.60) | 1.08 (1.47) | 0.12 | 2.49 (2.43) | 2.22 (2.30) | 0.11 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 2.03 (2.43) | 1.92 (2.30) | 0.05 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 0.47 (0.76) | 0.55 (0.79) | -0.10 | 0.28 (0.60) | 0.34 (0.65) | -0.10 | 0.38 (0.69) | 0.44 (0.72) | -0.09 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.69) | 0.00 (0.72) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.27 (2.79) | 0.30 (2.78) | -0.01 | 0.16 (0.78) | 0.16 (0.96) | 0.00 | 0.22 (2.07) | 0.22 (2.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (2.07) | 0.00 (2.02) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.58 (0.81) | 0.61 (0.80) | -0.04 | 0.39 (0.83) | 0.44 (0.85) | -0.06 | 0.49 (0.82) | 0.52 (0.83) | -0.04 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.82) | 0.00 (0.83) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.06 (0.33) | 0.06 (0.34) | 0.00 | 0.06 (0.33) | 0.03 (0.22) | 0.11 | 0.06 (0.33) | 0.04 (0.28) | 0.07 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.33) | 0.00 (0.28) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.04 (0.27) | 0.04 (0.27) | 0.00 | 0.03 (0.23) | 0.02 (0.16) | 0.05 | 0.04 (0.25) | 0.03 (0.22) | 0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.25) | 0.00 (0.22) | 0.00 |
| Number of tests for microalbuminuria | | | | / > | | | | | |
| mean (sd) | 0.28 (0.78) | 0.34 (0.81) | -0.08 | 0.14 (0.53) | 0.16 (0.56) | -0.04 | 0.21 (0.67) | 0.24 (0.69) | -0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.67) | 0.00 (0.69) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at | | | | | | | | | |
| the 3rd digit level | 11 70 /12 20\ | 12 42 (11 20) | 0.14 | C 4C (0.02) | 7.00 (0.45) | 0.17 | 0.10/10.70 | 10 45 (0 03) | 0.12 |
| mean (sd) | 11.78 (12.28) | 13.43 (11.39) | -0.14<br>-0.25 | 6.46 (8.93)<br>0.00 [0.00, 13.00] | 7.90 (8.45) | -0.17<br>-0.69 | 9.19 (10.78) | 10.45 (9.92) | -0.12<br>-0.40 |
| median [IQR] For PS | 9.00 [0.00, 18.00] | 12.00 [4.00, 19.00] | -0.23 | 0.00 [0.00, 15.00] | 6.00 [0.00, 14.00] | -0.09 | 4.61 (10.78) | 8.77 (9.92) | -0.40 |
| Hemorrhagic stroke+Other | 1,184 (3.5%) | 166 (2.3%) | 0.07 | 615 (1.9%) | 81 (1.0%) | 0.08 | 1799 (2.7%) | 247 (1.6%) | 0.08 |
| cerebrovascular disease+Cerebrovascular | 1,164 (5.5%) | 100 (2.3%) | 0.07 | 013 (1.5%) | 81 (1.0%) | 0.08 | 1799 (2.770) | 247 (1.0%) | 0.08 |
| procedure (for PS); n (%) | | | | | | | | | |
| Occurrence of creatinine tests ordered (for | 1,600 (4.7%) | 304 (4.3%) | 0.02 | 1,402 (4.3%) | 222 (2.7%) | 0.09 | 3,002 (4.5%) | 0,526 (3.4%) | 0.06 |
| PS); n (%) | 1,000 (4.770) | 304 (4.370) | 0.02 | 1,102 (1.370) | 222 (2.770) | 0.03 | 3,002 (4.370) | 0,320 (3.470) | 0.00 |
| Occurrence of BUN tests ordered (for PS); n | 910 (2.7%) | 177 (2.5%) | 0.01 | 786 (2.4%) | 120 (1.5%) | 0.07 | 1,696 (2.5%) | 0,297 (1.9%) | 0.04 |
| (%) | ( | ( , | | ( | , | | , , | -, - ( , | |
| Occurrence of chronic renal insufficiency | 4,154 (12.1%) | 710 (10.0%) | 0.07 | 1,526 (4.7%) | 247 (3.0%) | 0.09 | 5,680 (8.5%) | 0,957 (6.2%) | 0.09 |
| w/o CKD (for PS) ; n (%) | | | | | | | | | |
| Chronic kidney disease Stage 1-2 (for PS); n | 1,225 (3.6%) | 289 (4.1%) | -0.03 | 380 (1.2%) | 84 (1.0%) | 0.02 | 1605 (2.4%) | 373 (2.4%) | 0.00 |
| (%) | | | | | | | | | |
| Chronic kidney disease Stage 3-6 (for PS); n | 5,711 (16.7%) | 1,118 (15.8%) | 0.02 | 2,015 (6.2%) | 365 (4.4%) | 0.08 | 7,726 (11.6%) | 1,483 (9.7%) | 0.06 |
| (%) | | | | | | | | | |
| Bladder stones+Kidney stones (for PS); n (%) | 990 (2.9%) | 223 (3.2%) | -0.02 | 535 (1.6%) | 151 (1.8%) | -0.02 | 1,525 (2.3%) | 0,374 (2.4%) | -0.01 |
| Diabetes with peripheral circulatory disorders+Gangrene+Osteomyelitis(for PS) with ICD10; n (%) | 2,069 (6.0%) | 493 (7.0%) | -0.04 | 735 (2.3%) | 166 (2.0%) | 0.02 | 2,804 (4.2%) | 0,659 (4.3%) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Alcohol abuse or dependence+Drug abuse | 1,634 (4.8%) | 350 (4.9%) | 0.00 | 886 (2.7%) | 219 (2.7%) | 0.00 | 2520 (3.8%) | 569 (3.7%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| or dependence (for PS); n (%) | | | | | | | | | |
| Diabetes with other ophthalmic | 338 (1.0%) | 73 (1.0%) | 0.00 | 549 (1.7%) | 116 (1.4%) | 0.02 | 0,887 (1.3%) | 0,189 (1.2%) | 0.01 |
| manifestations+Retinal detachment, | | | | | | | | | |
| vitreous hemorrhage, vitrectomy+Retinal | | | | | | | | | |
| laser coagulation therapy (for PS); n (%) | | | | | | | | | |
| Other atherosclerosis+Cardiac conduction | 17,674 (51.6%) | 3,269 (46.2%) | 0.11 | 12,419 (38.1%) | 2,749 (33.3%) | 0.10 | 30,093 (45.0%) | 6,018 (39.2%) | 0.12 |
| disorders+Other CVD (for PS); n (%) | | | | | | | | | |
| Previous cardiac procedure (CABG or PTCA | 27,865 (81.4%) | 6,730 (95.1%) | -0.44 | 25,351 (77.8%) | 7,635 (92.4%) | -0.42 | 53,216 (79.6%) | 14,365 (93.6%) | -0.42 |
| or Stent) + History of CABG or PTCA (for PS) | ' ' | 0,: 00 (00:=,:,) | | | ( = : : : : ) | | / ( , | , (, | **** |
| ; n (%) | | | | | | | | | |
| Hyperthyroidism + Hypothyroidism + | 6,302 (18.4%) | 1,303 (18.4%) | 0.00 | 3,926 (12.1%) | 923 (11.2%) | 0.03 | 10,228 (15.3%) | 2,226 (14.5%) | 0.02 |
| Other disorders of thyroid gland (for PS); n | | | | | | | | | |
| (%) | | | | | | | | | |
| Delirium + Psychosis (for PS); n (%) | 1,418 (4.1%) | 209 (3.0%) | 0.06 | 690 (2.1%) | 100 (1.2%) | 0.07 | 2108 (3.2%) | 309 (2.0%) | 0.08 |
| Any use of Meglitinides (for PS); n (%) | 95 (0.3%) | 21 (0.3%) | 0.00 | 112 (0.3%) | 31 (0.4%) | -0.02 | 207 (0.3%) | 52 (0.3%) | 0.00 |
| Any use of AGIs (for PS); n (%) | 35 (0.1%) | 7 (0.1%) | 0.00 | 40 (0.1%) | 10 (0.1%) | 0.00 | 30,093 (45.0%) | 6,018 (39.2%) | 0.12 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 5,711 (16.7%) | 1,118 (15.8%) | 0.02 | 2,015 (6.2%) | 365 (4.4%) | 0.08 | 7,726 (11.6%) | 1,483 (9.7%) | 0.06 |
| Use of thiazide; n (%) | 3,544 (10.3%) | 675 (9.5%) | 0.03 | 2,983 (9.2%) | 654 (7.9%) | 0.05 | 59,039 (88.4%) | 13,609 (88.7%) | -0.01 |
| Use of beta blockers; n (%) | 30,072 (87.8%) | 6,231 (88.0%) | -0.01 | 28,967 (89.0%) | 7,378 (89.3%) | -0.01 | 18,021 (27.0%) | 3,660 (23.9%) | 0.07 |
| Use of calcium channel blockers; n (%) | 9,975 (29.1%) | 1,923 (27.2%) | 0.04 | 8,046 (24.7%) | 1,737 (21.0%) | 0.09 | 18,802 (28.1%) | 4,954 (32.3%) | -0.09 |
| All antidiabetic medications except | 10,056 (29.4%) | 2,541 (35.9%) | -0.14 | 8,746 (26.9%) | 2,413 (29.2%) | -0.05 | 6,527 (9.8%) | 1,329 (8.7%) | 0.04 |
| Insulin; n (%) | | | | | | | | | |
| DM Medications - Insulin ; n (%) | 4,442 (13.0%) | 1,074 (15.2%) | -0.06 | 3,925 (12.1%) | 1,017 (12.3%) | -0.01 | 8,367 (12.5%) | 2,091 (13.6%) | -0.03 |
| Use of Low Intensity Statins; n (%) | 12,706 (37.1%) | 2,017 (28.5%) | 0.18 | 12,432 (38.2%) | 2,215 (26.8%) | 0.25 | 25138 (37.6%) | 4,232 (27.6%) | 0.21 |
| Use of High Intensity Statins; n (%) | 21,258 (62.1%) | 5,363 (75.8%) | -0.30 | 19,285 (59.2%) | 6,350 (76.8%) | -0.38 | 40543 (60.7%) | 11,713 (76.3%) | -0.34 |
| Malignant hypertension; n (%) | 2,762 (8.1%) | 322 (4.5%) | 0.15 | 17,029 (52.3%) | 2,783 (33.7%) | 0.38 | 19791 (29.6%) | 3,105 (20.2%) | 0.22 |
| Cardiovascular stress test; n (%) | 103 (0.3%) | 19 (0.3%) | 0.00 | 93 (0.3%) | 17 (0.2%) | 0.02 | 0,196 (0.3%) | 36 (0.2%) | 0.02 |
| Echocardiogram; n (%) | 26,110 (76.2%) | 5,478 (77.4%) | -0.03 | 22,761 (69.9%) | 5,951 (72.0%) | -0.05 | 48,871 (73.1%) | 11429 (74.5%) | -0.03 |
| Number of BNP tests | | | | | | | | | |
| mean (sd) | 0.12 (0.48) | 0.11 (0.45) | 0.02 | 0.12 (0.43) | 0.12 (0.38) | 0.00 | 0.12 (0.46) | 0.12 (0.41) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.46) | 0.00 (0.41) | 0.00 |
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.62 (1.74) | 0.59 (1.81) | 0.02 | 0.67 (1.58) | 0.66 (1.58) | 0.01 | 0.64 (1.66) | 0.63 (1.69) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.66) | 0.00 (1.69) | 0.00 |
| Number of Ambulatory Blood pressure | | | | | | | | | |
| monitoring tests | | () | | /> | | | / , | /> | |
| mean (sd) | 0.00 (0.03) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.03) | 0.00 | 0.00 (0.03) | 0.00 (0.03) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.03) | 0.00 |
| N of days on antihypertensive medications | | | | | | | | | |
| during baseline | 405 60 (77 47) | 100.06 (70.12) | 0.00 | 02 62 (70 42) | 02.02.(70.54) | 0.40 | 00 04 (70 42) | 04.74.70.00\ | 0.40 |
| mean (sd) | 105.69 (77.47) | 100.86 (78.13) | 0.06 | 93.62 (79.43) | 83.92 (79.54) | 0.12 | 99.81 (78.43) | 91.74 (78.89) | 0.10 |
| median [IQR] | 147.00 [1.00, 179.00] | 135.00 [1.00, 1/8.00] | 0.15 | 115.00 [1.00,<br>177.00] | 78.00 [1.00, 173.00] | 0.47 | 131.40 (78.43) | 104.30 (78.89) | 0.34 |
| N of days in database anytime prior | | | | 1//.00] | | | | | |
| 1 ,, , | 1 | | | | | | | | Ī |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| 1 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 1,835.09 (1,422.04) | 1,784.22 (1,449.19) | 0.04 | 2,135.45 (1,386.94) | 2,271.61 (1,503.12) | -0.09 | 1981.48 (1405.04) | 2046.75 (1478.48) | -0.05 |
| median [IQR] | 1,433.00 [681.00, | 1,315.00 [637.75, | 0.08 | 1,880.00 [915.00, | 1,999.00 [950.00, | -0.08 | 1650.86 (1405.04) | 1683.44 (1478.48) | -0.02 |
| | 2,665.00] | 2,606.25] | | 3,295.00] | 3,558.00] | | | | |
| Mean Copay for per prescription cost | | | | | | | | | |
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 23.29 (34.93) | 22.94 (32.38) | 0.01 | 18.45 (26.28) | 16.63 (21.49) | 0.08 | 20.93 (31.02) | 19.54 (27.06) | 0.05 |
| median [IQR] | 14.29 [5.85, 29.58] | 13.92 [5.00, 29.49] | 0.01 | 12.82 [5.08, 24.33] | 10.80 [3.33, 22.51] | 0.08 | 13.57 (31.02) | 12.24 (27.06) | 0.05 |
| Missing; n (%) | 3,156 (9.2%) | 609 (8.6%) | 0.02 | 3,809 (11.7%) | 993 (12.0%) | -0.01 | 6,965 (10.4%) | 1602 (10.4%) | 0.00 |
| Colonos; n (%) | 1,177 (3.4%) | 279 (3.9%) | -0.03 | 991 (3.0%) | 292 (3.5%) | -0.03 | 2,168 (3.2%) | 571 (3.7%) | -0.03 |
| Fecal occult blood (FOB) test; n (%) | 1,073 (3.1%) | 200 (2.8%) | 0.02 | 886 (2.7%) | 180 (2.2%) | 0.03 | 1,959 (2.9%) | 380 (2.5%) | 0.02 |
| Flu vaccine; n (%) | 5,381 (15.7%) | 1,085 (15.3%) | 0.01 | 3,101 (9.5%) | 723 (8.7%) | 0.03 | 8,482 (12.7%) | 1808 (11.8%) | 0.03 |
| Mammogram; n (%) | 2,131 (6.2%) | 468 (6.6%) | -0.02 | 1,397 (4.3%) | 322 (3.9%) | 0.02 | 3,528 (5.3%) | 790 (5.1%) | 0.01 |
| Pap smear; n (%) | 485 (1.4%) | 114 (1.6%) | -0.02 | 654 (2.0%) | 136 (1.6%) | 0.03 | 1,139 (1.7%) | 250 (1.6%) | 0.01 |
| Pneumonia vaccine; n (%) | 5,203 (15.2%) | 1,341 (18.9%) | -0.10 | 2,015 (6.2%) | 721 (8.7%) | -0.10 | 7,218 (10.8%) | 2062 (13.4%) | -0.08 |
| PSA test or Prostate exam for DRE; n (%) | 4,519 (13.2%) | 1,008 (14.2%) | -0.03 | 3,148 (9.7%) | 932 (11.3%) | -0.05 | 7,667 (11.5%) | 1940 (12.6%) | -0.03 |
| Bone mineral density; n (%) | 847 (2.5%) | 171 (2.4%) | 0.01 | 371 (1.1%) | 87 (1.1%) | 0.00 | 1,218 (1.8%) | 258 (1.7%) | 0.01 |
| Use of Sympatomimetic agents; n (%) | 190 (0.6%) | 47 (0.7%) | -0.01 | 249 (0.8%) | 94 (1.1%) | -0.03 | 0,439 (0.7%) | 141 (0.9%) | -0.02 |
| Use of CNS stimulants; n (%) | 102 (0.3%) | 24 (0.3%) | 0.00 | 162 (0.5%) | 48 (0.6%) | -0.01 | 0,264 (0.4%) | 72 (0.5%) | -0.01 |
| Use of estrogens, progestins, androgens; n | 845 (2.5%) | 197 (2.8%) | -0.02 | 1,332 (4.1%) | 328 (4.0%) | 0.01 | 2,177 (3.3%) | 525 (3.4%) | -0.01 |
| (%) | 17 (0.0%) | 5 (0.1%) | -0.04 | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 0,017 (0.0%) | 6 (0.0%) | #DIV/0! |
| Use of Angiogenesis inhibitors; n (%) Use of Oral Immunosuppressants; n (%) | 52 (0.2%) | 5 (0.1%)<br>15 (0.2%) | 0.04 | 75 (0.2%) | 22 (0.3%) | #DIV/0!<br>-0.02 | 0,017 (0.0%) | 37 (0.2%) | #DIV/0!<br>0.00 |
| | ' ' | , , | | , , | , , | | | , , | |
| Use of fondaparinux or Bivalirudin; n (%) | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 9 (0.0%) | 0 (0.0%) | #DIV/0! | 0,012 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of other direct thrombin inhibitors (lepirudin, desirudin, argatroban); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Prasugrel ON CED; n (%) | 148 (0.4%) | 29 (0.4%) | 0.00 | 155 (0.5%) | 34 (0.4%) | 0.01 | 0,303 (0.5%) | 63 (0.4%) | 0.01 |
| Use of Prasugrel 180 to 1 day prior; n (%) | 213 (0.6%) | 65 (0.9%) | -0.03 | 205 (0.6%) | 59 (0.7%) | -0.01 | 0,418 (0.6%) | 124 (0.8%) | -0.02 |
| Duration of index hospitalization (i.e. | 213 (0.0%) | 03 (0.976) | -0.03 | 203 (0.0%) | 39 (0.778) | -0.01 | 0,418 (0.0%) | 124 (0.8%) | -0.02 |
| anchor hospitalization (i.e. | | | | | | | | | |
| mean (sd) | 4.54 (3.88) | 3.98 (3.03) | 0.16 | 3.97 (2.44) | 3.38 (1.57) | 0.29 | 4.26 (3.26) | 3.66 (2.36) | 0.21 |
| median [IQR] | 4.00 [3.00, 5.00] | 3.00 [3.00, 4.00] | 0.29 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.51 (3.26) | 3.00 (2.36) | 0.18 |
| Number of D-dimer tests | 4.00 [5.00, 5.00] | 3.00 [3.00, 4.00] | 0.23 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.31 (3.20) | 3.00 (2.30) | 0.10 |
| mean (sd) | 0.04 (0.23) | 0.04 (0.23) | 0.00 | 0.05 (0.23) | 0.06 (0.26) | -0.04 | 0.04 (0.23) | 0.05 (0.25) | -0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.23) | 0.00 (0.25) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.23) | 0.00 (0.23) | 0.00 |
| mean (sd) | 0.06 (0.33) | 0.06 (0.30) | 0.00 | 0.04 (0.27) | 0.04 (0.27) | 0.00 | 0.05 (0.30) | 0.05 (0.28) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.30) | 0.00 (0.28) | 0.00 |
| Number of PT or aPTTt tests | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.50) | 0.00 (0.20) | 0.00 |
| mean (sd) | 0.59 (1.97) | 0.40 (1.37) | 0.11 | 0.48 (1.37) | 0.37 (0.98) | 0.09 | 0.54 (1.70) | 0.38 (1.18) | 0.11 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.40 (1.37) | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.70) | 0.00 (1.18) | 0.00 |
| Number of Bleeding time tests | 0.00 [0.00, 0.00] | 3.00 [0.00, 0.00] | 0.00 | 3.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.70) | 0.00 (1.10) | 0.00 |
| mean (sd) | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| days | | | | | | | | | |
| mean (sd) | 4.05 (0.76) | 3.90 (0.75) | 0.20 | 3.57 (0.66) | 3.36 (0.59) | 0.34 | 3.82 (0.71) | 3.61 (0.67) | 0.30 |
| (3u) | 4.03 (0.70) | 3.30 (0.73) | 0.20 | 3.37 (0.00) | 3.30 (0.33) | 0.54 | 3.02 (0.71) | 3.01 (0.07) | 0.50 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| median [IQR] | 4.00 [4.00, 4.00] | 4.00 [3.00, 4.00] | 0.00 | 4.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 1.60 | 4.00 (0.71) | 3.46 (0.67) | 0.78 |
|---|---|---|---|---|---|---|---|---|---|
| Drug eluting stent; n (%) | 8,430 (24.6%) | 1,218 (17.2%) | 0.18 | 10,014 (30.8%) | 2,371 (28.7%) | 0.05 | 18,444 (27.6%) | 3589 (23.4%) | 0.10 |
| Bare metal stent; n (%) | 18,447 (53.9%) | 5,947 (84.0%) | -0.69 | 15,203 (46.7%) | 7,011 (84.8%) | -0.88 | 33,650 (50.4%) | 12958 (84.5%) | -0.78 |
| Use of CYP inhibitors; n (%) | 7,802 (22.8%) | 1,443 (20.4%) | 0.06 | 6,227 (19.1%) | 1,374 (16.6%) | 0.07 | 14,029 (21.0%) | 2817 (18.4%) | 0.07 |
| Use of CYP inducers; n (%) | 41 (0.1%) | 7 (0.1%) | 0.00 | 64 (0.2%) | 9 (0.1%) | 0.03 | 0,105 (0.2%) | 16 (0.1%) | 0.03 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code - CORRECT ONE - | | | | | | | | | |
| TRUVEN | | | | | | | | | |
| Commercial; n (%) | 9,219 (26.9%) | 2,194 (31.0%) | -0.09 | 15,361 (47.2%) | 2,555 (30.9%) | 0.34 | 24,580 (36.8%) | 4749 (31.0%) | 0.12 |
| Medicare Advantage; n (%) | 25,032 (73.1%) | 4,884 (69.0%) | 0.09 | 17,204 (52.8%) | 5,709 (69.1%) | -0.34 | 42,236 (63.2%) | 10593 (69.0%) | -0.12 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 9,219 (26.9%) | 2,194 (31.0%) | -0.09 | - | - | #VALUE! | 9,219 (26.9%) | 2,194 (31.0%) | -0.09 |
| MCR = MEDICARE; n (%) | 25,032 (73.1%) | 4,884 (69.0%) | 0.09 | - | - | #VALUE! | 25,032 (73.1%) | 4,884 (69.0%) | 0.09 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| in 2015); n (%) | | | | | | | | | |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data | | | | | | | | | |
| Туре | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 15,223 (46.7%) | 5,158 (62.4%) | -0.32 | 15,223 (46.7%) | 5,158 (62.4%) | -0.32 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 1,981 (6.1%) | 551 (6.7%) | -0.02 | 1,981 (6.1%) | 551 (6.7%) | -0.02 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 13,443 (41.3%) | 2,290 (27.7%) | 0.29 | 13,443 (41.3%) | 2,290 (27.7%) | 0.29 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 1,918 (5.9%) | 265 (3.2%) | 0.13 | 1,918 (5.9%) | 265 (3.2%) | 0.13 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural (non-MSA) | | | | | | | | | |
| Urban; n (%) | - | - | #VALUE! | 23,495 (72.1%) | 5,859 (70.9%) | 0.03 | 23,495 (72.1%) | 5,859 (70.9%) | 0.03 |
| Rural; n (%) | - | - | #VALUE! | 1,316 (4.0%) | 628 (7.6%) | -0.15 | 1,316 (4.0%) | 628 (7.6%) | -0.15 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 7,754 (23.8%) | 1,777 (21.5%) | 0.05497 | 7,754 (23.8%) | 1,777 (21.5%) | 0.05 |
| N of Generic name drugs | | | | | | | | | |
| mean (sd) | 17.06 (13.53) | 15.92 (13.38) | 0.08 | 13.50 (10.40) | 12.08 (9.64) | 0.14 | 15.32 (12.11) | 13.85 (11.52) | 0.12 |
| median [IQR] | 14.00 [8.00, 22.00] | 12.00 [7.00, 21.00] | 0.15 | 11.00 [6.00, 18.00] | 10.00 [5.00, 16.00] | 0.10 | 12.54 (12.11) | 10.92 (11.52) | 0.14 |
| N of Brand name drugs | | | | | | | | | |
| mean (sd) | 3.13 (4.46) | 3.86 (4.39) | -0.16 | 3.48 (4.24) | 3.82 (3.89) | -0.08 | 3.30 (4.35) | 3.84 (4.13) | -0.13 |
| median [IQR] | 1.00 [0.00, 4.00] | 2.00 [1.00, 5.00] | -0.226 | 2.00 [1.00, 5.00] | 2.00 [1.00, 5.00] | 0 | 1.49 (4.35) | 2.00 (4.13) | -0.12 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| | | | PS-m | atched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opt | tum | | Truv | /en | | POO | LED | |
| Variable | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. |
| Number of patients | 6,697 | 6,697 | | 7,283 | 7,283 | | 13,980 | 13,980 | ļ |
| Age | | | | | | | | | |
| mean (sd) | 68.19 (10.96) | 68.38 (10.66) | -0.02 | 62.57 (11.12) | 62.72 (10.33) | -0.01 | 65.26 (11.04) | 65.43 (10.49) | -0.02 |
| median [IQR] | 69.00 [61.00, 76.00] | 69.00 [62.00, 76.00] | 0.00 | 62.00 [56.00, | 62.00 [57.00, | 0.00 | 65.35 (11.04) | 65.35 (10.49) | 0.00 |
| Age categories | | | | <del>-</del> | · · · · <del>·</del> | | | | ļ |
| 18 - 54; n (%) | 761 (11.4%) | 716 (10.7%) | 0.02 | 1,548 (21.3%) | 1,372 (18.8%) | 0.06 | 2,309 (16.5%) | 2,088 (14.9%) | 0.04 |
| 55 - 64; n (%) | 1,531 (22.9%) | 1,473 (22.0%) | 0.02 | 3,310 (45.4%) | 3,451 (47.4%) | -0.04 | 4,841 (34.6%) | 4,924 (35.2%) | -0.01 |
| 65 - 74; n (%) | 2,461 (36.7%) | 2,515 (37.6%) | -0.02 | 1,339 (18.4%) | 1,446 (19.9%) | -0.04 | 3,800 (27.2%) | 3,961 (28.3%) | -0.02 |
| >= 75; n (%) | 1,944 (29.0%) | 1,993 (29.8%) | -0.02 | 1,086 (14.9%) | 1,014 (13.9%) | 0.03 | 3,030 (21.7%) | 3,007 (21.5%) | 0.00 |
| Gender | 2,5 (2510,5) | 2,555 (25.575) | 0.02 | 1,000 (1 1.570) | 2,02 (20.570) | 0.00 | 3,000 (2117,0) | 3,007 (22.370) | 0.00 |
| Males; n (%) | 4,290 (64.1%) | 4,277 (63.9%) | 0.00 | 5,161 (70.9%) | 5,145 (70.6%) | 0.01 | 9,451 (67.6%) | 9,422 (67.4%) | 0.00 |
| Females; n (%) | 2,407 (35.9%) | 2,420 (36.1%) | 0.00 | 2,122 (29.1%) | 2,138 (29.4%) | -0.01 | 4,529 (32.4%) | 4,558 (32.6%) | 0.00 |
| Region | 2,407 (33.370) | 2,420 (30.170) | 0.00 | 2,122 (23.170) | 2,130 (23.470) | 0.01 | 4,323 (32.470) | 4,550 (52.070) | 0.00 |
| negion | | | | | | | | | ļ |
| Northeast; n (%) | 777 (11.6%) | 772 (11.5%) | 0.00 | 1,356 (18.6%) | 1,386 (19.0%) | -0.01 | 2,133 (15.3%) | 2,158 (15.4%) | 0.00 |
| South; n (%) | 3,136 (46.8%) | 3,102 (46.3%) | 0.01 | 2,027 (27.8%) | 2,009 (27.6%) | 0.00 | 5,163 (36.9%) | 5,111 (36.6%) | 0.01 |
| Midwest; n (%) | 1,524 (22.8%) | 1,566 (23.4%) | -0.01 | 3,064 (42.1%) | 3,047 (41.8%) | 0.01 | 4,588 (32.8%) | 4,613 (33.0%) | 0.00 |
| West; n (%) | 1,260 (18.8%) | 1,257 (18.8%) | 0.00 | 796 (10.9%) | 803 (11.0%) | 0.00 | 2,056 (14.7%) | 2,060 (14.7%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 40 (0.5%) | 38 (0.5%) | 0.00 | 40 (0.3%) | 38 (0.3%) | 0.00 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 6,697 (100.0%) | 6,697 (100.0%) | #DIV/0! | 7,283 (100.0%) | 7,283 (100.0%) | #DIV/0! | 13,980 (100.0%) | 13,980 (100.0%) | #DIV/0! |
| Acute MI; n (%) | 6,135 (91.6%) | 6,128 (91.5%) | 0.00 | 6,879 (94.5%) | 6,876 (94.4%) | 0.00 | 13014 (93.1%) | 13004 (93.0%) | 0.00 |
| ACS/unstable angina; n (%) | 2,839 (42.4%) | 2,840 (42.4%) | 0.00 | 2,601 (35.7%) | 2,637 (36.2%) | -0.01 | 5440 (38.9%) | 5477 (39.2%) | -0.01 |
| Old MI; n (%) | 1,126 (16.8%) | 1,128 (16.8%) | 0.00 | 684 (9.4%) | 652 (9.0%) | 0.01 | 1810 (12.9%) | 1780 (12.7%) | 0.01 |
| Stable angina; n (%) | 1,622 (24.2%) | 1,691 (25.3%) | -0.03 | 1,196 (16.4%) | 1,199 (16.5%) | 0.00 | 2,818 (20.2%) | 2,890 (20.7%) | -0.01 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 6,437 (96.1%) | 6,433 (96.1%) | 0.00 | 6,745 (92.6%) | 6,733 (92.4%) | 0.01 | 13,182 (94.3%) | 13,166 (94.2%) | 0.00 |
| Other atherosclerosis with ICD10; n (%) | 86 (1.3%) | 81 (1.2%) | 0.01 | 98 (1.3%) | 85 (1.2%) | 0.01 | 184 (1.3%) | 166 (1.2%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or | 6,024 (90.0%) | 6,183 (92.3%) | -0.08 | 6,519 (89.5%) | 6,549 (89.9%) | -0.01 | 12543 (89.7%) | 12732 (91.1%) | -0.05 |
| Stent); n (%) | ,,,,, | 0,200 (02.07.7) | | 0,000 (00.07.7) | 5,5 15 (551511) | | ( | | |
| History of CABG or PTCA; n (%) | 2,490 (37.2%) | 2,351 (35.1%) | 0.04 | 1,494 (20.5%) | 1,309 (18.0%) | 0.06 | 3,984 (28.5%) | 3,660 (26.2%) | 0.05 |
| Any stroke; n (%) | 622 (9.3%) | 601 (9.0%) | 0.01 | 406 (5.6%) | 416 (5.7%) | 0.00 | 1,028 (7.4%) | 1,017 (7.3%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | , , | 598 (8.9%) | 0.01 | 406 (5.6%) | 416 (5.7%) | 0.00 | 1,022 (7.3%) | 1,014 (7.3%) | 0.00 |
| infarction); n (%) | 0 = 0 (0 := ; : ) | (0.07.7) | | (3.37.7) | (=,-, | | _,=== (: :=::, | _,== : (: :=,=, | |
| Hemorrhagic stroke; n (%) | 13 (0.2%) | 7 (0.1%) | 0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 13 (0.1%) | 7 (0.1%) | 0.00 |
| TIA; n (%) | 120 (1.8%) | 125 (1.9%) | -0.01 | 83 (1.1%) | 77 (1.1%) | 0.00 | 203 (1.5%) | 202 (1.4%) | 0.01 |
| Other cerebrovascular disease; n (%) | 143 (2.1%) | 151 (2.3%) | -0.01 | 72 (1.0%) | 73 (1.0%) | 0.00 | 215 (1.5%) | 224 (1.6%) | -0.01 |
| Late effects of cerebrovascular disease; n (%) | 134 (2.0%) | 135 (2.0%) | 0.00 | 51 (0.7%) | 50 (0.7%) | 0.00 | 185 (1.3%) | 185 (1.3%) | 0.00 |
| Cerebrovascular procedure; n (%) | 8 (0.1%) | 8 (0.1%) | 0.00 | 7 (0.1%) | 4 (0.1%) | 0.00 | 15 (0.1%) | 12 (0.1%) | 0.00 |
| Heart failure (CHF); n (%) | 1,722 (25.7%) | 1,720 (25.7%) | 0.00 | 1,134 (15.6%) | 1,134 (15.6%) | 0.00 | 2,856 (20.4%) | 2,854 (20.4%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD<br>Surgery ; n (%) | 874 (13.1%) | 843 (12.6%) | 0.01 | 397 (5.5%) | 394 (5.4%) | 0.00 | 1,271 (9.1%) | 1,237 (8.8%) | 0.01 |
| Atrial fibrillation; n (%) | 815 (12.2%) | 823 (12.3%) | 0.00 | 598 (8.2%) | 561 (7.7%) | 0.02 | 1,413 (10.1%) | 1,384 (9.9%) | 0.01 |
| Other cardiac dysrhythmia; n (%) | 2,463 (36.8%) | 2,524 (37.7%) | -0.02 | 2,216 (30.4%) | 2,204 (30.3%) | 0.00 | 4,679 (33.5%) | 4,728 (33.8%) | -0.01 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Cardiac conduction disorders; n (%) | 1,075 (16.1%) | 1,041 (15.5%) | 0.02 | 749 (10.3%) | 748 (10.3%) | 0.00 | 1824 (13.0%) | 1789 (12.8%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Other CVD; n (%) | 2,475 (37.0%) | 2,563 (38.3%) | -0.03 | 1,945 (26.7%) | 1,998 (27.4%) | -0.02 | 4,420 (31.6%) | 4,561 (32.6%) | -0.02 |
| Diabetes-related complications | , , , | . , , | | | , , , | | , , , | | |
| Diabetic retinopathy; n (%) | 267 (4.0%) | 253 (3.8%) | 0.01 | 144 (2.0%) | 132 (1.8%) | 0.01 | 0,411 (2.9%) | 0,385 (2.8%) | 0.01 |
| Diabetes with other ophthalmic | 25 (0.4%) | 36 (0.5%) | -0.01 | 67 (0.9%) | 63 (0.9%) | 0.00 | 0,092 (0.7%) | 0,099 (0.7%) | 0.00 |
| manifestations; n (%) | - ( / | , | | ( / | , | | ( , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| Retinal detachment, vitreous hemorrhage, | 28 (0.4%) | 15 (0.2%) | 0.04 | 21 (0.3%) | 21 (0.3%) | 0.00 | 49 (0.4%) | 36 (0.3%) | 0.02 |
| vitrectomy; n (%) | | | | | | | | | |
| Retinal laser coagulation therapy; n (%) | 27 (0.4%) | 28 (0.4%) | 0.00 | 34 (0.5%) | 30 (0.4%) | 0.01 | 61 (0.4%) | 58 (0.4%) | 0.00 |
| Occurrence of Diabetic Neuropathy; n (%) | 871 (13.0%) | 833 (12.4%) | 0.02 | 389 (5.3%) | 371 (5.1%) | 0.01 | 1,260 (9.0%) | 1,204 (8.6%) | 0.01 |
| . , , , | | | | | | | | | |
| Occurrence of diabetic nephropathy with | 814 (12.2%) | 805 (12.0%) | 0.01 | 220 (3.0%) | 224 (3.1%) | -0.01 | 1,034 (7.4%) | 1,029 (7.4%) | 0.00 |
| ICD10 ; n (%) | | | | | | | | | |
| Hypoglycemia ; n (%) | 56 (0.8%) | 40 (0.6%) | 0.02 | 97 (1.3%) | 91 (1.2%) | 0.01 | 0,153 (1.1%) | 0,131 (0.9%) | 0.02 |
| Hyperglycemia; n (%) | 600 (9.0%) | 604 (9.0%) | 0.00 | 444 (6.1%) | 442 (6.1%) | 0.00 | 1,044 (7.5%) | 1,046 (7.5%) | 0.00 |
| Disorders of fluid electrolyte and acid-base | 1,318 (19.7%) | 1,332 (19.9%) | -0.01 | 681 (9.4%) | 709 (9.7%) | -0.01 | 1,999 (14.3%) | 2,041 (14.6%) | -0.01 |
| balance; n (%) | | | | | | | | | |
| Diabetic ketoacidosis; n (%) | 43 (0.6%) | 35 (0.5%) | 0.01 | 45 (0.6%) | 43 (0.6%) | 0.00 | 88 (0.6%) | 78 (0.6%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK); n (%) | 31 (0.5%) | 32 (0.5%) | 0.00 | 12 (0.2%) | 12 (0.2%) | 0.00 | 43 (0.3%) | 44 (0.3%) | 0.00 |
| Diabetes with peripheral circulatory disorders with ICD-10; n (%) | 444 (6.6%) | 441 (6.6%) | 0.00 | 132 (1.8%) | 127 (1.7%) | 0.01 | 0,576 (4.1%) | 0,568 (4.1%) | 0.00 |
| Diabetic Foot; n (%) | 105 (1.6%) | 101 (1.5%) | 0.01 | 67 (0.9%) | 67 (0.9%) | 0.00 | 172 (1.2%) | 168 (1.2%) | 0.00 |
| Gangrene ; n (%) | 10 (0.1%) | 9 (0.1%) | 0.00 | 8 (0.1%) | 3 (0.0%) | 0.04 | 18 (0.1%) | 12 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 50 (0.7%) | 45 (0.7%) | 0.00 | 12 (0.2%) | 14 (0.2%) | 0.00 | 62 (0.4%) | 59 (0.4%) | 0.00 |
| Osteomyelitis; n (%) | 23 (0.3%) | 29 (0.4%) | -0.02 | 13 (0.2%) | 19 (0.3%) | -0.02 | 36 (0.3%) | 48 (0.3%) | 0.00 |
| Skin infections ; n (%) | 309 (4.6%) | 313 (4.7%) | 0.00 | 252 (3.5%) | 253 (3.5%) | 0.00 | 0,561 (4.0%) | 0,566 (4.0%) | 0.00 |
| Erectile dysfunction; n (%) | 208 (3.1%) | 216 (3.2%) | -0.01 | 182 (2.5%) | 179 (2.5%) | 0.00 | 0,390 (2.8%) | 0,395 (2.8%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 373 (5.6%) | 364 (5.4%) | 0.01 | 225 (3.1%) | 216 (3.0%) | 0.01 | 0,598 (4.3%) | 0,580 (4.1%) | 0.01 |
| , | 0.0 (0.0,0) | 55 (61.77) | | (====, | (3.37.7) | | 2,222 (11272) | 2,222 (**=/-1) | |
| Diabetes mellitus without mention of | 3,495 (52.2%) | 3,487 (52.1%) | 0.00 | 2,994 (41.1%) | 2,965 (40.7%) | 0.01 | 6,489 (46.4%) | 6,452 (46.2%) | 0.00 |
| complications; n (%) | 5 702 (D.C. 40() | 5 024 (06 00() | 0.04 | 5 642 (77 40/) | 5 647 /77 40() | 0.00 | 44 205 (04 50/) | 44 420 (04 00() | 0.04 |
| Hypertension: 1 inpatient or 2 outpatient | 5,783 (86.4%) | 5,821 (86.9%) | -0.01 | 5,612 (77.1%) | 5,617 (77.1%) | 0.00 | 11,395 (81.5%) | 11,438 (81.8%) | -0.01 |
| claims within 365 days; n (%) | E E02 (02 E0/) | E C22 (04 40/) | 0.02 | F 462 (70 00/) | F 4F0 /70 00/) | 0.00 | 40.754/76.00() | 40 702 (77 20/) | 0.01 |
| Hyperlipidemia ; n (%) | 5,592 (83.5%) | 5,633 (84.1%) | -0.02 | 5,162 (70.9%) | 5,159 (70.8%) | 0.00 | 10,754 (76.9%) | 10,792 (77.2%) | -0.01 |
| Edema; n (%) | 447 (6.7%) | 442 (6.6%) | 0.00 | 214 (2.9%) | 220 (3.0%) | -0.01 | 0,661 (4.7%) | 0,662 (4.7%) | 0.00 |
| Renal Dysfunction (non-diabetic); n (%) | 2,007 (30.0%) | 2,049 (30.6%) | -0.01 | 999 (13.7%) | 969 (13.3%) | 0.01 | 3,006 (21.5%) | 3,018 (21.6%) | 0.00 |
| Occurrence of acute renal disease; n (%) | 928 (13.9%) | 919 (13.7%) | 0.01 | 419 (5.8%) | 425 (5.8%) | 0.00 | 1347 (9.6%) | 1344 (9.6%) | 0.00 |
| Occurrence of chronic renal insufficiency; n (%) | 1,520 (22.7%) | 1,503 (22.4%) | 0.01 | 534 (7.3%) | 520 (7.1%) | 0.01 | 2,054 (14.7%) | 2,023 (14.5%) | 0.01 |
| Chronic kidney disease ; n (%) | 1,486 (22.2%) | 1,464 (21.9%) | 0.01 | 516 (7.1%) | 494 (6.8%) | 0.01 | 2,002 (14.3%) | 1,958 (14.0%) | 0.01 |
| CKD Stage 3-4; n (%) | 1,056 (15.8%) | 1,045 (15.6%) | 0.01 | 336 (4.6%) | 330 (4.5%) | 0.00 | 1,392 (10.0%) | 1,375 (9.8%) | 0.01 |
| Occurrence of hypertensive nephropathy; n (%) | 1,199 (17.9%) | 1,177 (17.6%) | 0.01 | 362 (5.0%) | 363 (5.0%) | 0.00 | 1561 (11.2%) | 1540 (11.0%) | 0.01 |
| Occurrence of miscellaneous renal insufficiency | 580 (8.7%) | 598 (8.9%) | -0.01 | 306 (4.2%) | 307 (4.2%) | 0.00 | 0,886 (6.3%) | 0,905 (6.5%) | -0.01 |
| ; n (%)<br>Glaucoma or cataracts ; n (%) | 4.046 (45.60() | 1.061 (15.00/) | 0.01 | 047/44 20/) | 700 (44 00/) | 0.01 | 1 962 /12 20/\ | 1 050 (12 20/) | 0.00 |
| Gladcoma or cataracts, if (70) | 1,046 (15.6%) | 1,061 (15.8%) | -0.01 | 817 (11.2%) | 798 (11.0%) | 0.01 | 1,863 (13.3%) | 1,859 (13.3%) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Foot ulcer; n (%) | 107 (1.6%) | 104 (1.6%) | 0.00 | 63 (0.9%) | 67 (0.9%) | 0.00 | 170 (1.2%) | 171 (1.2%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Bladder stones; n (%) | 13 (0.2%) | 8 (0.1%) | 0.03 | 9 (0.1%) | 8 (0.1%) | 0.00 | 22 (0.2%) | 16 (0.1%) | 0.03 |
| Kidney stones; n (%) | 218 (3.3%) | 207 (3.1%) | 0.01 | 127 (1.7%) | 120 (1.6%) | 0.01 | 0,345 (2.5%) | 0,327 (2.3%) | 0.01 |
| Urinary tract infections (UTIs); n (%) | 588 (8.8%) | 597 (8.9%) | 0.00 | 291 (4.0%) | 280 (3.8%) | 0.01 | 0,879 (6.3%) | 0,877 (6.3%) | 0.00 |
| Dipstick urinalysis; n (%) | 1,825 (27.3%) | 1,872 (28.0%) | -0.02 | 1,486 (20.4%) | 1,441 (19.8%) | 0.01 | 3,311 (23.7%) | 3,313 (23.7%) | 0.00 |
| Non-dipstick urinalysis; n (%) | 1,275 (19.0%) | 1,303 (19.5%) | -0.01 | 748 (10.3%) | 734 (10.1%) | 0.01 | 2,023 (14.5%) | 2,037 (14.6%) | 0.00 |
| Urine function test; n (%) | 148 (2.2%) | 152 (2.3%) | -0.01 | 116 (1.6%) | 132 (1.8%) | -0.02 | 0,264 (1.9%) | 0,284 (2.0%) | -0.01 |
| Cytology; n (%) | 69 (1.0%) | 83 (1.2%) | -0.02 | 25 (0.3%) | 32 (0.4%) | -0.02 | 94 (0.7%) | 115 (0.8%) | -0.01 |
| Cystos; n (%) | 102 (1.5%) | 103 (1.5%) | 0.00 | 57 (0.8%) | 36 (0.5%) | 0.04 | 159 (1.1%) | 139 (1.0%) | 0.01 |
| Other Covariates | ` ′ | , , | | , , | , , | | , , | ` , | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0,000 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 1,393 (20.8%) | 1,383 (20.7%) | 0.00 | 848 (11.6%) | 881 (12.1%) | -0.02 | 2,241 (16.0%) | 2,264 (16.2%) | -0.01 |
| Other arthritis, arthropathies and | 2,587 (38.6%) | 2,593 (38.7%) | 0.00 | 2,193 (30.1%) | 2,215 (30.4%) | -0.01 | 4,780 (34.2%) | 4,808 (34.4%) | 0.00 |
| musculoskeletal pain; n (%) | , , , | , , , | | , , , | , , , | | , , , | , , , | |
| Dorsopathies; n (%) | 1,774 (26.5%) | 1,745 (26.1%) | 0.01 | 1,480 (20.3%) | 1,469 (20.2%) | 0.00 | 3,254 (23.3%) | 3,214 (23.0%) | 0.01 |
| Fractures; n (%) | 206 (3.1%) | 195 (2.9%) | 0.01 | 132 (1.8%) | 137 (1.9%) | -0.01 | 0,338 (2.4%) | 0,332 (2.4%) | 0.00 |
| Falls ; n (%) | 255 (3.8%) | 255 (3.8%) | 0.00 | 73 (1.0%) | 66 (0.9%) | 0.01 | 328 (2.3%) | 321 (2.3%) | 0.00 |
| Osteoporosis; n (%) | 310 (4.6%) | 314 (4.7%) | 0.00 | 155 (2.1%) | 156 (2.1%) | 0.00 | 0,465 (3.3%) | 0,470 (3.4%) | -0.01 |
| Hyperthyroidism; n (%) | 33 (0.5%) | 45 (0.7%) | -0.03 | 22 (0.3%) | 22 (0.3%) | 0.00 | 55 (0.4%) | 67 (0.5%) | -0.01 |
| Hypothyroidism ; n (%) | 1,142 (17.1%) | 1,098 (16.4%) | 0.02 | 706 (9.7%) | 734 (10.1%) | -0.01 | 1,848 (13.2%) | 1,832 (13.1%) | 0.00 |
| Other disorders of thyroid gland; n (%) | 203 (3.0%) | 236 (3.5%) | -0.03 | 174 (2.4%) | 164 (2.3%) | 0.01 | 0,377 (2.7%) | 0,400 (2.9%) | -0.01 |
| Depression; n (%) | 779 (11.6%) | 782 (11.7%) | 0.00 | 449 (6.2%) | 458 (6.3%) | 0.00 | 1,228 (8.8%) | 1,240 (8.9%) | 0.00 |
| Anxiety; n (%) | 947 (14.1%) | 939 (14.0%) | 0.00 | 586 (8.0%) | 601 (8.3%) | -0.01 | 1,533 (11.0%) | 1,540 (11.0%) | 0.00 |
| SleepDisorder; n (%) | 301 (4.5%) | 316 (4.7%) | -0.01 | 466 (6.4%) | 439 (6.0%) | 0.02 | 0,767 (5.5%) | 0,755 (5.4%) | 0.00 |
| Dementia; n (%) | 292 (4.4%) | 303 (4.5%) | 0.00 | 112 (1.5%) | 119 (1.6%) | -0.01 | 404 (2.9%) | 422 (3.0%) | -0.01 |
| Delirium; n (%) | 162 (2.4%) | 155 (2.3%) | 0.01 | 65 (0.9%) | 67 (0.9%) | 0.00 | 227 (1.6%) | 222 (1.6%) | 0.00 |
| Psychosis; n (%) | 67 (1.0%) | 61 (0.9%) | 0.01 | 32 (0.4%) | 34 (0.5%) | -0.01 | 99 (0.7%) | 95 (0.7%) | 0.00 |
| Obesity; n (%) | 1,796 (26.8%) | 1,832 (27.4%) | -0.01 | 1,445 (19.8%) | 1,357 (18.6%) | 0.03 | 3,241 (23.2%) | 3,189 (22.8%) | 0.01 |
| Overweight; n (%) | 484 (7.2%) | 489 (7.3%) | 0.00 | 218 (3.0%) | 217 (3.0%) | 0.00 | 0,702 (5.0%) | 0,706 (5.1%) | 0.00 |
| Smoking; n (%) | 3,128 (46.7%) | 3,124 (46.6%) | 0.00 | 2,083 (28.6%) | 2,118 (29.1%) | -0.01 | 5,211 (37.3%) | 5,242 (37.5%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 152 (2.3%) | 159 (2.4%) | -0.01 | 108 (1.5%) | 114 (1.6%) | -0.01 | 260 (1.9%) | 273 (2.0%) | -0.01 |
| Drug abuse or dependence; n (%) | 195 (2.9%) | 188 (2.8%) | 0.01 | 91 (1.2%) | 94 (1.3%) | -0.01 | 286 (2.0%) | 282 (2.0%) | 0.00 |
| COPD; n (%) | 1,228 (18.3%) | 1,230 (18.4%) | 0.00 | 671 (9.2%) | 640 (8.8%) | 0.01 | 1,899 (13.6%) | 1,870 (13.4%) | 0.01 |
| Asthma; n (%) | 484 (7.2%) | 494 (7.4%) | -0.01 | 363 (5.0%) | 369 (5.1%) | 0.00 | 0,847 (6.1%) | 0,863 (6.2%) | 0.00 |
| Obstructive sleep apnea; n (%) | 770 (11.5%) | 783 (11.7%) | -0.01 | 630 (8.7%) | 612 (8.4%) | 0.01 | 1,400 (10.0%) | 1,395 (10.0%) | 0.00 |
| Pneumonia; n (%) | 425 (6.3%) | 456 (6.8%) | -0.02 | 198 (2.7%) | 219 (3.0%) | -0.02 | 0,623 (4.5%) | 0,675 (4.8%) | -0.01 |
| Imaging; n (%) | 211 (3.2%) | 203 (3.0%) | 0.01 | 80 (1.1%) | 101 (1.4%) | -0.03 | 291 (2.1%) | 304 (2.2%) | -0.01 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 3,488 (52.1%) | 3,508 (52.4%) | -0.01 | 4,129 (56.7%) | 4,130 (56.7%) | 0.00 | 7,617 (54.5%) | 7,638 (54.6%) | 0.00 |
| Use of ARBs; n (%) | 1,623 (24.2%) | 1,647 (24.6%) | -0.01 | 1,544 (21.2%) | 1,551 (21.3%) | 0.00 | 3,167 (22.7%) | 3,198 (22.9%) | 0.00 |
| Use of Loop Diuretics - ; n (%) | 1,034 (15.4%) | 1,025 (15.3%) | 0.00 | 580 (8.0%) | 588 (8.1%) | 0.00 | 1,614 (11.5%) | 1,613 (11.5%) | 0.00 |
| Use of other diuretics-; n (%) | 318 (4.7%) | 327 (4.9%) | -0.01 | 322 (4.4%) | 302 (4.1%) | 0.01 | 0,640 (4.6%) | 0,629 (4.5%) | 0.00 |
| Use of nitrates-; n (%) | 2,918 (43.6%) | 2,928 (43.7%) | 0.00 | 3,267 (44.9%) | 3,251 (44.6%) | 0.01 | 6,185 (44.2%) | 6,179 (44.2%) | 0.00 |
| Use of other hypertension drugs; n (%) | 518 (7.7%) | 509 (7.6%) | 0.00 | 352 (4.8%) | 353 (4.8%) | 0.00 | 0,870 (6.2%) | 0,862 (6.2%) | 0.00 |
| Use of digoxin- ; n (%) | 72 (1.1%) | 71 (1.1%) | 0.00 | 70 (1.0%) | 62 (0.9%) | 0.01 | 142 (1.0%) | 133 (1.0%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 178 (2.7%) | 204 (3.0%) | -0.02 | 159 (2.2%) | 154 (2.1%) | 0.01 | 337 (2.4%) | 358 (2.6%) | -0.01 |
| Use of COPD/asthma meds-; n (%) | 1,024 (15.3%) | 1,023 (15.3%) | 0.00 | 885 (12.2%) | 894 (12.3%) | 0.00 | 1,909 (13.7%) | 1,917 (13.7%) | 0.00 |
| Use of statins; n (%) | 6,026 (90.0%) | 6,037 (90.1%) | 0.00 | 6,668 (91.6%) | 6,661 (91.5%) | 0.00 | 12,694 (90.8%) | 12,698 (90.8%) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Use of other lipid-lowering drugs; n (%) | 504 (7.5%) | 511 (7.6%) | 0.00 | 660 (9.1%) | 658 (9.0%) | 0.00 | 1,164 (8.3%) | 1,169 (8.4%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Use of oral anticoagulants (Dabigatran, | 367 (5.5%) | 349 (5.2%) | 0.01 | 346 (4.8%) | 312 (4.3%) | 0.02 | 0,713 (5.1%) | 0,661 (4.7%) | 0.02 |
| Rivaroxaban, Apixaban, Warfarin); n (%) | | | | | | | | | |
| Use of heparin and other low-molecular weight | 37 (0.6%) | 41 (0.6%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 37 (0.3%) | 41 (0.3%) | 0.00 |
| heparins; n (%) | | | | | | | | | |
| Use of NSAIDs; n (%) | 997 (14.9%) | 1,014 (15.1%) | -0.01 | 1,127 (15.5%) | 1,115 (15.3%) | 0.01 | 2,124 (15.2%) | 2,129 (15.2%) | 0.00 |
| Use of oral corticosteroids; n (%) | 1,231 (18.4%) | 1,215 (18.1%) | 0.01 | 1,145 (15.7%) | 1,119 (15.4%) | 0.01 | 2,376 (17.0%) | 2,334 (16.7%) | 0.01 |
| Use of bisphosphonate (); n (%) | 113 (1.7%) | 108 (1.6%) | 0.01 | 69 (0.9%) | 64 (0.9%) | 0.00 | 182 (1.3%) | 172 (1.2%) | 0.01 |
| Use of opioids- ; n (%) | 1,663 (24.8%) | 1,668 (24.9%) | 0.00 | 1,603 (22.0%) | 1,582 (21.7%) | 0.01 | 3,266 (23.4%) | 3,250 (23.2%) | 0.00 |
| Use of antidepressants; n (%) | 1,356 (20.2%) | 1,338 (20.0%) | 0.00 | 1,158 (15.9%) | 1,165 (16.0%) | 0.00 | 2,514 (18.0%) | 2,503 (17.9%) | 0.00 |
| Use of antipsychotics; n (%) | 128 (1.9%) | 139 (2.1%) | -0.01 | 63 (0.9%) | 68 (0.9%) | 0.00 | 0,191 (1.4%) | 0,207 (1.5%) | -0.01 |
| Use of anticonvulsants; n (%) | 975 (14.6%) | 907 (13.5%) | 0.03 | 612 (8.4%) | 577 (7.9%) | 0.02 | 1,587 (11.4%) | 1,484 (10.6%) | 0.03 |
| Use of lithium- ; n (%) | 10 (0.1%) | 11 (0.2%) | -0.03 | 6 (0.1%) | 6 (0.1%) | 0.00 | 16 (0.1%) | 17 (0.1%) | 0.00 |
| Use of Benzos- ; n (%) | 792 (11.8%) | 764 (11.4%) | 0.01 | 761 (10.4%) | 742 (10.2%) | 0.01 | 1,553 (11.1%) | 1,506 (10.8%) | 0.01 |
| Use of anxiolytics/hypnotics-; n (%) | 310 (4.6%) | 306 (4.6%) | 0.00 | 399 (5.5%) | 381 (5.2%) | 0.01 | 0,709 (5.1%) | 0,687 (4.9%) | 0.01 |
| Use of dementia meds- ; n (%) | 118 (1.8%) | 121 (1.8%) | 0.00 | 60 (0.8%) | 59 (0.8%) | 0.00 | 178 (1.3%) | 180 (1.3%) | 0.00 |
| Use of antiparkinsonian meds-; n (%) | 154 (2.3%) | 147 (2.2%) | 0.01 | 100 (1.4%) | 103 (1.4%) | 0.00 | 0,254 (1.8%) | 0,250 (1.8%) | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 15 (0.2%) | 16 (0.2%) | 0.00 | 6 (0.1%) | 3 (0.0%) | 0.04 | 21 (0.2%) | 19 (0.1%) | 0.03 |
| Labs | (0, | () | | J (J. 17.7) | - (0.0, c) | | (*:=/-/ | == (====,=, | |
| Lab values- HbA1c (%) ; n (%) | 1,404 (21.0%) | 1,381 (20.6%) | 0.01 | 128 (1.8%) | 103 (1.4%) | 0.03 | 1,532 (11.0%) | 1,484 (10.6%) | 0.01 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 920 (13.7%) | 888 (13.3%) | 0.01 | 75 (1.0%) | 74 (1.0%) | 0.00 | 0,995 (7.1%) | 0,962 (6.9%) | 0.01 |
| 200 10.000 110.120 (70) (11.11111.0 11.1011.11.15) 11.1(70) | 323 (23.77) | 000 (20.070) | 0.02 | 75 (2.675) | 7 1 (21070) | 0.00 | 0,555 (7.1270) | 0,302 (0.370) | 0.01 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 1,404 (21.0%) | 1,381 (20.6%) | 0.01 | 128 (1.8%) | 103 (1.4%) | 0.03 | 1,532 (11.0%) | 1,484 (10.6%) | 0.01 |
| Lab values- BNP; n (%) | 87 (1.3%) | 74 (1.1%) | 0.02 | 10 (0.1%) | 2 (0.0%) | 0.04 | 97 (0.7%) | 76 (0.5%) | 0.03 |
| Lab values- BNP (within 3 months); n (%) | 72 (1.1%) | 53 (0.8%) | 0.03 | 7 (0.1%) | 1 (0.0%) | 0.04 | 79 (0.6%) | 54 (0.4%) | 0.03 |
| Lab values-BNP (within 6 months); n (%) | 87 (1.3%) | 74 (1.1%) | 0.02 | 10 (0.1%) | 2 (0.0%) | 0.04 | 97 (0.7%) | 76 (0.5%) | 0.03 |
| Lab values- BUN (mg/dl); n (%) | 1,874 (28.0%) | 1,893 (28.3%) | -0.01 | 126 (1.7%) | 116 (1.6%) | 0.01 | 2,000 (14.3%) | 2,009 (14.4%) | 0.00 |
| Lab values- BUN (mg/dl) (within 3 months); n<br>(%) | 1,255 (18.7%) | 1,255 (18.7%) | 0.00 | 75 (1.0%) | 72 (1.0%) | 0.00 | 1,330 (9.5%) | 1,327 (9.5%) | 0.00 |
| Lab values-BUN (mg/dl) (within 6 months); n<br>(%) | 1,874 (28.0%) | 1,893 (28.3%) | -0.01 | 126 (1.7%) | 116 (1.6%) | 0.01 | 2,000 (14.3%) | 2,009 (14.4%) | 0.00 |
| Lab values- Creatinine (mg/dl); n (%) | 1,936 (28.9%) | 1,945 (29.0%) | 0.00 | 140 (1.9%) | 125 (1.7%) | 0.02 | 2,076 (14.8%) | 2,070 (14.8%) | 0.00 |
| Lab values- Creatinine (mg/dl) (within 3 | 1,301 (19.4%) | 1,295 (19.3%) | 0.00 | 83 (1.1%) | 81 (1.1%) | 0.00 | 1,384 (9.9%) | 1,376 (9.8%) | 0.00 |
| months); n (%) | | | | | | | | | |
| Lab values- Creatinine (mg/dl) (within 6 | 1,936 (28.9%) | 1,945 (29.0%) | 0.00 | 140 (1.9%) | 125 (1.7%) | 0.02 | 2,076 (14.8%) | 2,070 (14.8%) | 0.00 |
| months); n (%) | | | | | | | | | |
| Lab values- HDL level (mg/dl); n (%) | 1,456 (21.7%) | 1,486 (22.2%) | -0.01 | 118 (1.6%) | 96 (1.3%) | 0.03 | 1,574 (11.3%) | 1,582 (11.3%) | 0.00 |
| Lab values- HDL level (mg/dl) (within 3 months); | 890 (13.3%) | 898 (13.4%) | 0.00 | 58 (0.8%) | 55 (0.8%) | 0.00 | 0,948 (6.8%) | 0,953 (6.8%) | 0.00 |
| n (%) | | | | | | | | | |
| Lab values- HDL level (mg/dl) (within 6 months);<br>n (%) | 1,456 (21.7%) | 1,486 (22.2%) | -0.01 | 118 (1.6%) | 96 (1.3%) | 0.03 | 1,574 (11.3%) | 1,582 (11.3%) | 0.00 |
| Lab values- LDL level (mg/dl); n (%) | 1,496 (22.3%) | 1,555 (23.2%) | -0.02 | 130 (1.8%) | 102 (1.4%) | 0.03 | 1,626 (11.6%) | 1,657 (11.9%) | -0.01 |
| Lab values- LDL level (mg/dl) (within 3 months); | 911 (13.6%) | 952 (14.2%) | -0.02 | 71 (1.0%) | 61 (0.8%) | 0.02 | 0,982 (7.0%) | 1,013 (7.2%) | -0.01 |
| n (%) | | | | | | | | | |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 1,496 (22.3%) | 1,555 (23.2%) | -0.02 | 130 (1.8%) | 102 (1.4%) | 0.03 | 1,626 (11.6%) | 1,657 (11.9%) | -0.01 |
| Lab values- NT-proBNP; n (%) | 12 (0.2%) | 11 (0.2%) | 0.00 | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 12 (0.1%) | 12 (0.1%) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Lab values- NT-proBNP (within 3 months); n (%) | 10 (0.1%) | 7 (0.1%) | 0.00 | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 10 (0.1%) | 8 (0.1%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- NT-proBNP (within 6 months); n (%) | 12 (0.2%) | 11 (0.2%) | 0.00 | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 12 (0.1%) | 12 (0.1%) | 0.00 |
| Lab values-Total cholesterol (mg/dl); n (%) | 1,480 (22.1%) | 1,514 (22.6%) | -0.01 | 116 (1.6%) | 98 (1.3%) | 0.03 | 1,596 (11.4%) | 1,612 (11.5%) | 0.00 |
| Lab values- Total cholesterol (mg/dl) (within 3 months); n (%) | 899 (13.4%) | 912 (13.6%) | -0.01 | 58 (0.8%) | 55 (0.8%) | 0.00 | 0,957 (6.8%) | 0,967 (6.9%) | 0.00 |
| Lab values-Total cholesterol (mg/dl) (within 6 months); n (%) | 1,480 (22.1%) | 1,514 (22.6%) | -0.01 | 116 (1.6%) | 98 (1.3%) | 0.03 | 1,596 (11.4%) | 1,612 (11.5%) | 0.00 |
| Lab values-Triglyceride level (mg/dl); n (%) | 1,453 (21.7%) | 1,500 (22.4%) | -0.02 | 117 (1.6%) | 94 (1.3%) | 0.03 | 1,570 (11.2%) | 1,594 (11.4%) | -0.01 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n (%) | 881 (13.2%) | 906 (13.5%) | -0.01 | 57 (0.8%) | 54 (0.7%) | 0.01 | 0,938 (6.7%) | 0,960 (6.9%) | -0.01 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n (%) | 1,453 (21.7%) | 1,500 (22.4%) | -0.02 | 117 (1.6%) | 94 (1.3%) | 0.03 | 1,570 (11.2%) | 1,594 (11.4%) | -0.01 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 1,398 | 1,379 | | 123 | 100 | | 0 | 0 | |
| mean (sd) | 7.29 (1.75) | 7.27 (1.76) | 0.01 | 8.14 (1.81) | 7.66 (1.81) | 0.27 | 7.73 (1.78) | 7.47 (1.79) | 0.15 |
| median [IQR] | 6.90 [6.00, 8.10] | 6.75 [6.00, 8.00] | 0.09 | 8.00 [6.80, 9.20] | 7.18 [6.20, 8.95] | 0.45 | 7.47 (1.78) | 6.97 (1.79) | 0.28 |
| Missing; n (%) | 5,299 (79.1%) | 5,318 (79.4%) | -0.01 | 7,160 (98.3%) | 7,183 (98.6%) | -0.02 | 12,459 (89.1%) | 12,501 (89.4%) | -0.01 |
| Lab result number- BNP mean | 87 | 74 | | 10 | 2 | | 0 | 0 | |
| mean (sd) | 381.53 (1,230.47) | 345.14 (679.13) | 0.04 | 383.62 (605.09) | 334.50 (0.71) | 0.11 | 382.62 (957.10) | 339.60 (470.04) | 0.06 |
| median [IQR] | 94.00 [42.00, | 94.50 [44.42, | 0.00 | 163.00 [86.75, | 334.50 [334.00, | -0.40 | 129.95 (957.10) | 219.53 (470.04) | -0.12 |
| rearan [rear] | 253.00] | 276.17] | 0.00 | 463.25] | 335.00] | 0.40 | 123.33 (337.10) | 213.33 (470.04) | 0.12 |
| Missing; n (%) | 6,610 (98.7%) | 6,623 (98.9%) | -0.02 | 7,273 (99.9%) | 7,281 (100.0%) | -0.04 | 13,883 (99.3%) | 13,904 (99.5%) | -0.03 |
| Lab result number- BUN (mg/dl) mean | 1,874 | 1,893 | 0.02 | 126 | 116 | 0.04 | 0 | 0 | 0.03 |
| mean (sd) | 18.97 (8.52) | 18.95 (7.66) | 0.00 | 1,128.51<br>(12,470.63) | 3,361.89<br>(21,189.20) | -0.13 | 596.99 (9001.01) | 1760.48 (15293.87) | -0.09 |
| median [IQR] | 17.00 [14.00, 22.00] | 17.00 [14.00, 22.00] | 0.00 | 17.00 [14.00,<br>20.75] | 17.00 [14.00,<br>21.00] | 0.00 | 17.00 (9001.01) | 17.00 (15293.87) | 0.00 |
| Missing; n (%) | 4,823 (72.0%) | 4,804 (71.7%) | 0.01 | 7,157 (98.3%) | 7,167 (98.4%) | -0.01 | 11,980 (85.7%) | 11,971 (85.6%) | 0.00 |
| Lab result number- Creatinine (mg/dl) mean | 1,913 | 1,927 | | 121 | 103 | | 2,034 | 2,030 | |
| (only 0.1 to 15 included) | _,==== | _, | | | | | _,,,, | _,,,,, | |
| mean (sd) | 1.09 (0.45) | 1.08 (0.40) | 0.02 | 1.01 (0.23) | 1.00 (0.24) | 0.04 | 1.05 (0.35) | 1.04 (0.33) | 0.03 |
| median [IQR] | 1.00 [0.84, 1.21] | 1.00 [0.84, 1.22] | 0.00 | 1.00 [0.86, 1.13] | 1.00 [0.88, 1.12] | 0.00 | 1.00 (0.35) | 1.00 (0.33) | 0.00 |
| Missing; n (%) | 4,784 (71.4%) | 4,770 (71.2%) | 0.00 | 7,162 (98.3%) | 7,180 (98.6%) | -0.02 | 11,946 (85.5%) | 11,950 (85.5%) | 0.00 |
| Lab result number- HDL level (mg/dl) mean (only =<5000 included) | 1,456 | 1,486 | | 117 | 96 | | 1,573 | 1,582 | |
| mean (sd) | 46.40 (14.74) | 46.63 (14.02) | -0.02 | 41.80 (11.50) | 42.00 (12.11) | -0.02 | 44.00 (13.15) | 44.22 (13.06) | -0.02 |
| median [IQR] | 44.00 [36.00, 54.00] | | 0.00 | 41.00 [33.50,<br>48.50] | 41.00 [35.25,<br>48.00] | 0.00 | 42.44 (13.15) | 42.44 (13.06) | 0.00 |
| Missing; n (%) | 5,241 (78.3%) | 5,211 (77.8%) | 0.01 | 7,166 (98.4%) | 7,187 (98.7%) | -0.03 | 12,407 (88.7%) | 12,398 (88.7%) | 0.00 |
| Lab result number-LDL level (mg/dl) mean (only =<5000 included) | | 1,522 | | 111 | 89 | | 1,574 | 1,611 | |
| mean (sd) | 101.93 (45.14) | 103.69 (43.77) | -0.04 | 101.62 (50.86) | 96.09 (46.22) | 0.11 | 101.77 (48.20) | 99.73 (45.06) | 0.04 |
| median [IQR] | 101.00 [75.00,<br>128.00] | 100.00 [75.00,<br>131.00] | 0.02 | 99.00 [69.00,<br>134.50] | 104.50 [61.00,<br>129.00] | -0.11 | 99.96 (48.20) | 102.34 (45.06) | -0.05 |
| Missing; n (%) | 5,234 (78.2%) | 5,175 (77.3%) | 0.02 | 7,172 (98.5%) | 7,194 (98.8%) | -0.03 | 12,406 (88.7%) | 12,369 (88.5%) | 0.01 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included) | 1,476 | 1,510 | | 115 | 97 | | 1,591 | 1,607 | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 188.01 (53.70) | 187.17 (49.11) | 0.02 | 190.24 (53.63) | 187.50 (45.93) | 0.05 | 189.17 (53.66) | 187.34 (47.48) | 0.04 |
| median [IQR] | 183.00 [153.00,<br>214.00] | 182.00 [154.00,<br>216.00] | 0.02 | 197.00 [148.50,<br>230.00] | 186.00 [156.50,<br>219.25] | 0.22 | 190.29 (53.66) | 184.08 (47.48) | 0.12 |
| Missing; n (%) | 5,221 (78.0%) | 5,187 (77.5%) | 0.01 | 7,168 (98.4%) | 7,186 (98.7%) | -0.03 | 12,389 (88.6%) | 12,373 (88.5%) | 0.00 |
| Lab result number-Triglyceride level (mg/dl)<br>mean (only =<5000 included) | 1,450 | 1,500 | | 116 | 93 | | 1,566 | 1,593 | |
| mean (sd) | 178.04 (146.67) | 171.98 (120.25) | 0.05 | 191.07 (122.18) | 207.13 (136.39) | -0.12 | 184.83 (134.47) | 190.29 (128.91) | -0.04 |
| median [IQR] | 143.00 [104.00,<br>209.25] | 143.50 [104.00,<br>203.88] | 0.00 | 163.50 [103.12,<br>239.50] | 165.00 [122.00,<br>245.00] | -0.01 | 153.68 (134.47) | 154.70 (128.91) | -0.01 |
| Missing; n (%) | 5,247 (78.3%) | 5,197 (77.6%) | 0.02 | 7,167 (98.4%) | 7,190 (98.7%) | -0.03 | 12,414 (88.8%) | 12,387 (88.6%) | 0.01 |
| Lab result number- Hemoglobin mean (only >0 included) | 1,451 | 1,430 | | 97 | 75 | | 1,548 | 1,505 | |
| mean (sd) | 13.81 (1.81) | 13.82 (1.78) | -0.01 | 13.82 (2.15) | 135,417.06<br>(1,154,595.69) | -0.17 | 13.82 (1.99) | 70553.29<br>(833360.19) | -0.12 |
| median [IQR] | 13.90 [12.60, 15.10] | 14.00 [12.60, 15.01] | -0.06 | 14.00 [12.80,<br>15.30] | 14.10 [13.00,<br>15.00] | 0.00 | 13.95 (1.99) | 14.05 (833360.19) | 0.00 |
| Missing; n (%) | 5,246 (78.3%) | 5,267 (78.6%) | -0.01 | 7,186 (98.7%) | 7,208 (99.0%) | -0.03 | 12,432 (88.9%) | 12,475 (89.2%) | -0.01 |
| Lab result number- Serum sodium mean (only > 90 and < 190 included) | 1,869 | 1,891 | | 133 | 111 | | 2,002 | 2,002 | |
| mean (sd) | 139.98 (2.88) | 140.05 (2.79) | -0.02 | 138.91 (2.64) | 139.51 (2.55) | -0.23 | 139.42 (2.76) | 139.77 (2.67) | -0.13 |
| median [IQR] | 140.00 [138.33,<br>142.00] | 140.00 [138.50,<br>142.00] | 0.00 | 139.00 [137.00,<br>141.00] | 140.00 [138.00,<br>141.00] | -0.39 | 139.48 (2.76) | 140.00 (2.67) | -0.19 |
| Missing; n (%) | 4,828 (72.1%) | 4,806 (71.8%) | 0.01 | 7,150 (98.2%) | 7,172 (98.5%) | -0.02 | 11,978 (85.7%) | 11,978 (85.7%) | 0.00 |
| Lab result number- Albumin mean (only >0 and <=10 included) | 1,708 | 1,714 | | 115 | 94 | | 1,823 | 1,808 | |
| mean (sd) | 4.19 (0.35) | 4.20 (0.34) | -0.03 | 4.11 (0.54) | 4.04 (0.45) | 0.14 | 4.15 (0.46) | 4.12 (0.40) | 0.07 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.10 [4.00, 4.40] | 4.00 [4.00, 4.40] | 0.20 | 4.15 (0.46) | 4.10 (0.40) | 0.12 |
| Missing; n (%) | 4,989 (74.5%) | 4,983 (74.4%) | 0.00 | 7,168 (98.4%) | 7,189 (98.7%) | -0.03 | 12,157 (87.0%) | 12,172 (87.1%) | 0.00 |
| Lab result number-Glucose (fasting or random) mean (only 10-1000 included) | 1,858 | 1,885 | | 133 | 113 | | 1,991 | 1,998 | |
| mean (sd) | 135.97 (63.19) | 134.68 (61.29) | 0.02 | 167.91 (62.54) | 152.10 (61.99) | 0.25 | 152.61 (62.85) | 143.76 (61.66) | 0.14 |
| median [IQR] | 114.00 [96.00,<br>156.00] | 113.00 [97.00,<br>151.00] | 0.02 | 153.00 [119.50,<br>202.00] | 139.00 [110.33,<br>179.80] | 0.22 | 134.32 (62.85) | 126.54 (61.66) | 0.12 |
| Missing; n (%) | 4,839 (72.3%) | 4,812 (71.9%) | 0.01 | 7,150 (98.2%) | 7,170 (98.4%) | -0.02 | 11,989 (85.8%) | 11,982 (85.7%) | 0.00 |
| Lab result number- Potassium mean (only 1-7 included) | 1,914 | 1,926 | | 124 | 108 | | 2,038 | 2,034 | |
| mean (sd) | 4.44 (0.44) | 4.46 (0.44) | -0.05 | 4.29 (0.48) | 4.16 (0.44) | 0.28 | 4.36 (0.46) | 4.30 (0.44) | 0.13 |
| median [IQR] | 4.40 [4.15, 4.70] | 4.40 [4.20, 4.70] | 0.00 | 4.29 [4.00, 4.60] | 4.10 [4.00, 4.40] | 0.41 | 4.34 (0.46) | 4.24 (0.44) | 0.22 |
| Missing; n (%) | 4,783 (71.4%) | 4,771 (71.2%) | 0.00 | 7,159 (98.3%) | 7,175 (98.5%) | -0.02 | 11,942 (85.4%) | 11,946 (85.5%) | 0.00 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 3.71 (2.43) | 3.71 (2.43) | 0.00 | 2.24 (1.64) | 2.24 (1.64) | 0.00 | 2.94 (2.06) | 2.94 (2.06) | 0.00 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 2.48 (2.06) | 2.48 (2.06) | 0.00 |
| Frailty Score (mean): Empirical Version 365 | | | | | | | | | |
| days, | | | | | | | | | |
| mean (sd) | 0.20 (0.05) | 0.20 (0.05) | 0.00 | 0.18 (0.04) | 0.18 (0.04) | 0.00 | 0.19 (0.05) | 0.19 (0.05) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| median [IQR] Healthcare Utilization | 0.19 [0.16, 0.22] | 0.19 [0.16, 0.22] | 0.00 | 0.17 [0.15, 0.19] | 0.17 [0.15, 0.19] | 0.00 | 0.18 (0.05) | 0.18 (0.05) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization; n (%) | 6,686 (99.8%) | 6,690 (99.9%) | -0.03 | 7,283 (100.0%) | 7,283 (100.0%) | #DIV/0! | 13,969 (99.9%) | 13,973 (99.9%) | 0.00 |
| Any hospitalization during prior 31-180 days; n | ' ' ' | 411 (6.1%) | -0.05 | 176 (2.4%) | 192 (2.6%) | -0.01 | 0,512 (3.7%) | 0,603 (4.3%) | -0.03 |
| (%) | 333 (3.074) | (0.170) | 0.00 | 170 (21170) | 132 (2.070) | 0.01 | 0,012 (0.770) | 0,000 (110,0) | 0.00 |
| Endocrinologist Visit; n (%) | 464 (6.9%) | 450 (6.7%) | 0.01 | 405 (5.6%) | 390 (5.4%) | 0.01 | 0,869 (6.2%) | 0,840 (6.0%) | 0.01 |
| Endocrinologist Visit (30 days prior); n (%) | 239 (3.6%) | 227 (3.4%) | 0.01 | 198 (2.7%) | 210 (2.9%) | -0.01 | 0,437 (3.1%) | 0,437 (3.1%) | 0.00 |
| | | (•, | | | (, | | 0,101 (012,1) | 0,101 (012/1) | |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 294 (4.4%) | 294 (4.4%) | 0.00 | 253 (3.5%) | 234 (3.2%) | 0.02 | 0,547 (3.9%) | 0,528 (3.8%) | 0.01 |
| Internal medicine/family medicine visits; n (%) | 5,736 (85.7%) | 5,717 (85.4%) | 0.01 | 5,239 (71.9%) | 5,227 (71.8%) | 0.00 | 10,975 (78.5%) | 10,944 (78.3%) | 0.00 |
| Internal medicine/family medicine visits (30 days prior); n (%) | 4,788 (71.5%) | 4,783 (71.4%) | 0.00 | 3,320 (45.6%) | 3,241 (44.5%) | 0.02 | 8,108 (58.0%) | 8,024 (57.4%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 days prior); n (%) | 4,341 (64.8%) | 4,335 (64.7%) | 0.00 | 4,170 (57.3%) | 4,231 (58.1%) | -0.02 | 8,511 (60.9%) | 8,566 (61.3%) | -0.01 |
| Cardiologist visit; n (%) | 6,365 (95.0%) | 6,231 (93.0%) | 0.08 | 2,849 (39.1%) | 2,776 (38.1%) | 0.02 | 9,214 (65.9%) | 9,007 (64.4%) | 0.03 |
| Number of Cardiologist visits (30 days prior); n | 6,321 (94.4%) | 6,192 (92.5%) | 0.08 | 2,372 (32.6%) | 2,275 (31.2%) | 0.03 | 8,693 (62.2%) | 8,467 (60.6%) | 0.03 |
| (%) | | | | | | | | | |
| Number of Cardiologist visits (31 to 180 days prior); n (%) | 1,442 (21.5%) | 1,466 (21.9%) | -0.01 | 923 (12.7%) | 952 (13.1%) | -0.01 | 2,365 (16.9%) | 2,418 (17.3%) | -0.01 |
| Electrocardiogram ; n (%) | 6,294 (94.0%) | 6,275 (93.7%) | 0.01 | 4,153 (57.0%) | 4,022 (55.2%) | 0.04 | 10,447 (74.7%) | 10,297 (73.7%) | 0.02 |
| Use of glucose test strips; n (%) | 121 (1.8%) | 127 (1.9%) | -0.01 | 106 (1.5%) | 102 (1.4%) | 0.01 | 0,227 (1.6%) | 0,229 (1.6%) | 0.00 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 10.48 (5.17) | 10.46 (5.10) | 0.00 | 9.41 (4.44) | 9.33 (4.38) | 0.02 | 9.92 (4.80) | 9.87 (4.74) | 0.01 |
| median [IQR] | 10.00 [7.00, 13.00] | 10.00 [7.00, 13.00] | 0.00 | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 9.48 (4.80) | 9.48 (4.74) | 0.00 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 1.13 (0.42) | 1.13 (0.44) | 0.00 | 1.06 (0.27) | 1.06 (0.27) | 0.00 | 1.09 (0.35) | 1.09 (0.36) | 0.00 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.35) | 1.00 (0.36) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 4.37 (3.32) | 4.42 (3.60) | -0.01 | 3.62 (2.00) | 3.64 (2.13) | -0.01 | 3.98 (2.71) | 4.01 (2.93) | -0.01 |
| median [IQR] | 3.00 [3.00, 5.00] | 3.00 [3.00, 5.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 (2.71) | 3.00 (2.93) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 1.18 (1.53) | 1.19 (1.76) | -0.01 | 3.37 (5.61) | 3.33 (5.97) | 0.01 | 2.32 (4.19) | 2.30 (4.48) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 0.00 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.00 | 1.52 (4.19) | 1.52 (4.48) | 0.00 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 4.04 (3.89) | 4.00 (3.76) | 0.01 | 3.12 (3.28) | 3.09 (3.24) | 0.01 | 3.56 (3.59) | 3.53 (3.50) | 0.01 |
| median [IQR] | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 0.00 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.00 | 2.48 (3.59) | 2.48 (3.50) | 0.00 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.29 (1.73) | 0.30 (1.91) | -0.01 | 0.22 (1.30) | 0.23 (1.48) | -0.01 | 0.68 (1.41) | 0.69 (1.62) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.48 (1.41) | 0.48 (1.62) | 0.00 |
| Number of internal medicine/family medicine | | | | | | | | | |
| visits | | | | | | | | | |
| mean (sd) | 9.83 (13.95) | 9.77 (13.26) | 0.00 | 4.68 (7.55) | 4.58 (7.32) | 0.01 | 7.15 (11.09) | 7.07 (10.59) | 0.01 |
| median [IQR] | 6.00 [2.00, 12.00] | 6.00 [2.00, 12.00] | 0.00 | 2.00 [0.00, 6.00] | 2.00 [0.00, 6.00] | 0.00 | 3.92 (11.09) | 3.92 (10.59) | 0.00 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Number of Cardiologist visits | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 9.71 (7.61) | 9.65 (6.80) | 0.01 | 1.28 (2.49) | 1.30 (2.66) | -0.01 | 5.32 (5.57) | 5.30 (5.08) | 0.00 |
| median [IQR] | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 4.31 (5.57) | 4.31 (5.08) | 0.00 |
| Number electrocardiograms received | | | | | | | | | |
| mean (sd) | 3.62 (3.22) | 3.57 (3.02) | 0.02 | 1.13 (1.46) | 1.10 (1.48) | 0.02 | 2.32 (2.47) | 2.28 (2.35) | 0.02 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.96 (2.47) | 1.96 (2.35) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 0.56 (0.81) | 0.55 (0.79) | 0.01 | 0.34 (0.66) | 0.32 (0.63) | 0.03 | 0.45 (0.74) | 0.43 (0.71) | 0.03 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.74) | 0.00 (0.71) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.27 (1.06) | 0.31 (2.85) | -0.02 | 0.14 (0.58) | 0.16 (0.99) | -0.02 | 0.20 (0.84) | 0.23 (2.10) | -0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.84) | 0.00 (2.10) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.61 (0.81) | 0.61 (0.80) | 0.00 | 0.44 (0.88) | 0.43 (0.85) | 0.01 | 0.52 (0.85) | 0.52 (0.83) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.85) | 0.00 (0.83) | 0.00 |
| Number of creatinine tests ordered | | - · · | | | - · · | | , , | . , | |
| mean (sd) | 0.06 (0.29) | 0.06 (0.34) | 0.00 | 0.04 (0.24) | 0.04 (0.23) | 0.00 | 0.05 (0.27) | 0.05 (0.29) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.27) | 0.00 (0.29) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.03 (0.22) | 0.04 (0.27) | -0.04 | 0.02 (0.16) | 0.02 (0.17) | 0.00 | 0.02 (0.19) | 0.03 (0.22) | -0.05 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.19) | 0.00 (0.22) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | | | |
| mean (sd) | 0.33 (0.81) | 0.33 (0.81) | 0.00 | 0.17 (0.58) | 0.15 (0.54) | 0.04 | 0.25 (0.70) | 0.24 (0.68) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.70) | 0.00 (0.68) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the | | | | | | | , , | | |
| 3rd digit level | | | | | | | | | |
| mean (sd) | 13.25 (11.46) | 13.42 (11.51) | -0.01 | 7.61 (8.40) | 7.68 (8.58) | -0.01 | 10.31 (9.98) | 10.43 (10.09) | -0.01 |
| median [IQR] | 12.00 [4.00, 19.00] | 12.00 [4.00, 20.00] | 0.00 | 4.00 [0.00, 14.00] | 4.00 [0.00, 14.00] | 0.00 | 7.83 (9.98) | 7.83 (10.09) | 0.00 |
| For PS | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | 155 (2.3%) | 163 (2.4%) | -0.01 | 78 (1.1%) | 77 (1.1%) | 0.00 | 233 (1.7%) | 240 (1.7%) | 0.00 |
| disease+Cerebrovascular procedure (for PS); n | | | | | | | | | |
| (%) | | | | | | | | | |
| Occurrence of creatinine tests ordered (for PS); | 299 (4.5%) | 291 (4.3%) | 0.01 | 204 (2.8%) | 211 (2.9%) | -0.01 | 0,503 (3.6%) | 0,502 (3.6%) | 0.00 |
| n (%) | | | | | | | | | |
| Occurrence of BUN tests ordered (for PS); n (%) | 168 (2.5%) | 167 (2.5%) | 0.00 | 115 (1.6%) | 117 (1.6%) | 0.00 | 0,283 (2.0%) | 0,284 (2.0%) | 0.00 |
| Occurrence of chronic renal insufficiency w/o | 704 (10.5%) | 682 (10.2%) | 0.01 | 244 (3.4%) | 229 (3.1%) | 0.02 | 0,948 (6.8%) | 0,911 (6.5%) | 0.01 |
| CKD (for PS) ; n (%) | | | | | | | | | |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 290 (4.3%) | 267 (4.0%) | 0.02 | 72 (1.0%) | 72 (1.0%) | 0.00 | 362 (2.6%) | 339 (2.4%) | 0.01 |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 1,070 (16.0%) | 1,060 (15.8%) | 0.01 | 340 (4.7%) | 337 (4.6%) | 0.00 | 1,410 (10.1%) | 1,397 (10.0%) | 0.00 |
| Bladder stones+Kidney stones (for PS); n (%) | 224 (3.3%) | 209 (3.1%) | 0.01 | 133 (1.8%) | 122 (1.7%) | 0.01 | 0,357 (2.6%) | 0,331 (2.4%) | 0.01 |
| Dish standith a sigh and signal stand | 464 (6.00() | 454(5,00%) | 0.00 | 4.47 (2.00/) | 1.4.4 (2.00() | 0.00 | 0.644./4.40/3 | 0.000 (4.30() | 0.00 |
| Diabetes with peripheral circulatory disorders+Gangrene+Osteomyelitis(for PS) with | 464 (6.9%) | 464 (6.9%) | 0.00 | 147 (2.0%) | 144 (2.0%) | 0.00 | 0,611 (4.4%) | 0,608 (4.3%) | 0.00 |
| ICD10; n (%) | | | | | | | | | |
| 10010,11(/0) | | | | | | | | | |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| Alcohol abuse or dependence+Drug abuse or dependence (for PS); n (%) | 331 (4.9%) | 334 (5.0%) | 0.00 | 186 (2.6%) | 200 (2.7%) | -0.01 | 517 (3.7%) | 534 (3.8%) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Diabetes with other ophthalmic<br>manifestations+Retinal detachment, vitreous<br>hemorrhage, vitrectomy+Retinal laser<br>coagulation therapy (for PS); n (%) | 67 (1.0%) | 70 (1.0%) | 0.00 | 106 (1.5%) | 99 (1.4%) | 0.01 | 0,173 (1.2%) | 0,169 (1.2%) | 0.00 |
| Other atherosclerosis+Cardiac conduction disorders+Other CVD (for PS); n (%) | 3,094 (46.2%) | 3,129 (46.7%) | -0.01 | 2,466 (33.9%) | 2,510 (34.5%) | -0.01 | 5,560 (39.8%) | 5,639 (40.3%) | -0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA (for PS); n (%) | 6,322 (94.4%) | 6,349 (94.8%) | -0.02 | 6,693 (91.9%) | 6,665 (91.5%) | 0.01 | 13,015 (93.1%) | 13,014 (93.1%) | 0.00 |
| Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland (for PS); n (%) | 1,250 (18.7%) | 1,239 (18.5%) | 0.01 | 816 (11.2%) | 838 (11.5%) | -0.01 | 2,066 (14.8%) | 2,077 (14.9%) | 0.00 |
| Delirium + Psychosis (for PS); n (%) | 213 (3.2%) | 202 (3.0%) | 0.01 | 92 (1.3%) | 91 (1.2%) | 0.01 | 305 (2.2%) | 293 (2.1%) | 0.01 |
| Any use of Meglitinides (for PS); n (%) | 23 (0.3%) | 21 (0.3%) | 0.00 | 18 (0.2%) | 29 (0.4%) | -0.04 | 41 (0.3%) | 50 (0.4%) | -0.02 |
| Any use of AGIs (for PS); n (%) | 9 (0.1%) | 7 (0.1%) | 0.00 | 2,466 (33.9%) | 2,510 (34.5%) | -0.01 | 5,560 (39.8%) | 5,639 (40.3%) | -0.01 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 1,070 (16.0%) | 1,060 (15.8%) | 0.01 | 340 (4.7%) | 337 (4.6%) | 0.00 | 1,410 (10.1%) | 1,397 (10.0%) | 0.00 |
| Use of thiazide; n (%) | 654 (9.8%) | 645 (9.6%) | 0.01 | 604 (8.3%) | 592 (8.1%) | 0.01 | 12,367 (88.5%) | 12,391 (88.6%) | 0.00 |
| Use of beta blockers; n (%) | 5,881 (87.8%) | 5,895 (88.0%) | -0.01 | 6,486 (89.1%) | 6,496 (89.2%) | 0.00 | 3,384 (24.2%) | 3,397 (24.3%) | 0.00 |
| Use of calcium channel blockers; n (%) | 1,824 (27.2%) | 1,833 (27.4%) | 0.00 | 1,560 (21.4%) | 1,564 (21.5%) | 0.00 | 4,418 (31.6%) | 4,404 (31.5%) | 0.00 |
| All antidiabetic medications except Insulin; n (%) | 2,329 (34.8%) | 2,328 (34.8%) | 0.00 | 2,089 (28.7%) | 2,076 (28.5%) | 0.00 | 1,258 (9.0%) | 1,237 (8.8%) | 0.01 |
| DM Medications - Insulin ; n (%) | 1,033 (15.4%) | 988 (14.8%) | 0.02 | 917 (12.6%) | 873 (12.0%) | 0.02 | 1,950 (13.9%) | 1,861 (13.3%) | 0.02 |
| Use of Low Intensity Statins; n (%) | 1,915 (28.6%) | 1,953 (29.2%) | -0.01 | 2,002 (27.5%) | 2,035 (27.9%) | -0.01 | 3917 (28.0%) | 3,988 (28.5%) | -0.01 |
| Use of High Intensity Statins; n (%) | 4,845 (72.3%) | 5,032 (75.1%) | -0.06 | 5,324 (73.1%) | 5,519 (75.8%) | -0.06 | 10169 (72.7%) | 10,551 (75.5%) | -0.06 |
| Malignant hypertension; n (%) | 283 (4.2%) | 317 (4.7%) | -0.02 | 2,690 (36.9%) | 2,670 (36.7%) | 0.00 | 2973 (21.3%) | 2,987 (21.4%) | 0.00 |
| Cardiovascular stress test; n (%) | 19 (0.3%) | 18 (0.3%) | 0.00 | 14 (0.2%) | 17 (0.2%) | 0.00 | 0,033 (0.2%) | 35 (0.3%) | -0.02 |
| Echocardiogram; n (%) | 5,122 (76.5%) | 5,169 (77.2%) | -0.02 | 5,207 (71.5%) | 5,195 (71.3%) | 0.00 | 10,329 (73.9%) | 10364 (74.1%) | 0.00 |
| Number of BNP tests | | | | | | | | | |
| mean (sd) | 0.11 (0.43) | 0.12 (0.45) | -0.02 | 0.13 (0.42) | 0.12 (0.38) | 0.02 | 0.12 (0.42) | 0.12 (0.42) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.42) | 0.00 (0.42) | 0.00 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.61 (1.83) | 0.60 (1.85) | 0.01 | 0.68 (1.49) | 0.66 (1.59) | 0.01 | 0.65 (1.66) | 0.63 (1.72) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.66) | 0.00 (1.72) | 0.00 |
| Number of Ambulatory Blood pressure | | | | | | | | | |
| monitoring tests | | | | | | | | | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| N of days on antihypertensive medications | | | | | | | | | |
| during baseline | | | | | | | | | |
| mean (sd) | 100.13 (78.50) | 101.32 (78.10) | -0.02 | 85.98 (79.37) | 85.78 (79.72) | 0.00 | 92.76 (78.95) | 93.22 (78.95) | -0.01 |
| median [IQR] | 135.00 [1.00,<br>178.00] | 137.00 [1.00,<br>178.00] | -0.03 | 89.00 [1.00,<br>173.00] | 88.00 [1.00,<br>174.00] | 0.01 | 111.04 (78.95) | 111.47 (78.95) | -0.01 |
| N of days in database anytime prior | - | | | | | | | | |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| mean (sd) | 1,800.74 (1,442.20) | 1,791.98 (1,450.03) | 0.01 | 2,250.83 | 2,264.37 | -0.01 | 2035.22 (1464.32) | 2038.08 (1467.96) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| . , | | | | (1,484.36) | (1,484.25) | | | | |
| median [IQR] | 1,342.00 [646.00,<br>2,614.00] | 1,327.00 [641.50,<br>2,621.50] | 0.01 | 1,996.00 [941.00,<br>3,521.00] | 1,990.00 [966.00,<br>3,538.00] | 0.00 | 1682.71 (1464.32) | 1672.40 (1467.96) | 0.01 |
| Mean Copay for per prescription cost (charges | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , | | .,. | .,, | | | | |
| in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 22.65 (29.77) | 22.98 (32.80) | -0.01 | 16.54 (20.34) | 16.64 (21.51) | 0.00 | 19.47 (25.30) | 19.68 (27.50) | -0.01 |
| median [IQR] | 13.37 [5.00, 30.00] | 13.80 [5.01, 29.28] | -0.01 | 10.61 [2.74, 23.07] | 10.96 [3.67, 22.35] | -0.02 | 11.93 (25.30) | 12.32 (27.50) | -0.01 |
| Missing; n (%) | 579 (8.6%) | 581 (8.7%) | 0.00 | 850 (11.7%) | 891 (12.2%) | -0.02 | 1,429 (10.2%) | 1472 (10.5%) | -0.01 |
| Colonos; n (%) | 254 (3.8%) | 266 (4.0%) | -0.01 | 263 (3.6%) | 250 (3.4%) | 0.01 | 0,517 (3.7%) | 516 (3.7%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) | 196 (2.9%) | 192 (2.9%) | 0.00 | 160 (2.2%) | 164 (2.3%) | -0.01 | 0,356 (2.5%) | 356 (2.5%) | 0.00 |
| Flu vaccine; n (%) | 974 (14.5%) | 1,032 (15.4%) | -0.03 | 646 (8.9%) | 637 (8.7%) | 0.01 | 1,620 (11.6%) | 1669 (11.9%) | -0.01 |
| Mammogram; n (%) | 422 (6.3%) | 439 (6.6%) | -0.01 | 277 (3.8%) | 298 (4.1%) | -0.02 | 0,699 (5.0%) | 737 (5.3%) | -0.01 |
| Pap smear; n (%) | 104 (1.6%) | 103 (1.5%) | 0.01 | 118 (1.6%) | 125 (1.7%) | -0.01 | 0,222 (1.6%) | 228 (1.6%) | 0.00 |
| Pneumonia vaccine; n (%) | 1,207 (18.0%) | 1,261 (18.8%) | -0.02 | 624 (8.6%) | 622 (8.5%) | 0.00 | 1,831 (13.1%) | 1883 (13.5%) | -0.01 |
| PSA test or Prostate exam for DRE; n (%) | 963 (14.4%) | 952 (14.2%) | 0.01 | 792 (10.9%) | 802 (11.0%) | 0.00 | 1,755 (12.6%) | 1754 (12.5%) | 0.00 |
| Bone mineral density; n (%) | 157 (2.3%) | 163 (2.4%) | -0.01 | 79 (1.1%) | 78 (1.1%) | 0.00 | 0,236 (1.7%) | 241 (1.7%) | 0.00 |
| Use of Sympatomimetic agents; n (%) | 38 (0.6%) | 43 (0.6%) | 0.00 | 79 (1.1%) | 80 (1.1%) | 0.00 | 0,117 (0.8%) | 123 (0.9%) | -0.01 |
| Use of CNS stimulants; n (%) | 17 (0.3%) | 23 (0.3%) | 0.00 | 38 (0.5%) | 42 (0.6%) | -0.01 | 0,055 (0.4%) | 65 (0.5%) | -0.01 |
| Use of estrogens, progestins, androgens; n (%) | 204 (3.0%) | 180 (2.7%) | 0.02 | 287 (3.9%) | 298 (4.1%) | -0.01 | 0,491 (3.5%) | 478 (3.4%) | 0.01 |
| Use of Angiogenesis inhibitors; n (%) | 8 (0.1%) | 5 (0.1%) | 0.00 | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 0,008 (0.1%) | 6 (0.0%) | 0.04 |
| Use of Oral Immunosuppressants; n (%) | 16 (0.2%) | 15 (0.2%) | 0.00 | 22 (0.3%) | 19 (0.3%) | 0.00 | 0,038 (0.3%) | 34 (0.2%) | 0.02 |
| Use of fondaparinux or Bivalirudin; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of other direct thrombin inhibitors | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0 (0.0%) | #DIV/0! |
| (lepirudin, desirudin, argatroban); n (%) | | | | | | | | | |
| Use of Prasugrel ON CED; n (%) | 22 (0.3%) | 29 (0.4%) | -0.02 | 34 (0.5%) | 33 (0.5%) | 0.00 | 0,056 (0.4%) | 62 (0.4%) | 0.00 |
| Use of Prasugrel 180 to 1 day prior; n (%) | 47 (0.7%) | 61 (0.9%) | -0.02 | 56 (0.8%) | 52 (0.7%) | 0.01 | 0,103 (0.7%) | 113 (0.8%) | -0.01 |
| Duration of index hospitalization (i.e. anchor hospitalization LOS) | | | | | | | | | |
| mean (sd) | 3.97 (2.97) | 4.01 (3.08) | -0.01 | 3.40 (1.60) | 3.43 (1.62) | -0.02 | 3.67 (2.36) | 3.71 (2.43) | -0.02 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [2.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 (2.36) | 3.00 (2.43) | 0.00 |
| Number of D-dimer tests | | | | | | | | | |
| mean (sd) | 0.04 (0.22) | 0.04 (0.23) | 0.00 | 0.05 (0.24) | 0.06 (0.26) | -0.04 | 0.05 (0.23) | 0.05 (0.25) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.23) | 0.00 (0.25) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | |
| mean (sd) | 0.06 (0.31) | 0.06 (0.31) | 0.00 | 0.04 (0.27) | 0.04 (0.26) | 0.00 | 0.05 (0.29) | 0.05 (0.29) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.29) | 0.00 (0.29) | 0.00 |
| Number of PT or aPTTt tests | | . , , | | . , . | . , . | | , , | , , | |
| mean (sd) | 0.41 (1.41) | 0.41 (1.40) | 0.00 | 0.39 (0.97) | 0.38 (1.01) | 0.01 | 0.40 (1.20) | 0.39 (1.21) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.20) | 0.00 (1.21) | 0.00 |
| Number of Bleeding time tests | | [] | | | [,] | | \/ | (/ | |
| mean (sd) | 0.00 (0.04) | 0.00 (0.02) | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | 0.00 [0.00, 0.00] | 3.55 [5.56, 6.66] | 0.00 | 3.00 [0.00, 0.00] | 3.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| mean (sd) | 3.91 (0.75) | 3.92 (0.74) | -0.01 | 3.40 (0.61) | 3.40 (0.60) | 0.00 | 3.64 (0.68) | 3.65 (0.67) | -0.01 |

Table 1: Ticagrelor 90 mg vs Clopidogrel 75 mg

| median [IQR] | 4.00 [3.00, 4.00] | 4.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.48 (0.68) | 3.48 (0.67) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Drug eluting stent; n (%) | 1,231 (18.4%) | 1,211 (18.1%) | 0.01 | 2,311 (31.7%) | 2,256 (31.0%) | 0.02 | 3,542 (25.3%) | 3467 (24.8%) | 0.01 |
| Bare metal stent; n (%) | 5,572 (83.2%) | 5,570 (83.2%) | 0.00 | 6,125 (84.1%) | 6,043 (83.0%) | 0.03 | 11,697 (83.7%) | 11613 (83.1%) | 0.02 |
| Use of CYP inhibitors; n (%) | 1,377 (20.6%) | 1,380 (20.6%) | 0.00 | 1,243 (17.1%) | 1,220 (16.8%) | 0.01 | 2,620 (18.7%) | 2600 (18.6%) | 0.00 |
| Use of CYP inducers; n (%) | 7 (0.1%) | 6 (0.1%) | 0.00 | 10 (0.1%) | 8 (0.1%) | 0.00 | 0,017 (0.1%) | 14 (0.1%) | 0.00 |
| Commercial vs Medicare Advantage- Business | | | | | | | | | |
| Type Code - CORRECT ONE - TRUVEN | | | | | | | | | |
| Commercial; n (%) | 1,994 (29.8%) | 1,995 (29.8%) | 0.00 | 2,433 (33.4%) | 2,455 (33.7%) | -0.01 | 4,427 (31.7%) | 4450 (31.8%) | 0.00 |
| Medicare Advantage; n (%) | 4,703 (70.2%) | 4,702 (70.2%) | 0.00 | 4,850 (66.6%) | 4,828 (66.3%) | 0.01 | 9,553 (68.3%) | 9530 (68.2%) | 0.00 |
| Commercial vs Medicare Advantage- Business | ,, | , - ( , | | , , | , ( , | | -, (, | , | |
| Type Code | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 1,994 (29.8%) | 1,995 (29.8%) | 0.00 | - | - | #VALUE! | 1,994 (29.8%) | 1,995 (29.8%) | 0.00 |
| MCR = MEDICARE; n (%) | 4,703 (70.2%) | 4,702 (70.2%) | 0.00 | - | - | #VALUE! | 4,703 (70.2%) | 4,702 (70.2%) | 0.00 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| 2015); n (%) | ( ) | , | , | | | | , | . ( , | , |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 4,383 (60.2%) | 4,356 (59.8%) | 0.01 | 4,383 (60.2%) | 4,356 (59.8%) | 0.01 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 467 (6.4%) | 472 (6.5%) | 0.00 | 467 (6.4%) | 472 (6.5%) | 0.00 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 2,169 (29.8%) | 2,198 (30.2%) | -0.01 | 2,169 (29.8%) | 2,198 (30.2%) | -0.01 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 264 (3.6%) | 257 (3.5%) | 0.01 | 264 (3.6%) | 257 (3.5%) | 0.01 |
| Metropolitan Statistical Area - Urban (any MSA) | | | | | | | | | |
| vs Rural (non-MSA) | | | | | | | | | |
| Urban; n (%) | - | - | #VALUE! | 5,129 (70.4%) | 5,146 (70.7%) | -0.01 | 5,129 (70.4%) | 5,146 (70.7%) | -0.01 |
| Rural; n (%) | - | - | #VALUE! | 559 (7.7%) | 533 (7.3%) | 0.02 | 559 (7.7%) | 533 (7.3%) | 0.02 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 1,595 (21.9%) | 1,604 (22.0%) | 0.00 | 1,595 (21.9%) | 1,604 (22.0%) | 0.00 |
| N of Generic name drugs | | | | | | | | | |
| mean (sd) | 16.07 (12.36) | 15.97 (13.43) | 0.01 | 12.49 (8.99) | 12.30 (9.86) | 0.020138 | 14.20 (10.74) | 14.06 (11.71) | 0.01 |
| median [IQR] | 13.00 [8.00, 21.00] | 13.00 [7.00, 21.00] | 0.00 | 10.00 [6.00, 16.00] | 10.00 [5.00, 16.00] | 0 | 11.44 (10.74) | 11.44 (11.71) | 0.00 |
| N of Brand name drugs | | | | | | | | | |
| mean (sd) | 3.76 (5.67) | 3.73 (4.17) | 0.01 | 3.65 (5.13) | 3.63 (3.53) | 0.00 | 3.70 (5.40) | 3.68 (3.85) | 0.07 |
| median [IQR] | 1.00 [0.00, 5.00] | 2.00 [1.00, 5.00] | -0.20 | 2.00 [0.00, 5.00] | 2.00 [1.00, 5.00] | 0 | 1.52 (5.40) | 2.00 (3.85) | 0.07 |